## Cover page

ID-054-304

## Statistical Analysis Plan

## Official Title:

A Prospective, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 3 Study to Assess the Efficacy and Safety of Clazosentan in Preventing Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI), in Adult Subjects With Aneurysmal Subarachnoid Hemorrhage (aSAH)

# ClinicalTrials.gov Identifier:

NCT03585270

Date of document:

26 January 2023



# **CLAZOSENTAN (ACT-108475)**

# STATISTICAL ANALYSIS PLAN

## FOR CLINICAL STUDY REPORT

ID-054-304

## **REACT**

pRevention and trEatment of vAsospasm with ClazosenTan

A prospective, multi-center, double-blind, randomized, placebo-controlled, parallel-group, Phase 3 study to assess the efficacy and safety of clazosentan in preventing clinical deterioration due to delayed cerebral ischemia (DCI), in adult subjects with aneurysmal subarachnoid hemorrhage (aSAH)

Version 4

Document Number: D-23.039

26 January 2023

Property of Idorsia Pharmaceuticals Ltd


May not be used, divulged, published or otherwise disclosed without the consent of Idorsia Pharmaceuticals Ltd

# TABLE OF CONTENTS

| LI | ST OF ABBREVI | ATIONS AND ACRONYMS | 7 |
|---|---|---|---|
| 1 | INTRODUCTIO | )N | 9 |
| 2 | STUDY DESIG | N AND FLOW | 9 |
| | 2.1 Study of | lesign | 9 |
| | | visit and assessment schedule | |
| | | ew of analysis periods | |
| 3 | OBJECTIVES | | 11 |
| | 3.1 Primar | y objective | 11 |
| | 3.2 Second | lary objectives | 12 |
| | | bjectives | |
| 4 | ANALYSIS SE | ГЅ | 12 |
| | 4.1 Definit | ions of analysis sets | 12 |
| | 4.1.1 | Screened analysis set | |
| | | Randomized analysis set | |
| | | Full analysis set. | |
| | 4.1.4 | Safety analysis set | |
| | 4.2 Usage | of the analysis sets | |
| 5 | STUDY SUBJE | CT VARIABLES AND ANALYSES | 13 |
| | 5.1 Subject | t disposition | 14 |
| | 5.1.1 | Screening failures | |
| | 5.1.2 | Study completion/discontinuation | |
| | 5.1.3 | Study treatment completion/discontinuation | |
| | | ol deviations | |
| | | is sets | |
| | | t characteristics | |
| | _ | Demographics | |
| | | Baseline disease characteristics | |
| | 5.4.2.1 | Stratification factors | |
| | 5.4.2.2 | | |
| | | hospital admission | |
| | 5.4.2.3 | Neurological scales after admission and prior to Study dr | |
| | | initiation | 17 |
| | 5.4.2.4 | aSAH-related characteristics | 17 |

| | | 5.4.3 | Other baseline characteristics | 18 |
|---|---|---|---|---|
| | | 5.4.3.1 | Computed tomography scan results | 18 |
| | | 5.4.4 | Medical history and concomitant diseases and/or diagnoses | 19 |
| | | 5.4.5 | Previous and concomitant therapies | |
| | | 5.4.5.1 | Previous/concomitant medications | 20 |
| | | 5.4.5.2 | Non-drug treatments/interventions | 21 |
| | | 5.4.5.3 | Rescue therapies | 21 |
| | 5.5 | Study | treatment exposure and compliance | 23 |
| | | 5.5.1 | Exposure | 23 |
| | | 5.5.2 | Compliance with study treatment | 24 |
| 6 | EFF | FICACY VA | ARIABLES AND ANALYSES | 24 |
| | 6.1 | Overv | iew | 24 |
| | | 6.1.1 | Overall testing strategy | 25 |
| | | 6.1.2 | Estimands | 26 |
| | | 6.1.3 | Overview of primary and secondary efficacy analyses | |
| | | | including subgroups | 34 |
| | 6.2 | | y endpoint | |
| | | 6.2.1 | Variable | |
| | | 6.2.2 | Intercurrent events for the main estimand | 36 |
| | | 6.2.3 | Handling of missing data | |
| | | 6.2.4 | Hypothesis, statistical model and assumptions | |
| | | 6.2.5 | Main analysis | |
| | | 6.2.6 | Supportive analyses | |
| | | 6.2.6.1 | $\mathcal{E}$ | |
| | | 6.2.6.2 | 1 2 | 38 |
| | | 6.2.6.3 | | |
| | | | death | 38 |
| | | 6.2.7 | Subgroup analyses | 38 |
| | | 6.2.8 | Other analyses | |
| | 6.3 | | secondary endpoint | |
| | | 6.3.1 | Variable | |
| | | 6.3.2 | Intercurrent events for the main estimand | |
| | | 6.3.3 | Handling of missing data | |
| | | 6.3.4 | Hypothesis, statistical model and assumptions | |
| | | 6.3.5 | Main analysis | |
| | | 6.3.6 | Supportive analyses | |
| | | 6.3.7 | Subgroup analyses | 42 |
| | | 6.3.8 | Other analyses | |
| | 6.4 | | secondary endpoint | |
| | | 6.4.1 | Modified Rankin Scale | |
| | | 6.4.1.1 | Variable | 43 |

| 6.4.1.2 | Intercurrent events for the main estimand | 43 |
|-------------|-----------------------------------------------------------|----|
| 6.4.1. | | |
| 6.4.1.4 | 4 Hypothesis, statistical model and assumptions | 44 |
| 6.4.1. | | 44 |
| 6.4.1. | 6 Supportive/sensitivity analyses | 45 |
| 6.4.1. | | |
| 6.4.1. | 8 Other analyses | 45 |
| 6.4.2 | Glasgow Outcome Scale – Extended | 46 |
| 6.4.2. | | |
| 6.4.2.2 | 2 Intercurrent events for the main estimand | 46 |
| 6.4.2. | 3 Handling of missing data | 46 |
| 6.4.2.4 | 4 Hypothesis, statistical model and assumptions | 47 |
| 6.4.2.: | 5 Main analysis | 47 |
| 6.4.2. | 6 Supportive/sensitivity analyses | 47 |
| 6.4.2. | 7 Subgroup analyses | 48 |
| 6.4.2. | 8 Other analyses | 48 |
| 6.5 Subject | ct-reported endpoints | 48 |
| 6.5.1 | Montreal Cognitive Assessment | 49 |
| 6.5.1. | 1 Variables | 49 |
| 6.5.1.2 | 2 Analysis | 49 |
| 6.5.2 | EQ-5D-5L | 51 |
| 6.5.2. | 1 Variables | 51 |
| 6.5.2.2 | $oldsymbol{J}$ | |
| 6.5.3 | Ox-PAQ | |
| 6.5.3. | | |
| 6.5.3.2 | $oldsymbol{J}$ | |
| 6.5.4 | Stroke-Specific Quality of Life | 53 |
| 6.5.4. | | |
| 6.5.4.2 | | |
| 6.6 Multiv | variate long-term outcome | |
| 6.6.1 | Variables | |
| 6.6.2 | Analysis | |
| 6.7 Analy | rsis of pharmaco-economic variables | |
| 6.7.1 | Rescue therapies | |
| 6.7.2 | Specific (pre-specified) medical treatments and therapies | |
| 6.7.3 | Subject location/rehabilitation | |
| 6.7.3. | | |
| 6.7.3.2 | | |
| 6.7.4 | Employment status | |
| 6.7.4. | | |
| 6.7.4.2 | | |
| 6.7.4. | 3 Analysis | 58 |

| | 6.8 | Biomarker endpoints analysis | 58 |
|---|---|---|---|
| | 6.8 | .1 Variables | 59 |
| | 6.8 | .2 Analysis | 59 |
| 7 | SAFET | Y VARIABLES AND ANALYSES | 59 |
| | 7.1 | Adverse events | 59 |
| | 7.1 | .1 Variables | 60 |
| | 7.1 | .2 Analysis | 62 |
| | 7.2 | Laboratory tests | 64 |
| | 7.3 | Electrocardiography | 65 |
| | 7.4 | Vital signs | 66 |
| | 7.5 | Other safety variables and analyses | 66 |
| | 7.5 | | |
| | 7.6 | Subgroup analysis of safety variables | 67 |
| 8 | GENER | AL STATISTICAL METHODOLOGY | 67 |
| 9 | INTERI | M ANALYSES AND DATA MONITORING COMMITTEES | 67 |
| 10 | GENER | AL DEFINITIONS AND DERIVATIONS | 68 |
| | 10.1 | Handling of missing date | 68 |
| | 10.2 | General analysis variables | |
| | 10.3 | Study treatment administration error | 69 |
| | 10.4 | Other derivations | |
| 11 | CHANG | GES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE | |
| | | PROTOCOL | 70 |
| | 11.1 | Changes in the conduct of the study / data collection | 70 |
| | 11.1 | Changes to the analyses planned in the study protocol | |
| | 11.2 | Clarifications concerning endpoint definitions and related variables or | / 0 |
| | 11.5 | statistical methods. | 71 |
| | 11.4 | Additional analyses to those planned in the study protocol | |
| 12 | LIST O | F TABLES, LISTINGS AND FIGURES | 72 |
| | | ENCES | |
| 14 | APPEN | DICES | |
| | 14.1 | Revision History | |
| | 14.2 | Schedule of events | |
| | 14.3 | Change from pre-aSAH to post-aSAH status | |
| | 1/1/1 | Adverse events of special interest | 83 |

# LIST OF ABBREVIATIONS AND ACRONYMS

| AE | Adverse event |
|--------|--------------------------------------------------------|
| ALT | Alanine aminotransferase |
| aNIHSS | Abbreviated National Institutes of Health Stroke Scale |
| ANOVA | Analysis of variance |
| aSAH | Aneurysmal subarachnoid hemorrhage |
| AST | Aspartate aminotransferase |
| CEC | Clinical Event Committee |
| CI | Confidence interval |
| CMH | Cochran-Mantel-Haenszel |
| CSR | Clinical study report |
| CT | Computed tomography |
| DCI | Delayed cerebral ischemia |
| eCRF | Electronic case report form |
| EOS | End-of-Study |
| FAS | Full analysis set |
| GCS | Glasgow Coma Scale |
| GOSE | Glasgow Outcome Scale – Extended |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| ICU | Intensive care unit |
| IDMC | Independent Data Monitoring Committee |
| IE | Intercurrent event |
| IRC | Independent Radiology Committee |
| IRT | Interactive Response Technology |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mGCS | Modified Glasgow Coma Scale |
| MLA | Marked laboratory abnormality |
| MoCA | Montreal Cognitive Assessment |
| mRS | Modified Rankin Scale |
| OR | Odds ratio |
| Ox-PAQ | Oxford Participation and Activities Questionnaire |
| PCA | Principal Component Analysis |

| POM | Proportional odds model |
|--------|--------------------------------------------|
| PT | Preferred Term |
| QoL | Quality of life |
| RND | Randomized analysis set |
| RR | Relative risk |
| RRR | Relative risk reduction |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SCR | Screened analysis set |
| SI | Standard International |
| SOC | System Organ Class |
| SS-QoL | Stroke-Specific Quality of Life |
| TEAE | Treatment-emergent adverse event |
| VAS | Visual analog scale |
| WFNS | World Federation of Neurological Societies |
| WHO | World Health Organization |

# 1 INTRODUCTION

This statistical analysis plan (SAP) describes in detail the analyses and data presentation for the final clinical study report (CSR) for study ID-054-304 (REACT). Version 4 of the SAP is based on protocol version 7, dated 18 February 2022 [D-22.069] and replaces the previous SAP version 3, dated 27 September 2022. A revision history of the SAP is provided in Appendix 14.1.

Obvious corrections to address minor formatting errors or spelling mistakes may be performed at the time of analysis without amending this and related documentation (e.g., mock shells).

The study includes the study committees displayed in Table 1, each having a specific role.

Table 1 Study committees

| Committee | Responsibility |
|---|---|
| Independent Data Monitoring<br>Committee | Reviewing unblinded safety and efficacy data obtained in the study at regular intervals, and making appropriate recommendations based on the reported data. |
| Independent Radiology<br>Committee | Reviewing retrospectively (during the course of the study) the angiograms and CT scans submitted for each randomized subject to determine the presence of pre-defined radiological features and to perform required measurements. |
| Clinical Event Committee | Determining, based on a charter, whether the primary and main secondary endpoint (first component, see Section 6.3.1 for details) have been met. |

CT = computed tomography.

#### 2 STUDY DESIGN AND FLOW

## 2.1 Study design

This is a prospective, multi-center, double-blind, randomized, placebo-controlled, parallel-group, Phase 3 study.

Subjects will be randomized 1:1 to clazosentan 15 mg/h or placebo, stratified by their World Federation of Neurological Societies (WFNS) grade at hospital admission (I–II vs III–V), patient population (high-risk prevention vs early treatment), and age at hospital admission ( $\leq 60$  and > 60 years). Recruitment into the early treatment stratum was discontinued from protocol version 6 (29 April 2021) onwards.

Overall, the study will enroll 400 subjects in 2 treatment groups, 200 subjects per group.

The study will be conducted at approximately 100 sites in 15 countries.

Once randomized, the subjects will enter a double-blind treatment period of a maximum duration of 14 days. This will be sequentially followed by a safety follow-up period of 24 hours and an extended follow-up period for safety and efficacy assessment terminating with an End-of-Study (EOS) visit at Week 24 post aneurysmal subarachnoid hemorrhage (aSAH).


The overall study design for the high-risk prevention group is depicted in Figure 1.

Note: The study design of the early treatment stratum is provided in Figure 2 although recruitment into this group was discontinued from protocol version 6 onwards.

Figure 1 Study design for the high-risk prevention group



Figure 2 Study design for the early treatment stratum



## 2.2 Study visit and assessment schedule

The study periods and 'visits' with their respective time windows are listed in the Visit and assessment schedules [see Appendix 14.2].

Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

## 2.3 Overview of analysis periods

An overview of the study periods and 'visits' is provided below.

The study comprises the following consecutive periods:

**Screening period:** Starts with the signature of the informed consent form (ICF) and ends with subject randomization.

**Treatment period:** Starts immediately with the baseline assessments followed by the initiation of study drug infusion and ends with the permanent discontinuation of study drug.

**Observation period for the primary endpoint:** This period covers the interval over which the subject may qualify for the primary endpoint of the study. It starts with the initiation of study drug infusion and ends on and includes Day 14 post-study drug initiation.

**24-hour safety follow-up period:** Starts with the permanent discontinuation of study drug and ends 24 hours later.

The End-of-Treatment assessments are included in the 24-hour safety follow-up period. These assessments are performed within 2 hours following permanent discontinuation of study drug.

**Extended follow-up period:** Starts after the 24-hour safety follow-up period and ends with the EOS visit, occurring 24 weeks after the aSAH.

**EOS** (individual subject): This is defined as the last visit performed for the study (i.e., the EOS visit, performed 24 weeks after the aSAH), or the date of premature discontinuation from the study, if applicable.

**EOS** (study level): This time point occurs when the last subject completes his/her EOS visit.

#### 3 OBJECTIVES

The overall objective of this study is to determine the clinical efficacy of clazosentan in a population at high risk of developing ischemic complications post-aSAH, and to further evaluate its safety and tolerability in this population.

## 3.1 Primary objective

To determine the efficacy of clazosentan in preventing clinical deterioration due to delayed cerebral ischemia (DCI) in subjects with aSAH.

Efficacy will primarily be assessed based on a reduction in the clazosentan group compared to the placebo group in the occurrence of clinical deterioration due to DCI up to 14 days post-study drug initiation.

## 3.2 Secondary objectives

- To evaluate the effect of clazosentan on the occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation defined as:
- all-cause cerebral infarction  $\geq 5$  cm<sup>3</sup> or
- cerebral infarction < 5 cm<sup>3</sup> in subjects with clinical deterioration due to DCI.
- To evaluate the effect of clazosentan on long-term clinical outcome, cognition, and health-related Quality of Life (QoL) at Week 12 post-aSAH and QoL at Week 24 post-aSAH.
- To evaluate the safety and tolerability of clazosentan in the selected population up to 24 hours post-study drug discontinuation.

## 3.3 Other objectives

To evaluate the effect of clazosentan on healthcare resource utilization.

#### 4 ANALYSIS SETS

## 4.1 Definitions of analysis sets

#### 4.1.1 Screened analysis set

The Screened analysis set (SCR) includes all subjects for whom informed consent to participate in the study has been obtained and who have a subject identification number.

#### 4.1.2 Randomized analysis set

The Randomized analysis set (RND) comprises all subjects who have been assigned to a study treatment.

#### 4.1.3 Full analysis set

The Full analysis set (FAS) comprises all subjects from the RND who started the study treatment. The rationale for this choice of the FAS is that, per study design, due to the emergency setting, the investigator has the possibility to withdraw subjects from the study before study drug initiation for safety or other reasons (e.g., due to a sudden deterioration of the clinical status post randomization). Defining the FAS as all subjects who have started study treatment is expected to preserve the intent-to-treat principle, because: a) randomized but untreated subjects will be rare (in previous Phase 3 studies, i.e., CONSCIOUS-2 and -3, less than 1% of the randomized subjects were not treated), and b) the decision whether or not to begin treatment cannot be influenced by knowledge of the assigned treatment.

To adhere to the intent-to-treat principle, if not otherwise stated subjects will be evaluated according to their assigned study treatment (which might differ from the actual treatment received) and stratum information as recorded in the Interactive Response Technology (IRT) system.

#### 4.1.4 Safety analysis set

The Safety analysis set (SAF) comprises all subjects who have been assigned to a study treatment and who have started the study drug.

Subjects will be evaluated according to the actual treatment they received, which may differ from the randomly assigned treatment.

In the event of an administration error, i.e., a subject was administered both placebo and active treatment, the subject will be analyzed as 'active treatment' ('clazosentan').

## 4.2 Usage of the analysis sets

If not otherwise stated, the listings will be produced on the FAS for efficacy and on the SAF for safety.

For the tables and figures, the sets are indicated in Table 2.

Table 2 Overview of the different analysis sets and their usage

| | Analysis sets | | | |
|---|---|---|---|---|
| Analyses | SCR | RND | FAS | SAF |
| Subject disposition, | X | X | | |
| Analysis sets | | | X | X |
| Protocol deviations | | [x] | X | |
| Demographics characteristics | | [x] | X | [y] |
| Baseline disease characteristics | | [x] | X | [y] |
| Medical history and current medical conditions | | [x] | X | |
| Previous and concomitant therapies | | [x] | X | |
| Study treatment exposure | | | | X |
| Primary efficacy endpoint | | [x] | X | |
| Secondary efficacy endpoints | | [x] | X | |
| Exploratory efficacy endpoint | | | X | |
| Quality of life endpoints | | | X | |
| Pharmaco-economic endpoints | | | X | |
| Biomarker endpoints | | | X | |
| Safety endpoints | | | | X |

Note: X: main analysis set; [x]: if RND and FAS differ by more than 5%, some tables may be replicated on the RND; [y]: if FAS and SAF differ by more than 5%, some tables may be replicated on the SAF.

FAS = Full analysis set; RND = Randomized analysis set; SAF = Safety analysis set; SCR = Screened analysis set.

## 5 STUDY SUBJECT VARIABLES AND ANALYSES

A listing of the randomization scheme and codes will be produced for randomized subjects only (as per ICH E3 16.1.7).

The analyses defined in this section on the FAS will be repeated on the RND if the RND and FAS differ by more than 5%.

## 5.1 Subject disposition

An overview of the recruitment for each country/site will be presented for the SCR and will comprise the following variables:

- N (%) of subjects screened overall
- N (%) of subjects randomized

An overview of the number of subjects randomized in each treatment group (according to the assigned treatment group) and overall for each country/site will be presented for the RND.

An overview of subject disposition over the course of the study will be presented for the RND in a table by treatment group (except for Screened, which is only summarized for the total column) and overall, and comprises the following variables:

- N (%) of randomized subjects
- N (%) of treated subjects
- N (%) of subjects who completed the study treatment
- N (%) of subjects who prematurely discontinued the study treatment
- N (%) of subjects who completed the study
- N (%) of subjects who prematurely discontinued the study

A listing will be produced with the subjects randomized but not treated.

#### 5.1.1 Screening failures

The number and percentage of subjects who failed screening and the reasons for screening failure will be summarized for the SCR (Overall). All reasons for screening failure will be included in a listing together with the screening failure date. An additional listing will present the list of eligibility criteria not met for the screened set where the screen-failed subjects will be flagged.

#### 5.1.2 Study completion/discontinuation

The reasons for study discontinuation will be tabulated by treatment group and overall on the randomized set.

A listing will be produced for all the subjects of the FAS who discontinued the study. It will display the EOS date, the EOS day (relative to start of study treatment), and the reason for discontinuation from the study.

Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

## 5.1.3 Study treatment completion/discontinuation

The reasons for treatment discontinuation as collected in the study treatment infusion log in the electronic case report form (eCRF) will be tabulated by treatment group and overall on the FAS.

Subjects who prematurely discontinued the study treatment and subjects randomized but not treated are also included in the listing described in Section 5.1.2. The listing displays the end date of study treatment, the study day on which treatment was discontinued (relative to start of study treatment), and the reason for treatment discontinuation.

#### 5.2 Protocol deviations

The number and percentage of subjects with at least one important protocol deviation will be summarized in a table by treatment group and overall on the FAS. The number and percentage of subjects with at least one deviation in each category and sub-category will also be presented. Similar tables will be produced for:

- subjects with at least one protocol deviation, regardless of importance (i.e., important or non-important)
- subjects with at least one important protocol deviation related to COVID-19
- subjects with at least one protocol deviation related to COVID-19, regardless of importance (i.e., important or non-important)

These tables will be repeated on the RND if the RND and FAS differ by more than 5%.

Important and non-important protocol deviations will be displayed in a listing on the screened set. It will include all deviation descriptions, identifiers and categories. Subjects without any protocol deviations will not be included in this listing.

#### 5.3 Analysis sets

The number and percentage of subjects included in the RND and FAS will be summarized in a table, by planned treatment group (i.e., as randomized) and overall, for the RND.

A similar table will be produced for the SAF as treated.

The inclusion/exclusion of subjects for each analysis set will be listed for the SCR. A listing displaying both planned and actual treatment groups will be produced for subjects having received in error a treatment different from the one they were randomized to.

## 5.4 Subject characteristics

#### 5.4.1 Demographics

Demographic characteristics will be summarized by treatment group and overall using descriptive statistics for continuous and categorical data on the FAS. It will include the following characteristics:

- Age (years) at hospital admission (continuous; categorized according to EudraCT as: adults [18–64], and elderly [65–84 and  $\geq$  85])
- Sex (categorized as: Male, Female)
- Race (categorized as: American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or other Pacific Islander, White, Other, Not permitted as per legislation/regulation)
- Ethnicity (categorized as: Hispanic or Latino, Not Hispanic or Latino, Unknown, Not permitted as per legislation/regulation)
- Body weight (kg) at hospital admission
- Height (cm)
- Body mass index (kg/m<sup>2</sup>), derived as weight (kg) / (height [cm] / 100)<sup>2</sup>
- Geographical location, derived from the country of enrollment (categorized as: USA vs non-USA, Europe vs non-Europe)

All these characteristics will be displayed in a listing.

The variables 'Woman of childbearing potential' and 'Reason for not being of childbearing potential' will not be summarized but will be listed.

This table will be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

This table will also be produced for the good neurological recovery subgroup (subjects who had  $mGCS \ge 14$  and aNIHSS = 0 prior to study drug start) and its complement.

#### 5.4.2 Baseline disease characteristics

#### 5.4.2.1 Stratification factors

The following variables will be summarized by treatment group on the FAS using descriptive statistics for categorical variables:

- Age at hospital admission categorized as:  $\leq 60, > 60$
- WFNS grade as assessed in the IRT system (categorized as: I–II, III–V)
- Patient population: high-risk vs early treatment

This table will be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

This table will also be produced for the good neurological recovery subgroup (subjects who had  $mGCS \ge 14$  and aNIHSS = 0 prior to study drug start) and its complement.

# 5.4.2.2 WFNS, total Glasgow Coma Scale score and motor deficit at hospital admission

WFNS grade, total Glasgow Coma Scale (GCS) score and presence of motor deficit at hospital admission will be summarized by treatment group and overall using descriptive

statistics for continuous and categorical data on the FAS. This table will include the following characteristics:

- WFNS grade as assessed in the IRT system (categorized as: I, II, III, IV, V)
- GCS score (ranges from 3 [deep coma] to 15 [fully awake person], continuous and categorized as: 3–6, 7–12, 13–14, 15])
- Motor deficit (categorized as: Present, Absent)

This table will also be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

- As 'WFNS grade at hospital admission' is collected both in the eCRF and in the IRT system. If there is a confirmed discrepancy at the time of database lock between the eCRF and the IRT system the following table will be produced: WFNS grade as assessed by investigator (categorized as: I, II, III, IV, V)
- WFNS grade as assessed by investigator (categorized as: I–II, III–V)

It will also be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

These characteristics (WFNS grade, total GCS score, and presence of motor deficit) evaluated at hospital admission, post aneurysm-securing procedure, and prior to randomization will be displayed in a listing for the FAS.

The discrepancies between WFNS collected in eCRF and in the IRT system will be flagged in the listing and the value collected in the eCRF system will also be displayed.

## 5.4.2.3 Neurological scales after admission and prior to Study drug initiation

The last available modified GCS (mGCS) and abbreviated National Institutes of Health Stroke Scale (aNIHSS) collected prior to study drug initiation will be summarized by treatment group and overall using descriptive statistics for continuous variable on the FAS.

This table will be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

#### 5.4.2.4 aSAH-related characteristics

Current aSAH-related characteristics will be summarized by treatment group and overall, using descriptive statistics for continuous and categorical data on the FAS. It will include the following characteristics:

• Aneurysm-securing procedure(s) performed prior to study drug initiation (categorized as: surgical clipping, endovascular coiling, other). If the two procedures have been sequentially used, only the latest one will be used

- Time (hours, continuous) elapsed between date/time of the aneurysm rupture and stop date/time of the aneurysm-securing procedure(s) when they are both available (i.e., no imputation for missing or partial dates and times)
- Location of the ruptured aneurysm (Supraclinoid internal carotid artery segments, Middle cerebral artery segments, Anterior cerebral artery segments, Anterior communicating artery, Posterior communicating artery, Distal vertebral artery segments, Basilar artery, Posterior cerebral artery segments, Other)
- Largest diameter of the ruptured aneurysm (mm) (continuous and categorized as: ≤ 5,
   > 5)
- Total number of aneurysm(s) repaired (ruptured or unruptured, categorical).
- Time from aSAH to end of the securing procedure (until the end of the last procedure used)
- Number of previous aSAH episodes (categorical)
- Total number of unruptured aneurysm(s) repaired (categorical)
- Occurrence of complications of the aneurysm-securing procedure (categorical: yes, no) and by type (Intracranial hemorrhage, Intraoperative cerebral artery thrombosis, Cardiac arrest, Seizure, Intracranial hypertension, Brain edema or swelling, Cerebral infarction/ischemia, Cerebral vasospasm, Artery dissection, Severe hemodynamic event, Other coiling or other surgical complications). The categories are not mutually exclusive

This table will be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

This table will also be produced for the good neurological recovery subgroup (i.e., subjects who had  $mGCS \ge 14$  and aNIHSS = 0 prior to study drug start) and its complement.

Subject-level current aSAH history and the peri-operative complications will be provided in a listing. Another listing will be produced displaying the aneurysm-securing procedure(s) performed prior to study drug initiation for all subjects.

#### 5.4.3 Other baseline characteristics

## 5.4.3.1 Computed tomography scan results

The following common findings at hospital admission as adjudicated by the Independent Radiology Committee (IRC) Review will be summarized by treatment group and overall on the FAS:

- Hydrocephalus
- Intraparenchymal hemorrhage
- Intraventricular hemorrhage
- Extracerebral hematoma
- Ventricular drainage

- Intracranial pressure monitoring device
- Midline shift

The number and percentage of subjects with at least one finding will also be presented.

The clot thickness will be summarized overall and separately for the good neurological recovery subgroup (i.e., subjects who had  $mGCS \ge 14$  and aNIHSS = 0 prior to study drug start) and its complement, according to the following categories:

- Diffuse thick, Diffuse thin, Local thick, Local thin, None, Unable to assess.
- Diffuse thick, Other, Unable to assess.

All these tables will also be repeated on the RND if the RND and FAS differ by more than 5%, and on the SAF if the FAS and the SAF differ by more than 5%.

## 5.4.4 Medical history and concomitant diseases and/or diagnoses

Reported terms are mapped to Preferred Terms (PTs) using MedDRA v25.

**Medical history** covers all diseases or diagnoses ended before or on the day of ICF signature (i.e., ongoing question is answered "No" in the eCRF).

Concomitant diseases and/or diagnoses are all diseases or diagnoses started before the day of ICF signature and ongoing at time of ICF signature (i.e., ongoing question is answered "Yes" in the eCRF).

Concomitant diseases and/or diagnoses not related to a protocol mandated procedure are all diseases or diagnoses not related to a study protocol mandated procedure started between ICF signature (included) and study drug initiation.

Medical history and concomitant diseases and/or diagnoses will be summarized separately on the FAS, by treatment group and overall. The number and percentage of subjects with at least one item of medical history are presented overall and by individual PT. Medical history and concomitant diseases and/or diagnoses will be sorted by descending frequencies of preferred name based on all treatment groups combined. This table will also be repeated on the RND if the RND and FAS differ by more than 5%.

A listing will be produced for all subjects with medical history, concomitant diseases and/or diagnoses and concomitant diseases and/or diagnoses not related to study protocol mandated procedure. The concomitant diseases and/or diagnoses not related to study protocol mandated procedure and started between ICF signature and study drug initiation will be flagged.

## 5.4.5 Previous and concomitant therapies

#### 5.4.5.1 Previous/concomitant medications

Therapies collected will be coded using the WHO Drug Global reference dictionary that employs the WHO Anatomical Therapeutic Chemical (ATC) classification system. The WHO Drug Global version used for reporting (B format 1 March 2022) will be specified in the footnote of the applicable output.

The medications will be summarized on the FAS according to the categories displayed in Table 3.

Table 3 Definition of categories for reporting previous/concomitant medications

| Category | Definition |
|---|---|
| Previous medications | Start and end date before the signature of the ICF |
| Study concomitant medications | Ongoing or started after ICF |
| Study treatment concomitant | Ongoing at time of Study treatment initiation |
| medications | or |
| | Start date equal to or after study drug initiation but before or |
| | the day of study drug discontinuation |
| Study concomitant medications started | Start date after study drug discontinuation and up to 24 h |
| during the 24 h follow-up period | study drug discontinuation |
| following study drug discontinuation | |

ICF = informed consent form.

Number (%) of subjects having taken at least one previous or concomitant medication will be presented overall and by treatment group, by ATC class (level 4 or next highest available level), and preferred name within each ATC class. A table will be produced for each category described in Table 3. Previous and concomitant medications will be sorted by ATC class and preferred name within each ATC class by descending frequency based on all treatment groups combined. These tables will also be repeated on the RND if the RND and FAS differ by more than 5%.

If the start date/time is missing, the medication will be considered as concomitant with the study and with the study treatment unless the end date is before the signature of the ICF or before study drug initiation, respectively.

If both start and end date are missing, the medication will be considered as concomitant with the study and with the study treatment.

If the start and/or end date are partially missing, the medication will be considered as concomitant with the study treatment and/or with the study unless it contradicts with the partial information available. For general rules regarding management of partial dates see Section 10.1.

A listing will be produced for all subjects with previous/concomitant medications (all categories specified in Table 3). This listing will include a flag identifying the medication started after ICF signature and before study drug initiation.

## 5.4.5.2 Non-drug treatments/interventions

Non-drug therapies, except rescue therapies, are defined as follows:

- Intracranial pressure monitoring
- Ventricular drainage
- Shunt (ventriculoperitoneal or ventriculoatrial)
- Subdural/epidural hematoma evacuation
- Lumbar drainage
- Mechanical ventilation
- Tracheostomy
- Intra-Aortic Balloon Counter-Pulsation

The number and percentage of subjects having started at least one non-drug treatment/intervention will be presented (i) overall and by therapies and (ii) overall and by treatment group on the FAS. It will be displayed overall and by period of emergence (prior to randomization; from randomization [included] up to hospital discharge [included]; from hospital discharge up to Week 12 [included]; after Week 12). Therapies will be sorted by descending frequency based on all treatment groups combined.

For general rules regarding management of partial dates see Section 10.1.

A listing will be produced for all subjects who received a non-drug treatment/intervention.

## 5.4.5.3 Rescue therapies

Rescue therapies will be summarized on the FAS according to the categories displayed in Table 4.

Table 4 Definition of categories for rescue therapies

| Category | Definition |
|---|---|
| Protocol-Specific Rescue Therapy | <ul> <li>Non-drug treatment/intervention: balloon angioplasty<br/>reported as 'cerebral angioplasty'.</li> </ul> |
| | • Concomitant medications reported as: (i) Intravenous vasodilators which were preceded by intra-arterial vasodilators or cerebral angioplasty, or (ii) intra-arterial/intrathecal/intra-cisternal/intraventricular administration of vasodilators or ozagrel, i.e., CM ticked as rescue medication in the eCRF and with one of the following ATC codes: C08CA, C08DA, G04BE, C01DA, C01CE, B01AC, R03DX, A03AD and those started with C04. |
| Local rescue therapy | <ul> <li>Concomitant medications reported as 'Administered as a<br/>rescue medication for vasospasm', excluding Protocol-<br/>Specific Rescue Therapy defined above.</li> </ul> |
| | • All therapies reported as 'Other' on the 'Non-drug treatment/intervention' form. |

ATC = Anatomical Therapeutic Chemical.

The incidence of protocol-specific rescue therapy and local rescue therapy within each treatment group will be displayed overall and by period of emergence together with the exact 95% confidence interval (CI) (Clopper-Pearson formula). The corresponding between-treatment group difference will be tested using a Cochran-Mantel-Haenszel (CMH) stratified by factors used in the randomization, i.e., WFNS grade (I–II vs III–V) and age ( $\leq 60$  and > 60 years) at admission. Both will be tested at the two-sided significance level of alpha = 0.05. Treatment effect will be quantified by means of the relative risk reduction (RRR) for clazosentan together with its 95% CI.

The use of rescue therapy overview will be produced by treatment group and overall on the FAS and will display:

- Number (%) of subjects having received at least one protocol-specific rescue therapy
- Number (%) of subjects having received at least one local rescue therapy
- Number (%) of subjects having received at least one protocol-specific or local rescue therapy
- Number (%) of subjects having received at least one protocol-specific, non-drug treatment / intervention (balloon angioplasty reported as 'cerebral angioplasty')
- Total number of days with protocol-specific rescue therapy, excluding overlap, i.e., if several rescue therapies are given on the same day, then the duration under rescue therapy is one day

• Total number of days with protocol-specific rescue therapy or local rescue therapy, excluding overlap, i.e., if several rescue therapies are given on the same day, then the duration under rescue therapy is one day

The following tables will be produced by treatment group on the FAS, by period of emergence (from randomization up to hospital discharge (included), and from hospital discharge up to Week 12 (included):

- The number and percentage of subjects having received at least one protocol-specific non-drug treatment / intervention rescue therapy overall, and by ATC code
- The number and percentage of subjects having received at least one protocol-specific medication rescue therapy overall, and by ATC code
- The number and percentage of subjects having received at least one local non-drug treatment / intervention rescue therapy overall, and by ATC code
- The number and percentage of subjects having received at least one local medication rescue therapy overall, and by ATC code

Hospital discharge date (time) is defined as the latest end/discharge date (time) reported with subject location equal to 'Critical care unit or equivalent', 'Specialized care ward' or 'General care ward' among the location reported for the initial hospitalization.

For general rules regarding management of partial dates see Section 10.1.

Rescue medications will be sorted by descending frequency of the number of subjects in the clazosentan group.

Tables will also be repeated on the RND if the RND and FAS differ by more than 5%. Listings with all rescue medication defined in Table 4 will be produced on the FAS, including the category (protocol-specific vs local), the period of emergence and the number of days relative to study drug initiation.

## 5.5 Study treatment exposure and compliance

Study treatment duration and compliance are defined for the treatment period.

#### 5.5.1 Exposure

Study treatment duration (in days) is defined as the number of days between the study treatment start date/time and the study treatment end date/time, regardless of treatment interruptions.

The descriptive statistics on the study treatment duration will be displayed overall and by treatment group for the SAF, Duration in subject-years will also be summarized. The definition of a year is 365.25 days.

Study treatment duration will also be summarized using the following categories  $\leq 3$ ,  $> 3-\leq 5$ ,  $> 5-\leq 10$ ,  $> 10-\leq 14$  and > 14 days.

Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

A listing will be produced displaying the study treatment duration and include the reason for permanent study treatment discontinuation.

## 5.5.2 Compliance with study treatment

Compliance with study treatment will be assessed using the proportion of subjects having received the study treatment for the expected duration as per the protocol: for a maximum of 14 days, for at least 10 days in the high-risk stratum, and for at least 6 days in the early treatment stratum. For each subject the observed treatment duration (difference between datetime of study drug start and stop excluding periods of temporary study drug interruptions) will be categorized as:

- 'Lower than expected' if the observed treatment duration is < 10 days or < 6 days for subjects in the in the high-risk or early treatment stratum respectively.
- 'As expected' if the observed treatment duration is ≥ 10 and ≤ 14 days or ≥ 6 and ≤ 14 days for subjects in the in the high-risk or early treatment stratum respectively
- 'Higher than expected' if the observed treatment duration is > 14.

These categories will be summarized overall and by treatment group using descriptive statistics for categorical variable on the FAS separately for the high-risk and early treatment stratum.

Number of days treated will also be summarized overall and by treatment group using a frequency table on the FAS for the high-risk and early treatment stratum separately.

#### 6 EFFICACY VARIABLES AND ANALYSES

A listing will be produced on the FAS with the individual data used in the analyses of the primary endpoint (including sensitivity analyses), the main secondary endpoint (including the originally planned main secondary endpoint [see Section 11.1 for details]), and the other secondary endpoints (i.e., poor mRS and poor GOSE).

Tables displaying SAS procedure outputs will be produced for the main analysis of the four endpoints included in the hierarchical testing strategy.

#### 6.1 Overview

If not otherwise stated, and according to the intent-to-treat principle, all the analyses presented in this section will be performed 'as randomized' and 'as stratified', that is, according to the treatment group and stratum allocated in the IVRS system.

If not otherwise stated, all analyses stratified/adjusted on the randomization stratification factors will be stratified/adjusted on [see Section 11.2 for details]:

- Hospital admission WFNS grade (as collected in IVRS) dichotomized as I–II vs III–V
- Age at hospital admission  $\leq 60 \text{ vs} > 60 \text{ years}$

## **6.1.1** Overall testing strategy

Four null hypotheses will be tested according to a hierarchical procedure, at the two-sided significance level of 0.05 until first non-rejection.

The first null hypothesis  $H_{10}$ , is that there is no difference between clazosentan 15 mg/h and placebo in the occurrence of clinical deterioration due to DCI from study drug initiation up to 14 days post-study drug initiation. The alternative hypothesis  $H_{1a}$  is that there is a difference between these groups:

$$H_{10}$$
:  $p_{1,plac} = p_{1,clazo}$  vs  $H_{1a}$ :  $p_{1,plac} \neq p_{1,clazo}$ 

Here  $p_{1,plac}$  and  $p_{1,clazo}$  denote the incidence of clinical deterioration due to DCI in the placebo and clazosentan groups, respectively. This hypothesis will be tested at a two-sided significance level of 0.05.

Superiority will be concluded if the lower limit of the two-sided 95% CI for the RRR of clazosentan compared to placebo is greater than 0.

The second null hypothesis  $H_{20}$ , which will be tested only if H10 is rejected, is that there is no difference between clazosentan and placebo in the occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation defined as: all-cause cerebral infarction  $\geq 5$  cm<sup>3</sup> or cerebral infarction  $\leq 5$  cm<sup>3</sup> in subjects with clinical deterioration due to DCI. The alternative hypothesis H2a is that there is a difference between these groups:

$$H_{20}$$
:  $p_{2,plac} = p_{2,clazo}$  vs  $H_{2a}$ :  $p_{2,plac} \neq p_{2,clazo}$ 

Here  $p_{2,plac}$  and  $p_{2,clazo}$  denote the incidence of occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation defined as: all-cause cerebral infarction  $\geq 5$  cm<sup>3</sup> or cerebral infarction  $\leq 5$  cm<sup>3</sup> in subjects with clinical deterioration due to DCI in the placebo and clazosentan groups, respectively. This hypothesis will be tested at a two-sided significance level of 0.05.

Superiority will be concluded if the lower limit of the two-sided 95% CI for the RRR of clazosentan compared to placebo is greater than 0.

The third null hypothesis H<sub>30</sub>, which will be tested only if H<sub>20</sub> is rejected, is that there is no difference between clazosentan and placebo in the proportion of subjects with a poor mRS score at Week 12 post-aSAH. The alternative hypothesis H<sub>3a</sub> is that there is a difference between these groups:

$$H_{30}$$
:  $p_{3,plac} = p_{3,clazo}$  vs  $H_{3a}$ :  $p_{3,plac} \neq p_{3,clazo}$ 

Here p<sub>3,plac</sub> and p<sub>3,clazo</sub> denote the proportion of subjects with a poor mRS at Week 12 post-aSAH in the placebo and clazosentan groups, respectively. This hypothesis will be tested at a two-sided significance level of 0.05.

Superiority will be concluded if the lower limit of the two-sided 95% CI for the RRR of clazosentan compared to placebo is greater than 0.

The fourth null hypothesis  $H_{40}$ , which will be tested only if  $H_{30}$  is rejected, is that there is no difference between clazosentan and placebo in the proportion of subjects with a poor Glasgow Outcome Scale – Extended (GOSE) score at Week 12 post-aSAH. The alternative hypothesis  $H_{4a}$  is that there is a difference between these groups:

H<sub>40</sub>: 
$$p_{4,plac} = p_{4,clazo}$$
 vs H<sub>4a</sub>:  $p_{4,plac} \neq p_{4,clazo}$ 

Here p<sub>4,plac</sub> and p<sub>4,clazo</sub> denote the proportion of subjects with a poor GOSE at Week 12 post-aSAH in the placebo and clazosentan groups, respectively. This hypothesis will be tested at a two-sided significance level of 0.05.

Superiority will be concluded if the lower limit of the two-sided 95% CI for the RRR of clazosentan compared to placebo is greater than 0.

The study will be considered successful if the first null hypothesis  $(H_{10})$  is rejected.

#### 6.1.2 Estimands

The estimands [ICH 2019] associated with endpoints described in Section 6.1.1 and their four attributes are given in Table 5. Estimands are defined by four attributes: Target population, Endpoint, Strategy for addressing intercurrent events (IEs), and Population-level summary.

The IEs considered in this study are:

| Intercurrent Event | Affects<br>primary<br>endpoint | Affects main secondary endpoint | Affects other secondary endpoints |
|---|---|---|---|
| Death | Yes | Yes | Yes |
| Unevaluable for neurological status and received rescue therapy for relevant vasospasm | Yes | Yes | Yes |
| Unevaluable for neurological status for vasospasms-related-reason | Yes | No | No |
| Early discharge followed by rehospitalization due to DCI | Yes | No | No |
| Early discharge without follow-up at Day 14 | Yes | No | No |
| Withdrawal of consent | Yes | Yes | Yes |
| Rescue therapy for non-relevant vasospasm | Yes | Yes | Yes |

#### Confidential

Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

| Permanent/temporary treatment discontinuation | Yes | Yes | Yes |
|-----------------------------------------------|-----|-----|-----|
|-----------------------------------------------|-----|-----|-----|

DCI = delayed cerebral ischemia.

IEs considered for the primary endpoint (clinical deterioration due to DCI) can be categorized as:

- IE suggestive of a clinical deterioration: death, unevaluable for neurological status and received rescue therapy for relevant vasospasm, unevaluable for neurological status for vasospasms-related reason, early discharge followed by rehospitalization due to DCI
- IE precluding assessment of the endpoint: withdrawal of consent and early discharge without follow-up at day 14
- IE that may affect the occurrence of clinical deterioration: use of rescue therapy for non-relevant vasospasm
- IE that can impact the estimation of treatment effect: permanent/temporary treatment discontinuation

IEs considered for the main secondary endpoint (clinically relevant cerebral infarction) are:

- IE suggestive of a cerebral infarction: death
- IE precluding assessment of the endpoint: withdrawal of consent
- IE that may affect the occurrence of clinical deterioration and thus ultimately cerebral infarction: use of rescue therapy (independently of whether it was provided for a relevant or non-relevant vasospasm)
- IE that can impact the estimation of treatment effect: permanent/temporary treatment discontinuation

IEs considered for the other secondary endpoints are the same as those for the main secondary endpoint.

The strategies used in this study to address IEs are:

- Composite strategy: The IE is incorporated into the outcome variable, e.g., any subject who died is assumed to meet the endpoint
- Hypothetical strategy: When the IE occurred, the observed (or missing) values are substituted by the ones of a hypothetical scenario where the IE would have not occurred, e.g., final outcome for a subject that withdrew consent is predicted using the data collected up to the time of consent withdrawal
- Treatment policy: The data collected are analyzed irrespective of the occurrence of the IE, e.g., the final outcome of a subject is analyzed irrespective of whether the subject discontinued study treatment

Within a given estimand different strategies are employed depending on the type of IEs considered. The efficacy estimands are detailed in Table 5. The estimands' differences vs the primary or secondary estimand (as appropriate) are indicated in bold.

Table 5 Estimands for efficacy endpoints

| Estimand | Target population | Endpoint | Strategy for addressing intercurrent events | Population-level summary |
|---|---|---|---|---|
| Primary Efficacy Endpoint | | | | |
| Main Estimand | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | The primary efficacy endpoint is the occurrence of clinical deterioration due to DCI, from study drug initiation up to 14 days post-study drug initiation. | Composite strategy: Death, Unevaluable for neurological status and received Rescue therapy <sup>[c]</sup> for relevant vasospasm, Unevaluable for neurological status for vasospasm-related reason, early discharge followed by rehospitalization due to DCI Hypothetical <sup>[a]</sup> Withdrawal of consent, Early discharge without follow- up at Day 14 Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy <sup>[d]</sup> for non-relevant vasospasm | Proportion of subjects meeting the endpoint as per CEC by planned treatment group. Treatment effect expressed as Relative Risk Reduction and common Odds Ratio (clazosentan vs placebo) from CMH analysis |
| Supplementary Estimand 1 | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Occurrence of clinical deterioration due to DCI, from study drug initiation up to 14 days post-study drug initiation. | Composite strategy: Death, Unevaluable for neurological status and received Rescue therapy <sup>[c]</sup> for relevant vasospasm, Unevaluable for neurological status for vasospasm-related reason, early discharge followed by rehospitalization due to DCI Hypothetical <sup>[a]</sup> : Withdrawal of consent, Early discharge without follow- up at Day 14 Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy <sup>[d]</sup> for non-relevant vasospasm | proportion of subjects meeting the endpoint as per CEC by planned treatment group. Treatment effect expressed as adjusted Odds Ratio (clazosentan vs placebo) from logistic regression. |

| Estimand | Target population | Endpoint | Strategy for addressing intercurrent events | Population-level summary |
|---|---|---|---|---|
| Supplementary Estimand 2 | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Occurrence of clinical deterioration due to DCI, from study drug initiation up to 14 days post-study drug initiation. | Composite strategy: Death, Unevaluable for neurological status and received Rescue therapy <sup>[c]</sup> for relevant vasospasm, Unevaluable for neurological status for vasospasm-related reason, early discharge followed by rehospitalization due to DCI, use of rescue therapy <sup>[d]</sup> for non-relevant vasospasm Hypothetical <sup>[a]</sup> : Withdrawal of consent, Early discharge without follow- up at Day 14 Treatment policy: Permanent/temporary treatment discontinuation | Proportion of subjects meeting the endpoint by planned treatment group. Treatment effect expressed as Relative Risk Reduction and common Odds Ratio (clazosentan vs placebo) from CMH analysis |
| Supplementary Estimand 3 | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Occurrence of death or clinical deterioration due to DCI based on neuroscales only, from study drug initiation up to 14 days post-study drug initiation | Composite strategy: Death Hypothetical <sup>[a]</sup> : Withdrawal of consent, Early discharge without follow- up at day 14 Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy <sup>[d]</sup> for non-relevant vasospasm, Unevaluable for neurological status and received Rescue therapy <sup>[c]</sup> for relevant vasospasm, Unevaluable for neurological status for vasospasm-related reason, early discharge followed by rehospitalization due to DCI | Proportion of subjects meeting the endpoint as per CEC by planned treatment group. Treatment effect expressed as Relative Risk Reduction and common Odds Ratio (clazosentan vs placebo) from CMH analysis |

| Main Secondary Efficacy Endpoint | | | | |
|---|---|---|---|---|
| Main Estimand | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation | Composite strategy: Death Hypothetical <sup>[e]</sup> : Withdrawal of consent Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy | Proportion of subjects meeting the endpoint by planned treatment group. Treatment effect expressed as Relative Risk Reduction and common Odds Ratio (clazosentan vs placebo) from CMH analysis |
| Supplementary Estimand 1 | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Occurrence of<br>clinically relevant<br>cerebral infarction at<br>Day 16 post-study<br>drug initiation | Composite strategy: Death Hypothetical <sup>[e]</sup> : Withdrawal of consent Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy | Proportion of subjects meeting the endpoint by planned treatment group. Treatment effect expressed as adjusted Odds Ratio (clazosentan vs placebo) from logistic regression |

| Supplementary Estimand 2 | Adult subjects with aSAH as defined by the inclusion/exclusion | Occurrence of all-cause cerebral infarction ≥ 5 cm3 at | Composite strategy:<br>Death | Proportion of subjects<br>meeting the endpoint by<br>planned treatment group. |
|---|---|---|---|---|
| | criteria | Day 16 post-study | Hypothetical <sup>[e]</sup> : | Treatment effect expressed as |
| | | drug initiation | Withdrawal of consent | Relative Risk Reduction and common Odds Ratio |
| | | | Treatment policy: | (clazosentan vs placebo) from |
| | | | Permanent/temporary treatment discontinuation, rescue therapy | CMH analysis |
| Other Secondary Efficacy En | Other Secondary Efficacy Endpoint (mRS) | | | |
| Main Estimand | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Long-term clinical outcome assessed by the mRS at Week 12 post-aSAH dichotomized into poor outcome (score ≥ 3) and good outcome (score < 3) | Composite strategy: Death Hypothetical <sup>[b]</sup> : Withdrawal of consent Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy | Proportion of subjects with<br>poor outcome by planned<br>treatment group. Treatment<br>effect expressed as Relative<br>Risk Reduction (clazosentan<br>vs placebo) |

| Other Secondary Efficacy Endpoint (mRS) | | | | |
|---|---|---|---|---|
| Main Estimand | Adult subjects with aSAH as defined by the inclusion/exclusion criteria | Long-term clinical outcome assessed by the GOSE at Week 12 post-aSAH, dichotomized into poor outcome (score ≤ 4) and good outcome (score > 4) | Composite strategy: Death Hypothetical <sup>[b]</sup> : Withdrawal of consent Treatment policy: Permanent/temporary treatment discontinuation, rescue therapy | Proportion of subjects with<br>poor outcome by planned<br>treatment group. Treatment<br>effect expressed as Relative<br>Risk Reduction (clazosentan<br>vs placebo) |

- [a] outcome of the patients after the occurrence of the IE is a medical judgment made by the CEC based on the totality of the data available.
- [b] if the IE occurs then the observed values are replaced by the one imputed according to Section 6.4.1.3 and 6.4.2.3 for mRS and GOSE, respectively.
- [c] protocol-specific rescue therapy as defined in Section 5.4.5.3
- [d] protocol-specific rescue therapy or local rescue therapy as defined in Section 5.4.5.3
- [e] for the first component of the endpoint [see Section 6.3.1] the outcome of the subjects after the occurrence of the IE is a medical judgment made by the CEC based on the totality of the data available. For the subjects not meeting the first component, the second component is imputed according to imputation rules for missing data defined in Section 6.3.3.

aSAH = aneurysmal subarachnoid hemorrhage; CEC = Clinical Event Committee; CMH = Cochran-Mantel-Haenszel; DCI = delayed cerebral ischemia; GOSE = Glasgow Outcome Scale Extended; IE = intercurrent event; mRS = modified Rankin Scale.

score

including subgroups

Doc No D-23.039

# 6.1.3 Overview of primary and secondary efficacy analyses including subgroups Table 6 Overview of primary and secondary efficacy planned analyses,

**Endpoint Analysis** Model Analysis details set Primary efficacy endpoint: Occurrence of clinical deterioration due to DCI from study drug initiation up to 14 days post-study drug initiation FAS Main analysis CMH test stratified by WFNS and age at admission **FAS** Supportive analysis (alternative Logistic regression adjusted for WFNS and model) age at admission FAS CMH test stratified by WFNS and age at Supportive analysis (impact of rescue therapy) admission FAS CMH test stratified by WFNS and age at Supportive analysis (neurological deterioration admission assessed on neuroscales only) **FAS** CMH test stratified by WFNS and age.at Subgroups admission, by subgroup FAS Logistic regression adjusted for WFNS and Subgroups age at admission (treatment by subgroup interaction) Main secondary efficacy endpoint: Occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation. FAS Main analysis CMH test stratified by WFNS and age at admission FAS Logistic regression adjusted for WFNS and Supportive analysis (alternative model) age at admission CMH test stratified by WFNS and age at **FAS** Supportive analysis (initially planned analysis) admission CMH test stratified by WFNS and age.at Subgroups **FAS** admission, by subgroup Subgroups Logistic regression adjusted for WFNS and **FAS** age at admission (subgroup as a factor) Other secondary endpoint: Long-term clinical outcome assessed by the mRS at Week 12 post-aSAH Good vs Main analysis CMH test stratified by WFNS, age at **FAS** admission, and good neurological recovery poor Supportive analysis (alternative **FAS** Good vs Logistic regression adjusted for WFNS, age model) poor at admission, and good neurological Raw **FAS** Supportive analysis (alternative Proportional odds model adjusted for ordinal model) WFNS, age at admission, and good

neurological recovery

| Endpoint | Analysis | Model | Analysis |
|---|---|---|---|
| details | | | set |
| Good vs | Supportive analysis (out-of- | CMH with imputation of out of time window | FAS |
| poor | window assessments) | assessments | |
| Good vs | Subgroups | CMH test stratified by WFNS and age at | FAS |
| poor | | admission | |
| Good vs | Subgroups | Logistic regression adjusted on WFNS and | FAS |
| poor | | age at admission (treatment by subgroup | |
| | | interaction) | |
| Other seco | ndary endpoint: Long-term clinic | al outcome assessed by the GOSE at Week 12 p | ost-aSAH |
| Good vs | Main analysis | CMH test stratified by WFNS, age at | FAS |
| poor | | admission, and good neurological recovery | |
| Good vs | Supportive analysis (alternative | Logistic regression adjusted for WFNS, age | FAS |
| poor | model) | at admission, and good neurological | |
| | | recovery | |
| Raw | Supportive analysis (alternative | Proportional odds model adjusted for | FAS |
| ordinal | model) | WFNS, age at admission, and good | |
| score | | neurological recovery | |
| Good vs | Supportive analysis (out-of- | CMH with imputation of out of time window | FAS |
| poor | window assessments) | assessments | |
| Good vs | Subgroups | CMH test stratified by WFNS and age at | FAS |
| poor | | admission | |
| Good vs | Subgroups | Logistic regression adjusted on WFNS and | FAS |
| poor | | age at admission (treatment by subgroup | |
| | | interaction) | |

aNIHSS = abbreviated National Institutes of Health Stroke Scale; aSAH = aneurysmal subarachnoid hemorrhage, CMH = Cochran-Mantel-Haenszel; CT = computed tomography; DCI = delayed cerebral ischemia; FAS = Full analysis set; GOSE = Glasgow Outcome Scale - Extended; mGCS = modified Glasgow Coma Scale; mRS = modified Rankin Scale; WFNS = World Federation of Neurological Societies.

# 6.2 Primary endpoint

## 6.2.1 Variable

The primary endpoint is the occurrence of clinical deterioration due to DCI from study drug initiation up to 14 days post-study drug initiation.

The Clinical Event Committee (CEC) will indicate for each subject the absence/presence of clinical deterioration due to DCI according to the rules specified in the CEC charter.

During the primary review, the CEC member may answer 'Unknown' if and only if there is a lack of data overall or if poor imaging quality does not allow the assessment on the presence of clinical deterioration or the causality of clinical deterioration to be made with sufficient certainty.
In that case, the primary CEC reviewers will discuss the case and try to come to an agreement during the consensus meeting. If an agreement cannot be reached during the consensus meeting, an adjudication meeting will take place.

The final assessment cannot be 'Unknown'.

#### 6.2.2 Intercurrent events for the main estimand

IEs include death, unevaluable for neurological status and received rescue therapy for relevant vasospasm, unevaluable for neurological status for vasospasms-related reason, and early discharge followed by rehospitalization due to DCI. As these events may reflect the occurrence of a clinical deterioration due to DCI, they will be addressed using a composite strategy, i.e., they will all lead the CEC to conclude (as per CEC charter) that the subject met the primary efficacy endpoint.

The withdrawal of consent and the early discharge without follow-up at day 14 are two IEs precluding further assessment of the neurological status of the subjects. However, they are not systematically associated with the occurrence of clinical deterioration. For instance, subjects in good clinical condition might be discharged early from the intensive care unit (ICU) to free up space for more severe subjects. These IEs will thus be addressed using a hypothetical strategy. The CEC will make a medical judgment based on the totality of the data available up to the time of the occurrence of the IE to determine what would have been the outcome of the subject if neuroscales had been collected up until Day 14.

Use of rescue therapy for a non-relevant vasospasm is part of standard-of-care / current practices. So far, the real efficacy of these rescue therapies has not been demonstrated. They will thus be addressed using a treatment policy strategy.

Permanent/temporary treatment discontinuation will be addressed using a treatment policy strategy.

#### 6.2.3 Handling of missing data

## Subjects randomized and treated

The CEC will provide a final assessment (yes or no) on the primary endpoint, indicating for each subject whether it has been met, therefore it is assumed that there will not be any missing data for the primary endpoint.

There will be no missing data for the stratification variables included in the analysis since these variables are used as stratification factors for the randomization.

#### Subjects randomized but not treated

No further data will be collected for these subjects. They will not be reviewed by the CEC and will be considered as having met the primary endpoint, i.e., the worst possible outcome is assumed.

## 6.2.4 Hypothesis, statistical model and assumptions

The null hypothesis  $(H_0)$  is that the occurrence of clinical deterioration due to DCI in subjects treated with clazosentan is not different from placebo. The alternative hypothesis  $(H_A)$  is that the event rate in the clazosentan group differs from the placebo group.

## 6.2.5 Main analysis

The main analysis for the primary endpoint will be performed on the FAS, according to the intent-to-treat approach.

The observed incidence rates will be displayed together with the exact 95% confidence intervals (CIs) (Clopper-Pearson).

For the main estimand, the null hypothesis will be tested using a CMH test stratified by factors used in the randomization, i.e., WFNS grade (I–II vs III–V) and age ( $\leq 60$  and > 60 years) at admission, at the two-sided significance level of alpha = 0.05.

The treatment effect (clazosentan vs placebo) will be expressed in terms of RRR with corresponding 95% CIs. An RRR greater than 0 will indicate a response to treatment in favor of clazosentan over placebo.

Homogeneity of the treatment effect across strata will be investigated using the Breslow-Day test. Should there be any indication that the odds ratios (ORs) are not homogeneous, emphasis will be given to the within-strata OR rather than the common OR for the interpretation of the treatment effect.

The treatment effect will be described, each with its 95% CL, with:

- The absolute difference in the rates
- The OR
- The RRR

#### **6.2.6** Supportive analyses

#### 6.2.6.1 Logistic regression

As a supplementary estimand, a logistic regression model will be used instead of the CMH test on the FAS.

The primary endpoint is expected to follow a binomial distribution. Accordingly, the treatment effect of clazosentan relative to the placebo will be assessed using a logistic regression adjusted for stratification factors, i.e., hospital admission WFNS grade (I–II vs III–V), and age at hospital admission ( $\leq 60$  and > 60 years).

The generalized linear model used for estimating the treatment effect is:

$$log(p/(1-p)) = \alpha + \beta_1 \times WFNS + \beta_2 \times age + \beta_3 \times treatment$$

where:

- p refers to the probability of the event (i.e., the probability of meeting the endpoint)
- treatment refers to clazosentan and placebo (reference is placebo)
- WFNS refers to hospital admission WFNS grade dichotomized as I–II vs III–V
- age refers to that at hospital admission dichotomized as  $\leq 60$  and > 60 years.

The coefficients  $\alpha$ ,  $\beta_1$ ,  $\beta_2$ , and  $\beta_3$  will be estimated by the method of maximum likelihood.

Treatment effect will be summarized by the OR, the corresponding 95% Wald CI and the p-value derived from the Wald statistic (Type III analysis of effects). Least Squares means for adjusted event rate (probability scale) by treatment group with corresponding 95% CIs will also be computed.

## 6.2.6.2 Rescue therapy for non-relevant vasospasms

A supplementary estimand will evaluate the robustness of the primary analysis with regards to the rescue therapies (i.e., any rescue therapy as defined in Section 5.4.5.3) that may have been given for non-relevant vasospasms. In the main analysis, this IE is addressed using a treatment policy because the efficacy of these medications has not been demonstrated. To assess the robustness of the primary efficacy analysis with regards to rescue therapy given for non-relevant vasospasms, the primary analysis will be repeated but addresses this IE using a composite strategy, i.e., all subjects having received a rescue therapy between study drug initiation and Day 14 will be considered as meeting the primary endpoint.

## 6.2.6.3 Deterioration due to DCI (based on neuroscales only) and death

A supplementary estimand will evaluate the robustness of the primary analysis with regards to the substitution rules defined in the CEC charter to accommodate the situation where a subject was not evaluable and, consequently, the neuroscales were not assessed. The primary analysis will be repeated but considers an alternative definition of the primary endpoint that can only be met following: (i) the occurrence of death or (ii) a clinical deterioration due to DCI based on neuroscales only. Hence, all subjects alive at Day 14 and meeting the primary endpoint according to CEC but without evidence of clinical deterioration based on the neuroscale measurements (i.e., patients having a "Yes" for question 1 "Has the primary endpoint been met?" and a "No" for question 2 "Did the patient have at least one episode of clinical deterioration due to DCI?" of the CEC eCRF) will be considered in this analysis as not meeting the primary endpoint.

#### 6.2.7 Subgroup analyses

The aim of these exploratory subgroup analyses, classifying subjects according to important baseline characteristics, is to explore the consistency of treatment effect in a

variety of relevant subject subgroups to support the efficacy evaluation of clazosentan in this indication.

The following pre-specified subgroups may be considered for the analyses:

- WFNS grade at hospital admission dichotomized as I–II vs III–V
- Age (years) at hospital admission dichotomized as  $\leq 60 \text{ vs} > 60$
- Geographical location (USA vs non-USA; Europe vs non-Europe)
- Race (White; Black or African American; Asian).
- Sex (Female vs Male)
- Type of aneurysm-securing procedure (coiling vs clipping). If both were used, the last one is used for analysis.
- Good neurological recovery (Y/N): subjects who had mGCS ≥ 14 and aNIHSS = 0 prior to study drug start.
- Full neurological recovery (Y/N): subjects who had mGCS = 15 and aNIHSS = 0 prior to study drug start.

Results of the subgroup analyses will be displayed in a table as well as in a forest plot including:

- An estimate of the treatment effect (OR for clazosentan vs placebo) with its 95% CI for each level of each subgroup. It will be calculated using the CMH estimator of the common OR obtained separately in each subgroup level (i.e., including the subgroup and its complementary) as described for the main analysis. When a subgroup is defined by a stratification variable the corresponding stratification variable will be excluded from the analysis.
- A vertical reference line displayed at the level of the overall treatment effect.

The subgroup analyses will also be performed using a logistic regression model stratified by hospital admission WFNS grade (I–II vs III–V), and age at hospital admission ( $\leq 60$  and > 60 years) and including terms for 'subgroup', 'treatment' and 'treatment by subgroup' interaction. Results will be summarized in a table and will include:

- An estimate of the treatment effect (OR for clazosentan vs placebo) with its 95% CI for each level of each subgroup (i.e., including the subgroup and its complementary)
- A p-value for the interaction tests

Additional subgroup analyses for the primary endpoint may also be conducted for factors that are identified with a statistically significant treatment × factor interaction.

The study is not designed or powered to detect interactions, but an arbitrary two-sided significance level of alpha = 0.10 will be used for the interpretation of the interaction test. No multiplicity adjustment is introduced as the subgroup analyses are exploratory in nature.

If there are issues due to very small sample sizes (e.g., interaction test failing due to presence of observed zero cells), the use of other methods may be considered.

## 6.2.8 Other analyses

If the FAS and the RND populations differ by more than 5%, then the main analysis will be repeated on the RND.

The initially planned analysis of the primary endpoint (up to protocol version 6 dated 29 April 2021) will be performed as an exploratory analysis. It will consist of repeating the primary analysis defined in Section 6.2.5 but stratified by all the factors used in the randomization, i.e., WFNS grade, age at admission, and patient population (high-risk prevention vs early treatment) at the two-sided significance level of alpha = 0.05.

Number of episodes of clinical deterioration due to DCI from study drug initiation and up to 14 days post-study drug initiation as adjudicated by the CEC will be summarized with descriptive statistics for categorical variables (from 1 up to the highest number of episodes observed) by treatment group on the FAS.

If subjects were treated accidently, at least partially, during the study with a treatment different from the one they were randomized to, the main analysis will be repeated using the actual treatment group instead of the planned treatment group, i.e., the main analysis will be repeated on the SAF.

One listing will be produced displaying both scores (mGCS and aNIHSS), the date and time of the assessment, and the day relative to study drug initiation.

One listing will present the date and time of each cerebral angiogram and cerebral computed tomography (CT) scan performed over the course of the study.

Selected information from data collected on the 'Episode of clinical deterioration' eCRF page, in the IRC Review eCRF and IRC Adjudication eCRF will be displayed in listings. Selected information from data collected in the CEC eCRF will also be displayed in listings.

# 6.3 Main secondary endpoint

#### 6.3.1 Variable

The main secondary endpoint is the occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation as defined by the two following components:

- Component 1: all-cause cerebral infarction  $\geq 5$  cm<sup>3</sup>. This will be evaluated (yes/no) for all subjects by IRC and will be confirmed by the CEC
- Component 2: for all subjects with a "no" at component 1, then the presence of cerebral infarction < 5 cm³ (as assessed by IRC) will be evaluated in subjects with clinical deterioration due to DCI (as assessed by the CEC)

Cerebral infarction refers to new or worsened infarcts and is determined by central radiology review comparing the total volume of infarcts on the CT scan performed 16 days after study drug initiation with the total volume on the CT scan performed post-procedure. If the CT scan cannot be performed on Day 16, then it is acceptable for the CT to be performed within the 7 days following Day 16. If a subject is discharged from the hospital prior to Day 16, the CT scan is performed on the day of hospital discharge. Clinical deterioration due to DCI and cerebral infarctions  $\geq 5$  cm<sup>3</sup> are confirmed by the CEC. Cerebral infarctions  $\leq 5$  cm<sup>3</sup> in subjects with clinical deterioration due to DCI are derived from both the CEC data (primary endpoint) and IRC data (for infarct size).

#### 6.3.2 Intercurrent events for the main estimand

Similar to that stated for the primary endpoint regarding death and DCI, the occurrence of death prior to Day 16 may be related to cerebral infarction. Consequently, the occurrence of death will be addressed using a composite strategy, i.e., all subjects who died will be considered as meeting the main secondary endpoint.

The withdrawal of consent before Day 16 is an IE precluding the carrying out of the Day 16 CT scan. The first component of the endpoint withdrawal of consent will be addressed using a hypothetical strategy where the CEC will make a medical judgment based on the totality of the data available up to the time of consent withdrawal to determine what would have been the outcome of the subject if the Day 16 CT scan would have been available. For all subjects who (i) withdrew consent, (ii) met the primary endpoint, and (iii) do not meet the first component of the main secondary endpoint, then the second component of the main secondary endpoint cannot be derived if the Day 16 CT scan is missing. These subjects will thus be considered as meeting the main secondary endpoint (according to imputation rule for missing data defined in Section 6.3.3).

Use of rescue therapy as defined in this study are part of standard-of-care / current practices. So far, the real efficacy of these therapies/medications has not been demonstrated. Therefore, they will be addressed using a treatment policy strategy.

Permanent/temporary treatment discontinuation will be addressed using a treatment policy strategy.

## 6.3.3 Handling of missing data

## Subjects randomized and treated

The CEC will provide a final assessment (yes/no) on the first component of the main secondary endpoint, indicating for each subject whether it has been met. Therefore, it is assumed that there will not be any missing data for this component. However, patients not meeting the first component of the endpoint may have a missing Day 16 CT scan (no CT scan performed 14 days after study drug start or later) preventing the assessment of the second component of the endpoint. If the second component of the endpoint cannot be derived, then the subjects meeting the primary endpoint will be considered as meeting the

main secondary endpoint, i.e., the worst possible outcome is assumed. As per protocol, if a subject is discharged before Day 16 but not earlier than Day 14, the "Day 16 CT scan" can be done on the day of discharge. It follows that "Day 16 CT scan" will be considered missing for the evaluation of the second component of the endpoint when there is no CT scan performed 14 days after study drug start or later.

There will be no missing data for the variables included in the model since these variables are collected as stratification factors for the randomization.

## Subjects randomized and not treated

No further data will be collected for these subjects. They will not be reviewed by the CEC and will be considered to have met the primary endpoint [see Section 6.2.3] and the main secondary endpoint, i.e., the worst possible outcome is assumed.

## 6.3.4 Hypothesis, statistical model and assumptions

The null hypothesis  $(H_0)$  is that the occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation in subjects treated with clazosentan is not different from placebo. The alternative hypothesis  $(H_A)$  is that the event rate in the clazosentan group differs from the placebo group.

## 6.3.5 Main analysis

The proportion of subjects with occurrence of clinically relevant cerebral infarction at Day 16 post-study drug initiation will be analyzed in a similar manner as the primary efficacy endpoint [see Section 6.2.5 for details].

The main statistical analysis for the main secondary endpoint will be performed on the FAS according to the intent-to-treat approach.

The null hypothesis will be tested using a CMH test stratified by factors used in the randomization, i.e., WFNS grade and age at admission, at the two-sided significance level of alpha = 0.05.

## **6.3.6** Supportive analyses

## Logistic regression

As a supplementary estimand, a logistic regression model will be used on the FAS instead of the CMH test following the same approach as the one considered for the supportive analysis of the primary endpoint described in Section 6.2.6.1.

#### 6.3.7 Subgroup analyses

Exploratory subgroup analyses may be conducted using the same approach and on the same subgroups as the ones defined for the primary endpoint analysis described in Section 6.2.7.

The study is not designed or powered to detect interactions, but an arbitrary two-sided significance level of alpha = 0.10 will be used to interpret the interaction test. No multiplicity adjustment is introduced as the subgroup analyses are exploratory in nature.

If there are issues due to very small sample sizes (e.g., interaction test failing due to presence of observed zero cells), the use of other methods may be considered.

## 6.3.8 Other analyses

If the FAS and the RND populations differ by more than 5%, then the main analysis will be repeated on the RND.

The initially planned primary analysis of the main secondary endpoint (up to protocol version 6 dated 29 April 2021) will be performed as an exploratory analysis. It will consist of repeating the primary analysis defined in Section 6.3.5 on the first component only of the endpoint as defined in Section 6.3.1. For this analysis the CMH will be stratified by all the factors used in the randomization, i.e., WFNS grade at hospital admission (I–II vs III–V), age ( $\leq 60$  and > 60 years) at hospital admission, and patient population (high-risk prevention vs early treatment) at the two-sided significance level of alpha = 0.05.

If subjects were treated accidently, at least partially, during the study with a treatment different from the one they were randomized to, the main analysis will be repeated using the actual treatment group instead of the planned treatment group, i.e., the main analysis will be repeated on the SAF.

Listings will be produced on the RND displaying all the data collected in the IRC Review eCRF (e.g., common findings, clot size, vasospasm severity, reviewer's comment, total infarct volume on post-procedure CT scan, total infarct volume on Day 16 CT scan, volume of new and worsened infarcts on Day 16 CT scan).

## 6.4 Other secondary endpoint

The other secondary endpoint is long-term clinical outcome assessed by the mRS and the GOSE at Week 12 post-aSAH. The structured interview for the GOSE allows for simultaneous derivation of the mRS.

#### 6.4.1 Modified Rankin Scale

#### 6.4.1.1 Variable

The raw mRS scores range from 0 (no symptoms) to 6 (dead) and will be dichotomized for analysis into poor (a score of 3 to 6) vs good (a score of 0 to 2) outcome.

#### 6.4.1.2 Intercurrent events for the main estimand

Deaths are included in the mRS. Therefore, the occurrence of death will be addressed using a composite strategy where all subjects that died prior to Week12 (i.e., died prior to day 84 + 21 days post-aSAH) will have a mRS score of 6 irrespective of whether a prior assessment was available.

The withdrawal of consent before the collection of the mRS assessment (Week 12) will be addressed using a hypothetical scenario. The final outcome for the subject will be derived based on the mGCS data collected up to the time of consent withdrawal as per the imputation rule for missing data defined in Section 6.4.1.3.

Use of rescue therapy as defined in this study are part of standard-of-care / current practices. So far, the real efficacy of these therapies/medications has not been demonstrated. Therefore, they will be addressed using a treatment policy strategy.

Permanent/temporary treatment discontinuation and out-of-window assessments will be addressed using a treatment policy strategy.

# 6.4.1.3 Handling of missing data

## Subjects randomized and treated

If the mRS score from the Week 12 interview is missing, and the subject did not die prior to Week 12 (i.e., did not die prior to day 84 + 21 days post-aSAH), the missing mRS score is replaced by the score 4 (moderately severe disability) with the following exception:

• If the patient had their mGCS score reported at least once per day, from the study drug initiation up to 14 days post-study drug initiation (or up to the time of discharge if subject is discharged before Day 14 but after having completed study treatment as per protocol), and all reported scores, regardless of day and time point, are ≥ 14 and the location where the subject was discharged after the initial hospitalization at the investigational study center is home, then the missing mRS is substituted with 2 (slight disability).

#### Subjects randomized but not treated

If the subject is still alive at the time they withdraw from study, a missing mRS score will be replaced by the score 4 (moderately severe disability).

#### 6.4.1.4 Hypothesis, statistical model and assumptions

The null hypothesis  $(H_0)$  is that the proportion of subjects with poor clinical outcomes treated with clazosentan is not different from the placebo group. The alternative hypothesis  $(H_A)$  is that the event rate in the clazosentan group differs from the placebo group.

#### 6.4.1.5 Main analysis

The proportion of subjects for each possible score value will be summarized in a table and in a figure by treatment group on the FAS.

The proportion of subjects with poor (a score of 3 to 6) clinical outcomes (mRS) at Week 12 post-aSAH will be analyzed in a similar manner as the primary efficacy endpoint [see Section 6.2.5 for details] but adding the good neurological recovery (mGCS  $\geq$  14 and aNIHSS = 0, Yes/No) variable as an adjustment variable.

All available assessments (including out-of-window ones) will be used in the analysis.

## 6.4.1.6 Supportive/sensitivity analyses

## 6.4.1.6.1 Out-of-window assessments

The main analysis will be repeated but replacing the assessments outside of the  $84 \pm 21$  days post-aSAH time window by imputed ones according to the imputation rule for missing data defined in Section 6.4.1.3.

# 6.4.1.6.2 Logistic regression

This analysis relies on a logistic regression model on the FAS instead of the CMH test. The same approach as the one considered for the supportive analysis of the primary endpoint described in Section 6.2.6.1 will be used but adding the good neurological recovery (mGCS  $\geq$  14 and aNIHSS = 0, Yes/No) variable as an adjustment variable.

## 6.4.1.6.3 Proportional odds regression model

A proportional odds model (POM) adjusted on WFNS grade (I–II vs III–V), age ( $\leq 60$  and > 60 years) at admission and good neurological recovery (mGCS  $\geq 14$  and aNIHSS = 0, Yes/No) will be used as a supportive analysis to assess treatment effect on raw mRS data (i.e., on ordinal score) on the FAS. Results of the POM will be presented by the OR, the corresponding 95% Wald CL, and the p-value derived from the Wald statistic (type III analysis of effects). The validity of the proportional odds assumption will be assessed by fitting a fully non-proportional odds model. Departure from the proportional odds assumption will be evaluated on the forest plot displaying the departure of all individual slopes (and associated p-values) compared to the reference slope for each effect. If the proportional odds assumption is not satisfied for some variables, then partially proportional odds models could be considered to estimate and test treatment effect.

## 6.4.1.7 Subgroup analyses

The main analysis will be repeated on the following pre-defined subgroups (and corresponding complementary subgroups) but without adjusting for good neurological recovery:

- Good neurological recovery: subjects who had mGCS ≥ 14 and aNIHSS = 0 prior to study drug start.
- Full neurological recovery: subjects who had mGCS = 15 and aNIHSS = 0 prior to study drug start.

Additional exploratory subgroup analyses may also be conducted with the same approach as the one defined for the primary endpoint in Section 6.2.7.

## 6.4.1.8 Other analyses

If the FAS and the RAND populations differ by more than 5%, then the main analysis will be repeated on the RND analysis set.

## Listings

One listing will be produced displaying both scores (GOSE and mRS), the date and time of the assessment, the number of days elapsed since aSAH, and the respondent's identity (subject and/or proxy and/or legal representative).

### **Figures**

For the GOSE and mRS, the distribution of subjects for each level will be provided in a graphical format.

## 6.4.2 Glasgow Outcome Scale – Extended

#### 6.4.2.1 Variable

The raw GOSE scores range from 1 (dead) to 8 (upper good recovery) and will be dichotomized for analysis into poor outcome (score  $\leq 4$ ) and good outcome (score  $\geq 4$ ).

#### 6.4.2.2 Intercurrent events for the main estimand

Death is included in the GOSE. Therefore, occurrence of death will be addressed using a composite strategy where all subjects that died prior to Week 12 (i.e., died prior to day 84 + 21 days post-aSAH) will have a GOSE score of 1 irrespective of whether a prior assessment was available.

The withdrawal of consent before the collection of the GOSE assessment (Week 12) will be addressed using a hypothetical scenario. The final outcome for the subject will be derived based on the mGCS data collected up to the time of consent withdrawal as per the imputation rule for missing data defined in Section 6.4.2.3.

Use of rescue therapy as they are defined in this study are part of standard-of-care / current practices. So far, the real efficacy of these therapies/medications has not been demonstrated. Therefore, they will be addressed using a treatment policy strategy.

Permanent/temporary treatment discontinuation will be addressed using a treatment policy strategy.

#### 6.4.2.3 Handling of missing data

## Subjects randomized and treated

If the GOSE score from the Week 12 interview is missing, and the subject did not die prior to Week 12 (i.e., did not die prior to day 84 + 21 days post-aSAH), the missing GOSE score is replaced by the score 3 (lower severe disability), with the following exception:

• If the subject had their mGCS score reported at least once per day, from study drug initiation up to 14 days post-study drug initiation (or up to the time of discharge if subject is discharged before Day 14 but after having completed study treatment as per protocol), and all reported scores regardless of day and time point are ≥ 14, and the location where the subject was discharged after the initial hospitalization at the

investigational study center is home, then the missing GOSE is substituted with 5 (lower moderate disability).

## Subjects randomized but not treated

If the subject is still alive at the time they withdraw from study, a missing GOSE score will be replaced by the score 3 (lower severe disability).

## 6.4.2.4 Hypothesis, statistical model and assumptions

The null hypothesis  $(H_0)$  is that the proportion of subjects with poor clinical outcome treated with clazosentan is not different from placebo. The alternative hypothesis  $(H_A)$  is that the event rate in the clazosentan group differs from the placebo group.

## 6.4.2.5 Main analysis

The proportion of subjects for each possible score value will be summarized in a table and in a figure by treatment group on the FAS.

The proportion of subjects with poor (a score of 1 to 4) clinical outcome (GOSE) at Week 12 post-aSAH will be analyzed in a similar manner as for the primary efficacy endpoint [see Section 6.2.5 for details] but adding the good neurological recovery (mGCS  $\geq$  14 and aNIHSS = 0, Yes/No) variable as an adjustment variable.

All available assessments (including those performed out-of-window) will be used in the analysis.

#### 6.4.2.6 Supportive/sensitivity analyses

## 6.4.2.6.1 Out-of-window assessments

The main analysis will be repeated but replacing the assessments outside of the  $84 \pm 21$  days post-aSAH time window by imputed ones according to the imputation rule for missing data defined in Section 6.4.2.3.

#### 6.4.2.6.2 Logistic regression

This analysis relies on a logistic regression model on the FAS instead of the CMH test. The same approach as the one considered for the supportive analysis of the primary endpoint described in Section 6.2.6.1 will be used but adding the good neurological recovery (mGCS  $\geq$  14 and aNIHSS = 0, Yes/No) variable as an adjustment variable.

#### 6.4.2.6.3 Proportional odds regression model

A POM adjusted on WFNS grade (I–II vs III–V), age ( $\leq 60$  and > 60 years) at admission and good neurological recovery (mGCS  $\geq 14$  and aNIHSS = 0, Yes/No) will be used as a supportive analysis to assess treatment effect on raw GOSE data (i.e., on ordinal score) on the FAS. Results of the POM will be presented by the OR, the corresponding 95% Wald CL, and the p-value derived from the Wald statistic (type III analysis of effects). The validity of the proportional odds assumption will be assessed by fitting a fully non-

proportional odds model. Departure from the proportional odds assumption will be evaluated on the forest plot displaying the departure of all individual slopes (and associated p-values) compared to the reference slope for each effect. If the proportional odds assumption is not satisfied for some variables, then partially proportional odds models would be considered to estimate and test treatment effect.

## 6.4.2.7 Subgroup analyses

The main analysis will be repeated on the following pre-defined subgroups (and their corresponding complementary) but without adjusting for good neurological recovery:

- Good neurological recovery: subjects who had mGCS ≥ 14 and aNIHSS = 0 prior to study drug start.
- Full neurological recovery: subjects who had mGCS = 15 and aNIHSS = 0 prior to study drug start.

Additional exploratory subgroup analyses may also be conducted with the same approach as the one defined for the primary endpoint on subgroups including but not limited to the ones defined in Section 6.2.7.

## 6.4.2.8 Other analyses

If the FAS and the RND populations differ by more than 5%, then the main analysis will be repeated on the RND.

#### Listings

One listing will be produced displaying both scores (GOSE and mRS), the date and time of the assessment, the number of days elapsed since aSAH, and the respondent's identity (subject and/or proxy and/or legal representative).

#### **Figures**

For the GOSE and mRS, the distribution of subjects for each level will be provided in a graphical format: one bar per treatment group and per variable, where each bar shows 100% of the discrete value.

## 6.5 Subject-reported endpoints

The analysis of the effect of clazosentan on long-term clinical outcome, cognition, and health-related QoL at Week 12 post-aSAH will be described together as described in this section.

To evaluate the effect of clazosentan on cognition, the following endpoints will be used:

Cognitive status, as assessed by the change from baseline to Day 14 post-study drug
initiation on the Montreal Cognitive Assessment (MoCA), for those subjects that have
a score at both time points

- Cognitive status, as assessed by the change from baseline to Week 12 post-aSAH on the MoCA, for those subjects that have a score at both time points
- Cognitive status, as assessed by the change from Day 14 post-study drug initiation to Week 12 post-aSAH on the MoCA, for those subjects that have a score at both time points
- Cognitive status as assessed by the MoCA at Day 14 post-study drug initiation and at Week 12 post-aSAH

To evaluate the effect of clazosentan on health-related QoL post-aSAH, the following endpoints will be used:

- Generic QoL as measured by the EQ-5D-5L at Week 12 and Week 24 post-aSAH
- Oxford Participation and Activities Questionnaire (Ox-PAQ) at Week 12 post-aSAH
- Disease-specific QoL as measured by the Stroke-Specific Quality of Life (SS-QoL) at Week 12 post-aSAH

## **6.5.1** Montreal Cognitive Assessment

#### 6.5.1.1 Variables

The MoCA will be used to detect cognitive impairment. The variables that will be analyzed are:

- The value at each assessment for the domain scores and the total score.
- The change from baseline to each post-treatment visit (i.e., Day 14 post-study drug initiation and Week 12) for the domains scores and the total score.
- The change from Day 14 post-study drug initiation to Week 12 for the domains scores and the total score.

If the assessment for one domain is missing, the total score is not computed. All assessments performed after Day 14 will be analyzed as Week 12 assessments.

## **6.5.1.2** Analysis

The tables, figures and listings will be produced on the FAS.

#### **Tables**

Descriptive statistics for both domain scores and the total score will be computed by treatment group on the FAS for:

- change from baseline to each visit and the corresponding actual values at each visit
- change from Day 14 post-study drug initiation to Week 12 post-aSAH and the corresponding actual values at Day 14 post-study drug initiation and at Week 12 postaSAH
- actual values at each visit (including subjects having missing values at any visit)

A table with descriptive statistics (number and percentage of subjects) on the reason for not performing the test will also be produced.

Treatment effect in MoCA total score will be assessed using a mixed model for repeated measures for the actual values at each post-baseline visit (i.e., Day 14 post-study drug initiation and Week 12) using an unstructured variance/covariance matrix and the following covariates: WFNS grade (I–II vs III–V) at admission, age (≤ 60 and > 60 years) at admission, visit (as a factor), treatment group, and visit by treatment interaction. Least Squares means and 95% CI will be computed for each treatment group and visit and for the between-group difference at each visit.

In addition, changes from baseline to post-baseline visits will be analyzed using the same mixed model but with an additional covariate for baseline MoCA total score. Treatment effect in MoCA total score will also be assessed using an analysis of variance (ANOVA) fitted on change from Day 14 post-study drug initiation to Week 12 and including the following covariates: WFNS grade (I–II vs III–V) at admission, age ( $\leq$  60 and > 60 years) at admission, Day 14 MoCA total score, and treatment group. This treatment effect estimate could have been derived from the mixed model for repeated measures on the change from baseline to post-baseline visits defined above but because of the missing baseline values this analysis should provide a more precise estimate of the change from Day 14 to Week 12.

Additional analyses may also be conducted using the same approaches on pre-defined subsets such as:

- Good neurological recovery: subjects who had mGCS ≥ 14 and aNIHSS = 0 prior to study drug start.
- Full neurological recovery: subjects who had mGCS = 15 and aNIHSS = 0 prior to study drug start.

#### **Figures**

The evolution of the total score over time will be provided in a graphical format from baseline to Week 12 (one boxplot per treatment group and analysis visit).

## Listings

A listing will provide date and time of assessment, the reason for not performing the MoCA, the total score at each visit, the absolute change from baseline to each post-baseline visit in total score and the change from Day 14 post-study drug initiation to Week 12 post-aSAH in total score. The values taken into account for the analysis will be flagged. It will also include the day relative to study drug initiation and the number of days elapsed since aSAH.

#### 6.5.2 EQ-5D-5L

#### 6.5.2.1 Variables

The EQ-5D (5L version) questionnaire will be used at Week 12 and Week 24 post-aSAH to assess the subject's QoL. The variables that will be analyzed are:

- To characterize an EQ-5D **health state**: The responses of the 5 dimensions combined ranging from (full health) to (worst health)
- To characterize the **health utility**: The EQ-5D health state converted into a single summary index value and continuous value ranging from 0 to 1 (value less than 0 represent health states regarded as worse than death) using a crosswalk link function. Following the latest guidance of the NICE published in 2022, the value set provided by Hernández Alava et al. [Hernández-Alava 2017] for the UK will be used to derive the health utility score
- To characterize the **overall self-rated health status**: The value of the visual analog scale (VAS) score, ranging from 0 (worst imaginable health) to 100 (best imaginable health)

All assessments performed before Day 126 (midpoint between Week 12 and Week 24) will be analyzed as Week 12 assessments and all those performed after will be analyzed as Week 24 assessments. If a subject has two assessments allocated to the same week then only the last assessment will be used for analysis.

#### **6.5.2.2** Analysis

The tables, figures and listing will be produced on the FAS.

## **Tables**

The health state and corresponding respondent (e.g., subject, proxy) will be summarized by visit and treatment group, using descriptive statistics for categorical and continuous data. The health utility and VAS will be summarized by visit and treatment group, using descriptive statistics for continuous data.

Change from Week 12 to Week 24 in health utility and VAS will be summarized by treatment group, using descriptive statistics for continuous data.

For the health state, between-group comparison domain by domain will be performed using a POM (unadjusted). It will provide the OR and corresponding 95% CI (normal approximation) for each domain.

For the overall health status (VAS score) and the health utility, between-group comparisons at Week 12 and Week 24 will be performed using ANOVAs with factors for WFNS grade (I–II vs III–V) at admission, age (≤ 60 and > 60 years) at admission, and treatment group. Least Squares means and 95% CLs will be computed for each treatment group and for the difference between clazosentan and placebo groups. Between-group comparison of the

change from Week 12 to Week 24 will be done using the same model but adding the assessment at Week 12 as an adjustment variable.

If the assumptions underlying the ANOVA model (normality of the residuals, homogeneity of the variance) are not fulfilled, the same comparisons between treatment groups will also be performed by means of a non-parametric one-way ANOVA (Wilcoxon-Mann-Whitney test).

## Figures

For each domain, the distribution of subjects in each level will be provided in a graphical format.

For the VAS score, the distribution will also be provided in a graphical format: one histogram per treatment group.

For the utility index, the distribution will also be provided in a graphical format: one histogram per treatment group.

All the figures will be provided for both Week 12 and Week 24.

### Listings

One listing will be produced displaying the health profile (the value for each domain), health status (VAS score) and index value. It will also include the number of days elapsed since aSAH.

#### 6.5.3 Ox-PAO

#### 6.5.3.1 Variables

The Ox-PAQ at Week 12 post-aSAH will be used to assess health-related QoL and in particular to assess participation, activities, and level of independence. The variables that will be analyzed are:

- The value for each item, ranging from 0 (never) to 4 (always)
- The raw score for each domain, calculated as the sum of the scores for the items in that domain
  - Routine activities (14 items):
  - Emotional well-being (5 items):
  - Social engagement (4 items):
- The re-scaled score **for each domain**, ranging from 0 to 100, calculated according to the following formula:
- 100 × raw score / maximum score

The missing data will be imputed as recommended in the Ox-PAQ manual. If a single item within any domain is unanswered it is considered reasonable to impute the mean value representing all of the respondent's other item responses (the series mean) within that

domain to the missing item. If two or more questions on any domain are unanswered, the overall score for that domain/respondent should not be calculated.

## 6.5.3.2 Analysis

The tables, figures and listings will be produced on the FAS.

#### **Tables**

Descriptive statistics on the raw and re-scaled scores will be presented by domain and treatment group. The table will also include descriptive statistics (number and percentage of subjects) on missing data (imputed, missing).

Between-group comparison (clazosentan vs placebo) will be performed for each domain on the transformed score by means of ANOVAs with factors for WFNS grade (I–II vs III–V) at admission, age ( $\leq$  60 and > 60 years) at admission and treatment group. Least Squares means and 95% CLs will be computed for each treatment group and for the difference between clazosentan and placebo groups.

If the assumptions underlying the ANOVA model (normality of the residuals, homogeneity of the variance) are not fulfilled, the same comparison between treatment groups will also be performed by means of a non-parametric one-way ANOVA (Wilcoxon-Mann-Whitney test).

## **Figures**

For each domain score, the distribution/dispersion of the values will be displayed as boxplots: one figure per score and one boxplot per treatment group.

#### Listings

A listing will provide the raw score for each of the 3 domains together with the transformed scores. It will also include the number of days elapsed since aSAH.

## 6.5.4 Stroke-Specific Quality of Life

#### 6.5.4.1 Variables

The SS-QoL [Williams 1999] is evaluated at Week 12 post-aSAH to measure health-related QoL specific to patients with stroke. For the first part of the questionnaire (49 items), the following scores will be computed:

Domain scores, computed
 Total score, computed
 Physical component, computed
 Psychosocial component, compute

Missing items are handled in the following way: if more than half of the items in a given domain are missing, that domain is not scored and the resulting overall SS-QoL score is an average of the remaining domain scores. If fewer than half of the items in a given domain are missing, the scored items are averaged and rounded to the nearest integer. This imputed item score is then substituted for the missing item(s).

Overall SS-QoL score is an unweighted average of domain scores and ranges from 1.0 (worst) to 5.0 (best).

For the second part of the questionnaire collecting information regarding patient status prior to aSAH, the following scores are used:

- Domain scores,
- Total score,

No imputation for missing data will be performed.

## 6.5.4.2 Analysis

The tables, figures and listings will be produced on the FAS.

#### **Tables**

For the first part of the questionnaire, descriptive statistics for each computed score will be presented by treatment group on the FAS. The table will also include descriptive statistics (number and percentage of subjects) on missing data (imputed, missing).

Between-group comparison (clazosentan vs placebo) will be performed for each domain and on the total score by means of ANOVAs with factors for WFNS grade (I–II vs III–V) at admission, age (≤ 60 and > 60 years) at admission and treatment group. Least Squares means and 95% CLs will be computed for each treatment group and for the difference between clazosentan and placebo groups.

If the assumptions underlying the ANOVA model (normality of the residuals, homogeneity of the variance) are not fulfilled, the same comparisons between treatment groups will also be performed by means of a non-parametric one-way ANOVA (Wilcoxon-Mann-Whitney test).

The variables collected in the second part of the questionnaire will be summarized using descriptive statistics for categorical variables by treatment groups on the FAS.

#### **Figures**

In the first part of the questionnaire, the distribution/dispersion of the values will be provided by means of boxplots for each computed score: one figure per score and one boxplot per treatment group.

In the second part of the questionnaire, a bar plot will be produced by variable and treatment group displaying the proportions of subjects for each category.

## Listings

A listing will be produced to display all computed scores. A second listing will provide the answers to the second part of the questionnaire and related reported scores. It will also include the number of days elapsed since aSAH.

# 6.6 Multivariate long-term outcome

#### 6.6.1 Variables

The long-term clinical outcome of the patients will be evaluated by jointly analyzing the following variables:

- GOSE total score at Week 12
- mRS total score at Week 12
- EQ-5D utility value at Week 12
- EQ-5D utility value at Week 24
- Ox-PAO raw domain scores at Week 12
- SS-QoL total score at Week 12
- MoCA at Week 12
- Change from baseline to Week 12 in MoCA

#### 6.6.2 Analysis

All Week 12 assessments will be analyzed jointly using a normed Principal Component Analysis (PCA). This analysis will be done in R [R Core Team 2020] using the function "dudi.pca" of the R-package 'ade4" [Chessel 2004]. As the PCA requires complete cases, subjects with at least one missing value will be excluded from the analysis. The treatment effect will be characterized using a between-class analysis [Dolédec 1987] and tested using a permutation test [Romesburg 1985] at the two-sided significance level of alpha = 0.05 on the between-groups inertia (i.e., multi-dimensional between-treatment group variance) percentage. This analysis will be repeated but imputing missing assessment with the observed overall mean of the corresponding variable. The analysis might also be repeated excluding the variables with the highest frequencies of missing values and/or including change from baseline to Week 12 in MoCA and Week 24 assessment of EQ-5D.

The following outputs will be produced:

- Distribution of the eigen values of the PCA
- Contribution of the variables to the principal components of the PCA
- Factorial maps of the PCA
- Factorial maps of the between-class analysis
- Permutation test on the between-group inertia percentage

# 6.7 Analysis of pharmaco-economic variables

The tables, figures and listings will be produced on the FAS.

- Number and type of episodes of rescue therapy, from randomization up to hospital discharge and from hospital discharge up to Week 12 [see Section 5.4.5.3]
- Number and type of specific (pre-specified) medical treatments and therapies from randomization up to hospital discharge and from hospital discharge up to Week 12 [see Section 5.4.5.2]
- Length (in days) of initial and total ICU stay, length (in days) of total hospitalization, and duration (in days) in different hospital care units, from randomization up to hospital discharge and from hospital discharge until Week 12
- Intensity of rehabilitation care up to Week 12 post-aSAH
- First post-hospital discharge location
- Duration (in days) of home care support post-initial hospital discharge
- Employment status at Week 24 (6 months) post-aSAH

## 6.7.1 Rescue therapies

See Section 5.4.5.3 for details.

## 6.7.2 Specific (pre-specified) medical treatments and therapies

See Section 5.4.5.2 for details.

#### 6.7.3 Subject location/rehabilitation

#### 6.7.3.1 Variables

For each subject, the following variables will be derived:

- Length of initial ICU stay, defined as the time (days) elapsed between date of start/admission and date of end/discharge when location is recorded as 'Critical care unit or equivalent' (earliest record)
- Length of total ICU stay, defined as the sum of the lengths (days) of each stay recorded as 'Critical care unit or equivalent'
- Length of total hospitalization (in days), defined as the sum of the lengths of each stay recorded as 'Critical care unit or equivalent' or 'Specialized care ward' or 'General care ward'
- Length of stay in 'Specialized care ward' defined as the total time (days) elapsed between date of start/admission and date of end/discharge for each location recorded as 'Specialized care ward'
- Length of stay in 'General care ward' defined as the total time (days) elapsed between date of start/admission and date of end/discharge for each location recorded as 'General care ward'
- Intensity of rehabilitation care up to Week 12 post-aSAH, defined as the cumulative number of hours in each category (none, light, moderate, intense)

- Post-hospital discharge location, defined as the first location the subject is admitted to other than 'Critical care unit or equivalent' or 'Specialized care ward' or 'General care ward'
- Duration (days) of home care support post-hospital discharge, defined as the sum of the lengths of each stay in 'Inpatient rehabilitation facility' and 'Assisted living facility' or 'Home partially independent'

Other locations recorded as a free text will not be taken into account for the computation of any of these durations.

Duration in hours (for the intensity of rehabilitation care) will be derived by multiplying the duration of the rehabilitation in weeks by the mid class of rehabilitation intensity: 3.5, 10.5, 17.5 hours per week.

To compute duration in the event of a missing end date, when the question 'Ongoing at end of study' was ticked in the eCRF then the missing end date should be imputed with EOS date.

### **6.7.3.2** Analysis

Descriptive statistics will be provided for each of the aforementioned variables by treatment group.

A first listing will present the inpatient and outpatient locations (e.g., critical care unit or equivalent, specialized care ward, nursing facility) with corresponding date (time) of start/admission and date (time) of end/discharge as well as the various lengths of stay.

A second listing will present the intensity of the rehabilitation course and the corresponding start and end date as well as the corresponding duration.

## 6.7.4 Employment status

#### 6.7.4.1 Assessments

At Week 24 post-aSAH, the pre-aSAH employment/student status, the current employment/student status, and the date of return to work (or to an educational institution, for students, as applicable) will be collected via telephone or postal questionnaire and captured in the clinical database.

The employment status is collected as follows:

- Employed full time
- Employed part time
- Student full time
- Student part time
- On work disability
- Homemaker

- Retired
- Not employed
- Unknown

For both time points (pre-aSAH and Week 24 post-aSAH), the subject may select multiple possibilities.

#### 6.7.4.2 Variables

The following variables will be derived:

- The employment status at the given time point (including the reported combinations (e.g., Student part time/ Employed part time)
- The time (days) from aSAH to return to work, the time (days) from aSAH to return to education
- The change from pre- to post-aSAH status (fully back to pre-aSAH, partially back to pre-aSAH, not back to pre-aSAH) defined as the worst observed transition (see transition matrix in Appendix 14.3) between pre-aSAH and post-aSAH status.

## **6.7.4.3** Analysis

Tables and listings will be produced on the FAS.

A table will provide the number and percentage of subjects in each category (and reported combinations) by treatment group for each time point.

A table will provide the number and percentage of subjects in each category of change from pre- to post-aSAH status (fully back, partially back, not back) by treatment group with 95% Clopper-Pearson CI.

Employment status will also be described on the FAS using descriptive statistics for the following variables:

- Time from aSAH to return to work
- Time from aSAH to return to education
- Proportion of subjects fully back to pre-aSAH status, partially back to pre-aSAH status, not back to pre-aSAH

A listing will provide the status for each time point. It will also display the date of return to work (or to an educational institution, for students, as applicable) and the corresponding number of days elapsed since aSAH.

## 6.8 Biomarker endpoints analysis

The biomarker endpoints are:

 Presence of abnormal S100b protein concentration defined as the max observed concentration between study drug start and day14 in S100b being greater than or equal to 0.4 μg/L

#### 6.8.1 Variables

The presence of abnormal concentration of S100b between study drug start and Day 14 will be derived.

## 6.8.2 Analysis

#### **Tables**

Descriptive statistics for the level of S100b protein at baseline will be tabulated by treatment group on the FAS. The table will also display the percentages of subjects with S100b protein greater or equal to 0.4  $\mu$ g/L at any time between study drug start and Day 14 with corresponding 95% Clopper-Pearson CI.

#### **Figures**

Values over time will be provided in graphical format (boxplots) by treatment group.

## Listings

One listing will be provided for the FAS. It will include all results from the central laboratory. The maximum concentration observed that will be used to derive the endpoint will be flagged. It will also include the day relative to study drug initiation.

#### 7 SAFETY VARIABLES AND ANALYSES

If not otherwise stated:

- All tables and listings will be produced on the SAF
- Subjects will be evaluated according to the actual treatment they received, which may differ from the randomly assigned treatment

In the event of an administration error, i.e., a subject was administered both placebo and active treatment, the subject will be analyzed as active treatment ('clazosentan').

For partial date handling see Section 10.1.

## 7.1 Adverse events

The original terms used by the investigators to describe adverse events (AEs) in the Adverse Events eCRF are assigned a PT and a System Organ Class (SOC) for classification and tabulation using MedDRA v25.

Subjects who experienced the same AE more than once (as qualified by the same PT) are counted only once.

#### 7.1.1 Variables

#### All adverse events

All AEs are those occurring from signature of the ICF until EOS visit, which are believed to be related to a protocol-mandated procedure as well as treatment-emergent adverse events (TEAEs).

## Treatment-emergent adverse events

An AE is treatment-emergent if the onset date/time  $\geq$  start date/time of study treatment up to 24 hours after study treatment discontinuation.

An incomplete (time, day or month missing) or missing AE date will be imputed as described in the Table 7. The 'lower limit' and 'upper limit' refer to the earliest and latest possible date/times, respectively. As an example: If AE onset date is MAR2017 (time and day missing), the lower limit is 01MAR2017 T00:00:01 and the upper limit is 31MAR2017 T23:59:59; if AE onset date is 2017 (time, day and month missing), the lower limit is 01JAN2017T00:00:01 and the upper limit is 31DEC2017T23:59:59.

Table 7 Imputation rules for an incomplete or missing AE datetime

| Field | Incomplete datetime | Missing datetime |
|---|---|---|
| AE resolution datetime | The upper limit. | No imputation: the AE is considered as ongoing. |
| AE onset datetime | The rules below apply in the order presented: 1. If the (imputed) AE end datetime is on or after the start of study treatment, and if the study treatment start falls within the upper and lower limits (inclusive), the study treatment start datetime is used. 2. If the AE resolution datetime is missing, and: if the study treatment start falls within the upper and lower limits (inclusive), the study treatment start datetime is used. 3. In all the other cases, the lower limit is used. | Whichever is the earlier of the AE resolution datetime or study treatment start datetime. |

AE = adverse event.

If the emergence of an AE cannot be determined based on the above imputation rules, the AE will be considered as treatment-emergent.

The purpose of imputing AE dates is only to determine the treatment emergence of an AE for the summary tables and listings. However, only the actual dates as reported in the eCRF will be listed. No imputed date is considered in the medical evaluation of an AE.

## Treatment-emergent adverse events related to study treatment

An AE is considered related to the study treatment if the investigator answered "related" to the question "Relationship to study treatment". If the relationship is missing, the AE is considered 'related'.

## Treatment-emergent adverse events by intensity

The intensity of an AE is determined by the investigator as 'mild', 'moderate' or 'severe'.

Subjects who experienced the same AE more than once (as qualified by the same PT), but with different intensities, are counted only once, using the worst reported intensity. If the intensity is missing, the event is considered severe.

#### Serious adverse events

An AE is considered serious if the investigator answered, "Yes" on the question "Serious?".

## Serious treatment-emergent adverse events

Serious AEs (SAEs) are considered treatment-emergent if their onset date/time  $\geq$  start date/time of study treatment up to 24 hours after study treatment discontinuation.

## Serious adverse events during the long-term follow-up

SAEs with an onset date/time  $\geq$  end date/time of study drug + 24 hours and up to EOS.

## Adverse events leading to death

An AE is considered fatal if the investigator ticked "Fatal" on the question "Outcome".

## Adverse events leading to premature discontinuation of study treatment

An AE is considered leading to premature discontinuation of study treatment if the investigator ticked "Permanently discontinued" on the question "Action taken with study treatment".

#### Adverse events of special interest

An AE is considered an AE of special interest (AESI) if it is treatment-emergent and belongs to any of the categories listed below (the corresponding MedDRA PTs/SMQs using MedDRA v25 are provided in Appendix 14.4):

- Brain oedema
- Cerebral haemorrhage
- Anaemia
- Lung complications
- Hypotension
- Oedema and fluid retention
- Tachyarrhythmia

## • Hepatic disorders

### Rescue therapy-specific adverse events

An AE is considered related to the rescue therapy if the investigator answered "related" to the question "Relationship to rescue therapy" in the AE page.

## 7.1.2 Analysis

An overview of the AEs by treatment group will be produced on the SAF. It will include the N (%) of subjects having at least one treatment-emergent:

- AE
- AE related to study treatment
- AE of severe intensity
- SAE
- SAE related to study treatment
- AE of special interest
- AE with a fatal outcome
- AE with a fatal outcome and related to study treatment
- AE leading to temporary interruption of study treatment
- AE leading to permanent discontinuation of study treatment

It will also include the N (%) of subjects having at least one:

- SAE during the long-term follow-up
- SAE during the long-term follow-up with fatal outcome

The tables specified in Table 8 will summarize the number (%) of subjects by treatment group based on the SAF.

Table 8 Summary of adverse event analyses

| Category | Approach |
|---|---|
| All AEs | |
| All TEAEs | <ul> <li>- N (%) of subjects having at least one event by SOC and PT (overall and by patient population high-risk prevention vs early treatment)</li> <li>- N (%) of subjects having at least one event by PT</li> <li>- N (%) of subjects having at least one event by SOC and PT and maximum intensity</li> </ul> |
| TEAEs of severe intensity | - N (%) of subjects having at least one event by SOC and PT |
| TEAEs related to study treatment | - N (%) of subjects having at least one event by and PT |
| TEAEs leading to temporary interruption of study treatment | - N (%) of subjects having at least one event by SOC and PT - N (%) of subjects having at least one event by PT |

| Category | Approach |
|---|---|
| TEAEs leading to permanent | - N (%) of subjects having at least one event by SOC and PT |
| discontinuation to study treatment | - N (%) of subjects having at least one event by PT |
| TEAEs with fatal outcome | - N (%) of subjects having at least one event by SOC and PT |
| | - N (%) of subjects having at least one event by PT |
| TEAEs with fatal outcome and | - N (%) of subjects having at least one event by SOC and PT |
| related to study treatment | - N (%) of subjects having at least one event by PT |
| Serious TEAEs | - N (%) of subjects having at least one event by SOC and PT (overall |
| | and by patient population high-risk prevention vs early treatment) |
| | - N (%) of subjects having at least one event by PT |
| SAEs during long-term follow-up | - N (%) of subjects having at least one event by SOC and PT |
| | - N (%) of subjects having at least one event by PT |
| Serious TEAEs related to study | - N (%) of subjects having at least one event by SOC and PT |
| treatment | - N (%) of subjects having at least one event by PT |
| SAEs with fatal outcome during | - N (%) of subjects having at least one event by SOC and PT |
| long-term follow-up | - N (%) of subjects having at least one event by PT |
| TEAEs of special interest | - N (%) of subjects having at least one event by category of interest |
| | and PT |
| Rescue therapy-specific AEs | - N (%) of subjects having at least one event by PT |

AE = adverse event; PT = preferred term; SAE = serious adverse event; SOC = system organ class; TEAE = treatment-emergent adverse event.

A table will display the most frequent TEAE (at least 5% in placebo or active group) by treatment group and by PT. The PTs will be sorted by decreasing frequency in the active group.

A table will display the primary cause of death for all deaths up to EOS by treatment group and by PT. The PTs will be sorted by decreasing frequency in the active group.

For disclosure to public database purposes the following table will also be produced:

- Treatment-emergent SAEs (including occurrences)
- Treatment-emergent SAEs related to study treatment (including occurrences)
- Most frequent (threshold to be defined at time of reporting) non-serious TEAEs (including occurrences)

For tables presented by SOC and PT, SOCs/PTs are sorted by descending frequency of the number of subjects in the clazosentan group. If the frequencies of SOCs or PTs are the same, alphabetical order is used.

For tables presented by PT, PTs are sorted by descending frequency of the number of subjects in the clazosentan group. If the frequencies of PTs are the same, alphabetical order is used.

All AEs captured from signature of ICF up to EOS will be reported in the subject listings, which include data collected in the eCRF as well as the coded terms (SOC, PT), a flag for treatment-emergent and a flag for waived event as defined in protocol section 9.1.3 [D-22.069].

The following additional listings will be produced:

- All deaths and associated primary cause of death will be listed
- All AEs of subjects randomized but not treated (RND)
- All the previous/concomitant medications for subjects with a waived SAE.
- All medical histories for subjects with a waived SAE.

## 7.2 Laboratory tests

Laboratory analyses are based on data received from the central laboratory. Laboratory data will be converted into Standard International (SI) units. Unless noted otherwise, summaries and listings will include scheduled, re-test, and unscheduled assessments.

Consistent with the AE emergence period, the study treatment period considered for the laboratory measurements analyses is defined as start date/time of study treatment up to 24 hours after study treatment discontinuation.

Descriptive summary statistics on the observed values and the change from baseline to last value (re-test and unscheduled assessments included) in the study treatment period for hematology and blood chemistry parameters will be summarized.

Marked laboratory abnormalities are defined in Table 9 in Appendix 14.5.

Treatment-emergent marked laboratory abnormalities (MLAs) are those which are not present at baseline (e.g., change from no marked abnormality to any marked abnormality) or if a worsening occurred from study drug initiation up to 24 hours after study drug discontinuation, as compared to the corresponding value at baseline (e.g., change from a pre-existing abnormality at baseline to a worse category of abnormality).

The number (%) of subjects with newly occurring or worsening MLAs during study treatment period will be tabulated. A subject will be counted only once but may be reported in more than one MLA criterion of a given parameter. Percentages will be based on the number of subjects at risk, i.e., those having at least one post-baseline value and not meeting the criteria at baseline (or having a missing baseline value) for a given parameter.

Treatment-emergent liver function abnormalities occurring at any time post-baseline are identified according to the following criteria; a subject is considered to have met the criteria if they have at least one abnormality based on the worst post-baseline value measured:

- ALT  $> 3, > 5, > 8 \times ULN, > 10 \times ULN$
- AST > 3, > 5, >  $8 \times ULN$ , >  $10 \times ULN$

- AST or ALT > 3, > 5, >  $8 \times ULN$ , >  $10 \times ULN$
- $TBL > 2 \times ULN$
- TBL  $> 2 \times ULN$  combined with ALT or AST  $> 3 \times ULN$
- ALT or AST  $> 3 \times ULN + TBL > 2 \times ULN + ALP < 2 \times ULN$

For criteria combining several parameters, the abnormality must be reported at the same visit (same sample date).

The number (%) of subjects meeting the criteria defined above will be tabulated by treatment group. Percentages will be based on the number of subjects at risk, i.e., those having at least one post-baseline value and not meeting the criteria at baseline for a given parameter. In the event a subject's baseline value is missing:

- the subject will be considered 'at risk' for an abnormality formulated as a post-baseline value, but:
- the subject will be considered not 'at risk' for an abnormality formulated as a change from baseline.

A similar table will be produced on all post-baseline marked abnormalities.

Individual results will be listed by category (e.g., Hematology, Blood chemistry), by subject number and by visit / study day for all subjects, including central laboratory results.

All laboratory data for subjects with at least one MLA during study treatment will be listed. Any local laboratory data collected will be listed separately.

# 7.3 Electrocardiography

Descriptive summary statistics on the observed values and the change from baseline to last value (re-test and unscheduled assessments included) in the study treatment period for the 12 lead ECG parameters will be summarized by treatment group on the SAF.

The QT corrected with Fridericia's formula (QTcF) will be derived from the reported QT and RR using the following formula:

$$QTcF (msec) = QT (msec) / RR^{1/3}$$

For this parameter, additional flags will be defined:

Marked ECG abnormalities are defined below for QTcF:

- Value > 450, Value > 480, Value > 500
- Increase from baseline > 30, Increase from baseline > 60
- Value > 450 and increase from baseline > 30
- Value > 450 and increase from baseline > 60
- Value > 500 and increase from baseline > 30
- Value > 500 and increase from baseline > 60.

Number (%) of subjects with a marked QTcF abnormality during the study treatment period will be tabulated by treatment group. Percentages will be based on the number of subjects at risk, i.e., those having at least one post-baseline value and not meeting the criteria at baseline for a given parameter. In the event a subject's baseline value is missing:

- the subject will be considered 'at risk' for an abnormality formulated as a post-baseline value, but:
- the subject will be considered not 'at risk' for an abnormality formulated as a change from baseline.

All data (values and changes) will be listed by assessment. The listing will include date and time of measurements as well as the day, relative to study drug initiation.

## 7.4 Vital signs

Descriptive summary statistics on the average daily values and the change from baseline to each daily average post-baseline value in the study treatment period will be summarized for the following parameters:

- Systolic blood pressure (mmHg)
- Diastolic blood pressure (mmHg)
- Heart rate (beats/min)
- Central venous pressure (mmHg)
- Intracranial pressure (mmHg)
- Body temperature (°C)

All data (values and changes) will be listed by assessment. The listing will include date and time of measurements as well as the day, relative to study drug initiation.

## 7.5 Other safety variables and analyses

#### 7.5.1 Fluid balance

Daily fluid balance will be computed by subtracting the daily input and the daily output when they are both available and will be categorized according to the following classes:

| Imbalance categories | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Class boundaries (L) | >0,≤1 | > 1, \le 2 | >2,≤3 | >3, <u>&lt;</u> 4 | >4, ≤5 | >5, ≤6 | >6 |

Negative fluid balance will not be categorized. For each subject the periods of at least two consecutive days with fluid balance of category 2 or higher will be flagged.

A table displaying the proportion of subjects with at least one episode of fluid balance of category 2 or higher lasting for at least two consecutive days by treatment group will be produced on the SAF. A listing displaying daily fluid balance for all subjects will be

produced on the SAF. Periods of at least two consecutive days with fluid balance of category 2 or higher will be flagged.

## 7.6 Subgroup analysis of safety variables

The following subgroups will be used for safety analyses:

- WFNS grade at hospital admission, dichotomized as I–II vs III–V
- Age (years) at hospital admission, dichotomized as < 60 and  $\ge 60$
- Geographical location (USA vs non-USA, Europe vs non-Europe)
- Race (White; Black or African American; Asian). Subjects in the "Other" category will be excluded from the analysis given the small number of subjects.
- Sex
- Type of aneurysm-securing procedure (coiling vs clipping). If both were used, the last one is used for analysis.
- Good neurological recovery (mGCS  $\geq$  14 and aNIHSS = 0 vs. complement)

The following tables [see Table 8 for details] will be repeated on the subgroups (and their complements) defined above:

- TEAEs
- TEAEs of special interest
- TEAEs leading to premature discontinuation of study treatment
- Serious TEAEs

## 8 GENERAL STATISTICAL METHODOLOGY

Descriptive statistics will be provided by treatment group depending on the nature of the variable:

- For continuous variables: number of observed values, mean, standard deviation, minimum, first quartile, median, third quartile and maximum
- For dichotomous or categorical variables: number of observed values, and frequency with percentage per level/ category

Data are listed and summarized as described below.

The tables will use the following header structure (label and order):

| Clazosentan 15 mg/h | Placebo |
|---------------------|---------|
| N = xxx | N = xxx |

Where N indicates the total number randomized or treated appropriate to the analysis set in the corresponding treatment group, unless otherwise specified.

#### 9 INTERIM ANALYSES AND DATA MONITORING COMMITTEES

Not applicable, IDMC analyses are described in a separate SAP.

# 10 GENERAL DEFINITIONS AND DERIVATIONS

## 10.1 Handling of missing date

This section describes some general principles to be followed in the case of missing or incomplete dates.


Missing dates will not necessarily be replaced (e.g., medical history). Unless specified otherwise, partially known dates will be defined as:

- Partially known start date:
  - If only the day is missing, and month and year of the episode = month and year of study drug initiation, then otherwise
     Start date = date of study drug initiation, Start date = yyyy-mm-01.
  - If month and day are missing, and year of the episode = year of study drug initiation, then
    Start date = date of study drug initiation,
    otherwise
    Start date = yyyy-01-01
- Partially known end date:
- If only the day is missing, and month and year of the episode = month and year of study drug discontinuation, then the body drug discontinuation, then the body drug discontinuation, and the study drug discontinuation, then the body drug discontinuation, and the study drug discontinuation, and the study drug discontinuation, and the body drug discontinuation.
- If month and day are missing, and year of the episode = year of study drug discontinuation, then if start date is less than or equal to study drug discontinuation then
   End date = date of study drug discontinuation, otherwise
   End date = yyyy-12-31

The original dates without estimation will be presented in the listings.

Any missing EOS date will be substituted with the date of database lock.

# 10.2 General analysis variables

**Baseline value** is defined as the last non-missing value before study drug initiation based on date and time (when collected).

**Analysis value** is defined as the value at the visit (numeric result in standard units).

**Absolute change from baseline** is defined as post-baseline value minus baseline value, i.e., a positive sign indicates an increase as compared to baseline.

Percent change from baseline is defined as the absolute change from baseline divided by the baseline value (if the baseline value is > 0) and then multiplied by 100.

**Ratio to baseline** is defined as the value at the visit divided by the value at baseline (if the baseline value is  $\neq 0$ ).

**Analysis date** is defined as the numeric SAS date derived from the date/time of assessment. It may be an imputed date.

**Analysis start date** is defined as the numeric SAS date derived from the start date/time of an event. It may be an imputed date.

**Analysis end date** is defined as the numeric SAS date derived from the end date/time of an event. It may be an imputed date.

Analysis relative day is estimated for several assessments (e.g., vital signs, laboratory data). It refers to the number of days elapsed since study drug initiation date plus 1 (e.g., Day 1 is the day of study drug initiation). For dates prior to study drug initiation, study day is the negative number of days elapsed between the date under consideration and the day of study drug initiation. Therefore, the study day is never 0.

Analysis day relative to aSAH is estimated for several assessments performed during screening period and at EOS visit (e.g., MoCA, EQ-5D-5L). It refers to the number of days elapsed since aneurysm rupture (aSAH) date plus 1 (e.g., Day 1 is the day of aSAH).

Analysis end relative day is estimated for several assessments, including AE end, treatment interruptions, concomitant medication end. It refers to the number of days between the end of the specific event and the study drug initiation.

**Hospital discharge date (time)** is defined as the latest end/discharge date (time) reported with subject location equal to 'Critical care unit or equivalent', 'Specialized care ward' or 'General care ward' among the location reported for the initial hospitalization.

**Discharge home** is defined as being discharged home fully or partially independent.

**Day 14** is defined as per protocol as 14<sup>th</sup> day after study drug start. This corresponds to the analysis relative day 15.

#### 10.3 Study treatment administration error

In the event of an administration error, i.e., a subject was administered both placebo and active treatment, the subject will be analyzed as active treatment ('clazosentan') in all analyses based on the SAF (i.e., in all analyses based on the actual treatment group).

#### 10.4 Other derivations

**Length/Duration:** Lengths and durations based on dates will be computed as end date minus start date plus 1.

Good and Full neurological recovery subgroup variable: If one of these subgroups cannot be derived for a given subject due to missing data then the subject will be considered to be in the corresponding complementary subgroup.

# 11 CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL

# 11.1 Changes in the conduct of the study / data collection

Addition of the EQ-5D questionnaire at Week 24 post-aSAH:

In order to have at least one QoL assessment performed later than 12 weeks after aSAH subjects will be interviewed for the EQ-5D questionnaire at a second timepoint, Week 24 post-aSAH (from protocol version 4 dated 7 January 2020). Accordingly, the study duration was adjusted from 3 to 6 months for the collection of the employment status, the EQ-5D and SAE data collection.

## Early treatment stratum:

Following decision of the IDMC held on 2 April 2021, the recruitment into the early treatment stratum was stopped. This decision was based on a low rate of recruitment into this cohort since the outset of the study, making the contribution of these subjects to the overall study futile.

## Main secondary endpoint definition:

In protocol version 7 the main secondary endpoint definition was updated: in addition to the already existing all-cause infarcts  $\geq 5$  cm<sup>3</sup> at Day 16 post-study drug initiation, clinically relevant infarcts < 5 cm<sup>3</sup> have been added. The latter are defined as those new or worsened infarcts < 5 cm<sup>3</sup> that occur in subjects with CEC-adjudicated clinical deterioration due to DCI [see Section 6.3.1 for details]. The initially planned analysis (up to and including protocol version 6) will still be performed but as an exploratory analysis [see Section 6.3.8 for details].

## Other secondary endpoint and testing strategy:

Since protocol version 7 the mRS has been formally included in the statistical hierarchical testing strategy, just before the GOSE [see Section 6.1.1 for details].

## 11.2 Changes to the analyses planned in the study protocol

### Early treatment stratum:

The number of subjects randomized in this stratum being very low, and according to IDMC decision considering the contribution of these subjects to the overall study futile, this stratum was no longer considered as an adjustment/stratification variable in all the analyses adjusted/stratified on the stratification factors used for randomization. The initially planned analysis of the primary endpoint (i.e., stratified on the 3 stratification factors) will be done, but as an exploratory analysis [see Section 6.2.8 for details].

#### Estimands:

As the study started before the ICH E9 (R1) guidance became effective [ICH 2019], the estimands were not described in the protocol or in the CSR SAP version 1. They are now

defined in Section 6.1.2. Redefining the analyses with the estimand framework led to no longer using a Per-protocol analysis set and to rather defining the list of the IEs, and the different strategies considered to address them.

## Biomarker endpoints analysis:

In the protocol, the biomarker endpoints are the area under the plasma concentration-time curve of S100b protein from baseline to Day 10 and from baseline to Day 14 post-study drug initiation. To accommodate the heterogeneity of the timing of the assessment, because some subjects may have been discharged early, and to align with previous studies, the following endpoint definition will be used: presence of abnormal S100b protein concentration defined as the max observed concentration between study drug start and Day 14 being greater or equal to  $0.4\mu g/L$ .

#### GOSE/mRS:

In the protocol, the main analysis of the dichotomized GOSE and mRS was specified as a CMH test stratified on the variables used in the randomization (i.e., WFNS grade [I–II vs III–V] and age [ $\leq$  60 and > 60 years] at admission). However, in previous studies it was found that subjects who had recovered well from their initial bleeding episode and aneurysm-securing procedure had on average a better GOSE/mRS score. This subgroup of subjects called "good neurological recovery" is defined as subjects with an mGCS  $\geq$  14 and an aNIHSS = 0 (absence of motor deficit) within 60 minutes prior to study drug initiation. The complement subgroup is called "neurological impairment". To gain further precision in treatment effect estimates, the analyses of GOSE and mRS will, in addition, be adjusted for good neurological recovery variable (mGCS  $\geq$  14 and aNIHSS = 0, Yes/No).

# 11.3 Clarifications concerning endpoint definitions and related variables or statistical methods

In protocol version 7 dated 18 February 2022, the main secondary endpoint definition was updated: in addition to the already existing all-cause infarcts  $\geq 5$  cm<sup>3</sup> at Day 16 post-study drug initiation, clinically relevant infarcts < 5 cm<sup>3</sup> have been added. The latter are defined as those new or worsened infarcts < 5 cm<sup>3</sup> that occur in subjects with CEC-adjudicated clinical deterioration due to DCI [see Section 6.3.1 for details].

The protocol defines that the treatment effect for the main efficacy analyses will be summarized using: the absolute difference in the rates, the OR, the RR and the RRR. However, to avoid redundancy as RRR = 1 - RR the RR will not be presented in statistical outputs.

The protocol defines the following pharmaco-economic endpoint: Number and type of episodes of rescue therapy, from randomization up to hospital discharge and from hospital discharge up to Week 12 post-aSAH. Total duration in days, rather than the number of episodes of rescue therapy, will be analyzed, and more specifically: (i) the total number of
days with protocol-specific rescue therapy and (ii) the total number of days with protocol-specific rescue therapy or local rescue therapy [see Section 5.4.5.3 for details].

# **11.4** Additional analyses to those planned in the study protocol Not applicable.

### 12 LIST OF TABLES, LISTINGS AND FIGURES

The complete list of Tables, Listings and Figures is stored in the Idorsia Electronic Document Management System.

For the mock-up catalog to be used during programming, please refer to the document stored in the Biometry Computing Environment.

Since all Tables, Listings and Figures are produced using SAS®, the output actually generated may slightly differ from the mock-ups presented in the study specific mock-up catalog.

#### 13 REFERENCES

- [D-22.069] A prospective, multi-center, double-blind, randomized, placebo-controlled, parallel-group, Phase 3 study to assess the efficacy and safety of clazosentan in preventing clinical deterioration due to delayed cerebral ischemia (DCI), in adult subjects with aneurysmal subarachnoid hemorrhage (aSAH). Idorsia Pharmaceuticals Ltd; Protocol Version 7 ID-054-304, 18 February 2022.
- [Chessel 2004] Chessel D, Dufour A, Thioulouse J. The ade4 Package I: One-Table Methods. R News. 2004;4(1):5-10 Available from: https://cran.r-project.org/doc/Rnews/Rnews 2004-1.pdf
- [Dolédec 1987], Dolédec S, Chessel, D. Rythmes saisonniers et composantes stationnelles en milieu aquatique I- Description d'un plan d'observations complet par projection de variables. Acta Oecologica, Oecologia Generalis, 8, 3, 403–426. French.
- [Hernández-Alava 2017] Hernández-Alava M, Pudney, S. Econometric modelling of multiple self-reports of health states: the switch from EQ-5D-3L to EQ-5D-5L in evaluating drug therapies for rheumatoid arthritis. J Health Econ. 2017;55:139-152.
- [ICH 2019] ICH Harmonised Tripartite Guideline. Addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials E9 (R1). 20 November 2019 [accessed on 25 July 2022]. Available from: https://database.ich.org/sites/default/files/E9-R1\_Step4\_Guideline\_2019\_1203.pdf
- [R Core Team 2020] R-project.org [Internet]. R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. 2020 [cited 25 July 2022]. Available from: https://www.R-project.org/

[Romesburg 1985] Romesburg HC. Exploring, confirming and randomization tests. Computers & Geosciences. 1985;11(1):19–37.

[Williams 1999] Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke. 1999 Jul;30(7):1362-9.

# 14 APPENDICES

# **14.1 Revision History**

| Version Date | Version | Implemented Change(s) |
|---|---|---|
| 31-OCT-2018 | 1.0 | Initial version |
| 26-JUL-2022 | 2.0 | <ul> <li>Definition of Estimands added</li> <li>Incorporate changes in protocol: <ul> <li>New/revised exploratory endpoints were added (protocol version 3)</li> <li>EQ-5D questionnaire was added at Week 24 post-aSAH, EOS visit was moved from Week 12 to Week 24, SAEs collected until Week 24 (protocol version 4)</li> <li>Follow-up visit / phone call was added for subject discharged prior to Day 14 to allow assessment of primary endpoint (protocol version 5)</li> <li>Discontinuation of the recruitment into the early treatment group following a recommendation received by the study IDMC on 2 April 2021 (protocol version 6)</li> <li>Revised definition of main secondary endpoint, mRS explicitly added to the overall testing strategy (protocol version 7)</li> <li>Imputation rules for missing CT scan at Day 16 (to address FDA comment from November 2018 on SAP Version 1)</li> </ul> </li> </ul> |
| 27-SEP-2022 | 3.0 | <ul> <li>GOSE/mRS: All GOSE/mRS analyses are now also adjusted for the partial neurological recovery variable (mGCS ≥ 14 and aNIHSS = 0, Yes/No).</li> <li>Subgroup analyses for safety variables were added.</li> <li>Minor updates/corrections/clarifications throughout the document.</li> </ul> |
| 26-JAN-2023 | 4.0 | <ul> <li>Name of the subgroup "partial neurological recovery" changed to "good neurological recovery subgroup".</li> <li>New table displaying main cause of death.</li> <li>New table displaying SAS procedure outputs.</li> </ul> |

24 January 2023

Doc No D-23.039

| Version Date | Version | Implemented Change(s) |
|---|---|---|
| | | <ul> <li>EQ-5D: Rule to reallocate visit was added.</li> <li>Update definition of marked abnormalities for ALT and AST.</li> <li>Minor updates/corrections/clarifications throughout the document.</li> </ul> |

ALT = alanine aminotransferase; AST = aspartate aminotransferase; aNIHSS = abbreviated National Institutes of Health Stroke Scale; aSAH = aneurysmal subarachnoid hemorrhage; CT = computed tomography; EOS = End-of-Study; EQ-5D = Euro Quality of Life-5D; GOSE = Glasgow Outcome Scale – Extended; IDMC =Independent Data Monitoring Committee; mGCS = modified Glasgow Coma Scale; mRS = modified Rankin Scale; SAE = serious adverse event.

Visit and assessment schedule for subjects in the high-risk prevention group

| | | | 1 | | | OBSERVATION Peri | ind | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | days post-study drug | | | | |
| | | | | | | pective of treatment du | | Extende | d FU Period | |
| | | SCREENING | | l . | | FMENT Period | iration) | 24 h safety FU | | h safety FU Period |
| PERIOD | | Period | | | | . 14 days of treatment) | | Period | | il EOS) |
| TERIOD | | 1 er iou | | | (111111: 10, 1114) | | | | WEEK 12 | END OF STUDY |
| | | :41.: 06 1 | h C A I | т | | for 14 days | | until 24 h post-SD | WEEK 12<br>VISIT | |
| | | WILIIII 90 I | hours post-aSAI | 1<br> | | post-SD start | 1 | stop | V1511 | (EOS) <sup>19</sup> |
| Timing / assessment | | | | | | | *** | | | |
| | 77 | E ICE | D | CD | | D . 1 | Worsening of | E 1 675 4 4 | 04.1 | 24 weeks (168 days |
| | | | Prior to study | | D ii . ICH8 | During observation | ≥ 2 points on mGCS / | End-of-Treatment | 84 days post- | ± 14 days) |
| | admission | | drug (SD) start | start | Daily in ICU <sup>8</sup> | period <sup>8</sup> | aNIHSS <sup>8</sup> | (EOT) | aSAH (± 7 d) | post-aSAH |
| Informed consent | | X | | | | | | | | |
| <b>Demographics</b> | | X | 37 | | | | | | | |
| Medical history | | X | X | | | | | | | |
| Incl./Excl. criteria | | X | | | | | | | | |
| Height, weight | | X | | | | | | | | |
| Vital signs (BP, HR, ICP <sup>1</sup> , | | | X | | q6h | q6h ( $\pm$ 1 h)<br>(every 12 h if not in | | | | |
| CVP¹) | | | (within 60 min) | | (± 1 h) | ICU) | | | | |
| Body temperature | | | X<br>(within 60 min) | | (every | X<br>12 h ± 1 h) | | | | |
| Fluid balance (24 h) <sup>16</sup> | | | X | 1 | X | , | | | | |
| ECG parameters | | | X<br>(within 60 min) | | | X <sup>9</sup> | | X (within 2 h post-SD stop) | | |
| Laboratory tests<br>(local [l]/ central [c]) | | X (1) | X (c)<br>(within 60 min) | | X <sup>10</sup> (c) (E | OD for 14 days) | X (1) / SpO <sub>2</sub> | X <sup>10</sup> (c) (within 2 h<br>post-SD stop) | | |
| Biomarker | | | X (c)<br>(within 60 min) | | X (c) (EOD for 14 days) X (c) if CNS cause | | | X (c) (within 2 h<br>post-SD stop) | | |
| Pregnancy test | | X (serum, (1)) | , | | | | | | X (urine) | |
| Concomitant medications <sup>18</sup> | | X | | | | | X | | | |
| Non-drug treatments /<br>interventions | | | X | | | | X | | | |
| WFNS | $X^2$ | X, X <sup>3</sup> | | ĺ | | | | | | |
| Total GCS | $X^2$ | $X, X^3$ | | 1 | | | | | | |
| | | , | 1 | ı | L | | I . | 1 | | |

24 January 2023

| | | | | | (for 1 | OBSERVATION Peri<br>4 days post-study drug is<br>spective of treatment du | initiation | | Extende | d FU Period |
|---|---|---|---|---|---|---|---|---|---|---|
| PERIOD | | SCREENING<br>Period | | | TREA | TMENT Period a. 14 days of treatment) | , | 24 h safety FU<br>Period | (From end of 24 unt | From end of 24 h safety FU Period until EOS) |
| | | within 96 l | nours post-aSAI | I | | for 14 days<br>post-SD start | | until 24 h post-SD<br>stop | WEEK 12<br>VISIT | END OF STUDY<br>(EOS) <sup>19</sup> |
| Timing / assessment | | | Prior to study<br>drug (SD) start | | Daily in ICU <sup>8</sup> | During observation period <sup>8</sup> | Worsening of<br>≥ 2 points on mGCS / aNIHSS <sup>8</sup> | End-of-Treatment<br>(EOT) | 84 days post-<br>aSAH (± 7 d) | 24 weeks (168 days<br>± 14 days)<br>post-aSAH |
| mGCS/aNIHSS | | | X<br>(within 30 min) | | q6h <sup>11</sup><br>(± 1 h) | X <sup>12</sup> (± 1 h) | X<br>(hourly ± 15 min for<br>first 2 h) | | | |
| Angiogram<br>(DSA or CTA) | X <sup>4</sup> | X<br>(local standard-<br>of-care, not<br>assessed<br>centrally) | | | | | X<br>(if CNS cause) | | | |
| CT scan | X <sup>4</sup> | X <sup>5</sup> | | | | | X<br>(if CNS cause) | X <sup>13</sup> (16 days post-<br>SD start) | | |
| Subject narrative | | | | | | | X (14 days post-SD start) | , | | |
| MoCA <sup>6</sup> | | 2 | K <sup>7</sup> | | | $X (14 \pm 1 \text{ day post-SD} $ start) 17 | | | X | |
| GOSE | | | | | | , | | | X | |
| SS-QoL, Ox-PAQ | | | | | | | | | X | |
| EQ-5D | | | | 37 | 37 | | | | X | X |
| Study drug administration Adverse events <sup>14</sup> | | | X | X | X | | X | | | |
| Serious adverse events <sup>15</sup> | | | <u>х</u><br>Х | | X<br>X | | | | | |
| Pharmaco-economic assessments | | | X | | | | X | | | |
| Employment status | | | | | | | | | | X |

- 1. ICP/CVP will be measured and recorded for those subjects with ICP and/or CVP monitoring in place.
- 2. If the subject was transferred from another hospital, the GCS score and WFNS grade will correspond to the assessments made at the referral hospital, unless these were not done or not reliable.
- 3. Two assessments: post aneurysm-securing procedure and prior to randomization.
- 4. If performed at a referral hospital, is of acceptable quality, and is available in digital format at the investigational site at the time of screening, does not need to be repeated.
- 5. This CT scan is to be performed at least 8 hours after the aneurysm-securing procedure and within 24 hours prior to randomization.

Clazosentan (ACT-108475) ID-054-304 (REACT)

24 January 2023


Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

- 6. Only performed if subject is GCS  $\geq$  13 and extubated (if applicable).
- 7. As soon as possible after recovering from the aneurysm-securing procedure and prior to SD start.
- 8. If there is a worsening of at least 2 points in the mGCS and/or the aNIHSS the assessments in the "worsening" column must be performed on top of the regularly scheduled assessments. The mGCS and the aNIHSS must be repeated hourly for at least the first 2 hours after a 2-point worsening. If the deterioration is believed to be of CNS origin, a cerebral angiogram and a cerebral CT scan must be performed within 6 hours of the start of the symptoms and submitted for central review and a blood sample for S100b protein must be drawn within 1 hour of the confirmation of the neurological deterioration episode or no later than 3 hours from the initial worsening. Local lab tests should be obtained as close as possible to the time of the clinical worsening (max. 1 hour after time of confirmed worsening) [See Section 7.2.2.2.1 for details].
- 9. QT, QRS, PR, RR intervals, and HR will be measured and recorded in the eCRF if subject experiences an AE related to cardiac rhythm abnormalities [see Section 7.2.3.7].
- 10. Any clinically significant laboratory values must be reported as an AE/SAE as appropriate and those still abnormal at the time of the EOS assessment will be followed up based on local routine standard-of-care. A local laboratory may be requested by the sponsor to document the event and its resolution, and the results recorded in the eCRF [see Section 7.2.4.1].
- 11. At least once per day for subjects that require uninterrupted continuous sedation.
- 12. After the end of the study drug infusion, the mGCS and aNIHSS will continue to be assessed every 6 hours if the subject is still in the ICU (or equivalent ward), until 14 days after study drug initiation. They will be assessed at least once per day if the subject requires continuous uninterrupted sedation. If the subject is no longer in the ICU (i.e., has been sent to a regular/general ward), the mGCS and aNIHSS will be assessed at least once every 12 hours (± 1 h) until 14 days after study drug initiation. In the unavoidable situation where the subject is discharged from the study site before completing the observation period, their clinical status must be followed up to cover the period between discharge and Day 14 post-study drug start. The follow-up should be performed on Day 14 post-study drug initiation or as soon as possible after. This follow-up is not required if the subject was discharged on Day 13 and there is at least one set of neurological assessment scales available on this day.
- 13. If the CT scan cannot be performed on the 16<sup>th</sup> day post-SD start, then it is acceptable if the CT scan is performed up to 7 days after Day 16. The CT scan will be performed on the day of hospital discharge for those subjects who are discharged from the hospital prior to 16 days after study drug start. If no CT scan is available at hospital discharge, the last CT scan performed prior to discharge may be used for this assessment. For further details see Section 7.2.2.4.4.
- 14. All AEs that occur after signing the ICF and up to the EOS visit must be recorded if related to a study-mandated procedure. All other AEs are to be reported from SD initiation until 24 hours post-permanent SD discontinuation.
- 15. All SAEs that occur after signing the ICF and up to the EOS visit must be recorded if related to a study-mandated procedure. All other SAEs are to be reported from SD initiation until EOS. Waived SAEs do not require reporting to the sponsor's Drug Safety department within 24 hours of the knowledge of its occurrence [see Section 9.1.3].
- 16. Applicable during study drug administration only. Balance is captured if a urine catheter is present. Otherwise, 24-hour fluid intake will be measured and recorded.
- 17. This MoCA will be performed on the day of hospital discharge for those subjects who are discharged from the hospital prior to 14 days after study drug start.
- 18. For details on the concomitant medication recording refer to Section 5.2.5.
- 19. The EOS visit is conducted remotely as a telephone interview.

AE = adverse event; aNIHSS = abbreviated National Institutes of Health Stroke Scale; aSAH = aneurysmal subarachnoid hemorrhage; BP = blood pressure; CNS = central nervous system; CT = computerized tomography; CTA = computerized tomography angiography; CVP = central venous pressure; DSA = digital subtraction angiography; ECG = electrocardiogram; eCRF = electronic case report form; EOD = every other day; EOS = End-of-Study; EOT = End-of-Treatment; FU = follow-up; GCS = Glasgow Coma Scale; GOSE = Glasgow Outcome Scale Extended; HR = heart rate; ICF = informed consent form; ICP = intracranial pressure; ICU = intensive care unit; mGCS = modified Glasgow Coma Scale; MoCA = Montreal Cognitive Assessment; Ox-PAQ = Oxford Participation and Activities Questionnaire; SAE = serious adverse event; SD = study drug; SpO<sub>2</sub> = peripheral capillary oxygen saturation; SS-QoL = Stroke-Specific Quality of Life; WFNS = World Federation of Neurological Societies.

Visit and assessment schedule for subjects in the early treatment stratum (recruitment in this stratum was discontinued from protocol version 6, dated 29 April 2021 onwards)

| PERIOD | | SCREENING<br>Period | | (mir | (for 14 irres | DBSERVATION Perilog days post-study drug is pective of treatment dum MENT Period 14 days of treatment) | initiation | 24 h safety<br>FU Period | Extended FU Period (From end of 24 h safety FU period until EOS) | |
|---|---|---|---|---|---|---|---|---|---|---|
| TEMOS | | until max. Day 14<br>post-aSAH | within 24 h of randomization | pre-<br>on | , max | for 14 days<br>post-SD start | | until 24 h post-SD stop | WEEK 12<br>VISIT | END OF STUDY<br>(EOS) <sup>21</sup> |
| Timing / assessment | Hospital<br>Admission | from ICF to randomization | Prior to study<br>drug (SD) start | Prior to study SD drug (SD) start start | | During observation period <sup>9</sup> | Worsening of<br>≥ 2 points on<br>mGCS /<br>aNIHSS <sup>9</sup> | End-of-Treatment<br>(EOT) | 84 days post-<br>aSAH (± 7 d) | 24 weeks (168 days<br>± 14 days)<br>post-aSAH |
| Informed consent | | X | | | | | | | | |
| Demographics | | X | | | | | | | | |
| Medical history | | X | X | | | | | | | |
| Incl./Excl. criteria | | X | | | | | | | | |
| Height, weight | | X | | | | | | | | |
| Vital signs (BP, HR, ICP <sup>1</sup> ,<br>CVP <sup>1</sup> ) | | | X<br>(within 60 min) | | q6h<br>(± 1 h) | q6h (± 1 h)<br>(every 12 h if not in<br>ICU) | | | | |
| Body temperature | | | X<br>(within 60 min) | | | X<br>very 12 h ± 1 h) | | | | |
| Fluid balance (24 h) <sup>18</sup> | | | X | | X | | | | | |
| ECG parameters | | | X<br>(within 60 min) | | | $X^{10}$ | | X (within 2 h<br>post-SD stop) | | |
| Laboratory tests (local [l]/<br>central [c]) | | X (l) | X (c)<br>(within 60 min) | | X <sup>11</sup> (c)<br>(EOD for 14 days) X (l)/SpO <sub>2</sub> | | X <sup>11</sup> (c) (within 2 h<br>post-SD stop) | | | |
| Biomarker | | | X (c) (within 60 min) | | X (c) X (c) (EOD for 14 days) (if CNS cause) | | X (c) (within 2 h<br>post-SD stop) | | | |
| Pregnancy test | | X (serum, (l)) | | | | | X (urine) | | | |
| Concomitant medications <sup>20</sup> | | X | | | | | | X | | |
| Non-drug treatments / interventions | | | X | | | | | X | | |
| WFNS | $X^2$ | $X, X^3$ | | | | | | | | |
| Total GCS | $X^2$ | $X, X^3$ | | | | | | | | |


Statistical Analysis Plan for CSR Version 4 Doc No D-23.039

| | | | | | | (for 14 irres | OBSERVATION Per<br>days post-study drug<br>pective of treatment du | initiation | | | ed FU Period |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PERIOD | | | ENING<br>riod | | (min | | MENT Period 14 days of treatment) | | 24 h safety<br>FU Period | | 4 h safety FU period til EOS) |
| TERIOD | | until ma | x. Day 14<br>aSAH | within 24 h of<br>randomization | pre-<br>on | . 0, max. | for 14 days post-SD star | t | until 24 h post-SD<br>stop | WEEK 12<br>VISIT | END OF STUDY<br>(EOS) <sup>21</sup> |
| Timing / assessment | Hospital<br>Admission | | ICF to<br>nization | Prior to study<br>drug (SD) start | SD<br>start | Daily<br>in ICU <sup>9</sup> | During observation period <sup>9</sup> | Worsening of<br>≥ 2 points on<br>mGCS /<br>aNIHSS <sup>9</sup> | End-of-Treatment<br>(EOT) | 84 days post-<br>aSAH (± 7 d) | 24 weeks (168 days<br>± 14 days)<br>post-aSAH |
| mGCS/aNIHSS | | | | X (within 30 min) | | q6h <sup>12</sup><br>(± 1 h) | X <sup>13</sup> (± 1 h) | X<br>(hourly ± 15 min<br>for first 2 h) | | | |
| Angiogram<br>(DSA or CTA) | X <sup>4</sup> | X <sup>17</sup> | X <sup>5</sup> | | | | | X<br>(if CNS cause) | | | |
| CT scan | X <sup>4</sup> | 2 | $X^6$ | | | | | X (if CNS cause) | X <sup>14</sup> (16 days<br>post-SD start) | | |
| Subject narrative | | | | | | | | X (14 days post-SD start) | | | |
| MoCA <sup>7</sup> | | | X | 8 | | | $X (14 \pm 1 \text{ day})$<br>post-SD start) 19 | | | X | |
| GOSE | | | | | | | | | | X | |
| SS-QoL, Ox-PAQ | | | | | | | | | | X | |
| EQ-5D | | | | | | | | 1 | | X | X |
| Study drug administration Adverse events <sup>15</sup> | | | X | | X | X | | | X | | |
| Serious adverse events <sup>16</sup> | | | X X | | | | | | X | | |
| Pharmaco-economic assessments | | | | X | | | | X | | | |
| Employment status | | | | | | | | | | | X |

- 1. ICP/CVP will be measured and recorded for those subjects with ICP and/or CVP monitoring in place.
- 2. If the subject was transferred from another hospital, the GCS score and WFNS grade will correspond to the assessments made at the referral hospital, unless these were not done or unreliable.
- 3. Two assessments: post aneurysm-securing procedure and prior to randomization.
- 4. If performed at a referral hospital, is of acceptable quality, and is available in digital format at the investigational site at the time of screening, does not need to be repeated.
- 5. The DSA or CTA which was performed according to local routine standard-of-care (preferably between Day 7 and 11 post-aSAH) and used to diagnose and document the vasospasm will be collected.
- 6. This CT scan is to be performed at least 8 hours after the aneurysm-securing procedure and within 24 hours prior to randomization.
- 7. Only performed if subject is  $GCS \ge 13$  and extubated (if applicable).

24 January 2023

- 8. As soon as possible after recovering from the aneurysm-securing procedure and prior to SD start.
- 9. If there is a worsening of at least 2 points in the mGCS and/or the aNIHSS the assessments in the "worsening" column must be performed on top of the regularly scheduled assessments. The mGCS and the aNIHSS must be repeated hourly for at least the first 2 hours after a 2-point worsening. If the deterioration is believed to be of CNS origin, a cerebral angiogram and a cerebral CT scan must be performed within 6 hours of the start of the symptoms and submitted for central review and a blood sample for S100b protein must be drawn within 1 hour of the confirmation of the neurological deterioration episode or no later than 3 hours from the initial worsening. Local lab tests should be obtained as close as possible to the time of the clinical worsening (max. 1 hour after time of confirmed worsening) [see Section 7.2.2.2.1 for details].
- 10. QT, QRS, PR, RR intervals, and HR will be measured and recorded in the eCRF if subject experiences an AE related to cardiac rhythm abnormalities [see Section 7.2.3.7].
- 11. Any clinically significant laboratory values must be reported as an AE/SAE as appropriate and those still abnormal at the time of the EOS assessment will be followed up based on local routine standard-of-care. A local laboratory may be requested by the sponsor to document the event and its resolution, and the results recorded in the eCRF [see Section 7.2.4.1].
- 12. At least once per day for subjects that require uninterrupted continuous sedation.
- 13. After the end of the study drug infusion, the mGCS and aNIHSS will continue to be assessed every 6 hours if the subject is still in the ICU (or equivalent ward), until 14 days after study drug initiation. They will be assessed at least once per day if the subject requires continuous uninterrupted sedation. If the subject is no longer in the ICU (i.e., has been sent to a regular/general ward), the mGCS and aNIHSS will be assessed at least once every 12 hours (± 1 h) until 14 days after study drug initiation. In the unavoidable situation where the subject is discharged from the study site before completing the observation period, their clinical status must be followed up to cover the period between discharge and Day 14 post-study drug start. The follow-up should be performed on Day 14 post-study drug initiation or as soon as possible after. This follow-up is not required if the subject was discharged on Day 13 and there is at least one set of neurological assessment scales available on this day.14. If the CT scan cannot be performed on the 16th day post-SD start, then it is acceptable if the CT scan is performed up to 7 days after Day 16. The CT scan will be performed on the day of hospital discharge for those subjects who are discharged from the hospital prior to 16 days after study drug start. If no CT scan is available at hospital discharge, the last CT scan performed prior to discharge may be used for this assessment. For further details see Section 7.2.2.4.4.
- 15. All AEs that occur after signing the ICF and up to the EOS visit must be recorded if related to a study-mandated procedure. All other AEs are to be reported from SD initiation until 24 hours post-permanent SD discontinuation.
- 16. All SAEs that occur after signing the ICF and up to the EOS visit must be recorded if related to a study-mandated procedure. All other SAEs are to be reported from SD initiation until EOS. Waived SAEs do not require reporting to the sponsor's Drug Safety department within 24 hours of the knowledge of its occurrence [see Section 9.1.3].
- 17. Angiogram performed as per local standard-of-care to confirm successful aneurysm-securing procedure. Angiogram not assessed centrally.
- 18. Applicable during study drug administration only. Balance is captured if a urine catheter is present. Otherwise, 24-hour fluid intake will be measured and recorded.
- 19. This MoCA will be performed on the day of hospital discharge for those subjects who are discharged from the hospital prior to 14 days after study drug start.
- 20. For details on the concomitant medication recording refer to Section 5.2.5.
- 21. The EOS visit is conducted remotely as a telephone interview.
- AE= adverse event; aNIHSS = abbreviated National Institutes of Health Stroke Scale; aSAH = aneurysmal subarachnoid hemorrhage; BP = blood pressure; CNS = central nervous system; CT = computerized tomography; CTA = computerized tomography angiography; CVP = central venous pressure; DSA = digital subtraction angiography; ECG = electrocardiogram; eCRF = electronic case report form; EOD = every other day; EOS = End-of-Study; EOT = End-of-Treatment; FU = follow-up; GCS = Glasgow Coma Scale; GOSE = Glasgow Outcome Scale Extended; HR = heart rate; ICF = informed consent form; ICP = intracranial pressure; ICU = intensive care unit; mGCS = modified Glasgow Coma Scale; MoCA = Montreal Cognitive Assessment; Ox-PAQ = Oxford Participation and Activities Questionnaire; SAE = serious adverse event; SD = study drug; SpO2 = peripheral capillary oxygen saturation; SS-QoL = Stroke-Specific Quality of Life; WFNS = World Federation of Neurological Societies.

# 14.3 Change from pre-aSAH to post-aSAH status

| Post-aSAH Pre-aSAH | Employed<br>full time | Employed part time | Employed<br>full time -<br>not yet<br>returned | Employed<br>part time -<br>not yet<br>returned | Employed<br>full time -<br>on work<br>disability | Employed<br>part time -<br>on work<br>disability | Retired | Unemployed | Homemaker | Student<br>full time | Student part time | Student<br>not yet<br>returned | Unknown |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Employed full time | F | P | NB | NB | NB | NB | P | P | P | P | P | NB | M |
| Employed part time | F | F | NB | NB | NB | NB | P | P | P | P | P | NB | M |
| Employed full time<br>- on work disability | F | P | NB | NB | NB | NB | P | P | P | P | P | NB | M |
| Employed part time - on work disability | F | F | NB | NB | NB | NB | P | P | P | P | P | NB | M |
| Retired | F | F | NB | NB | NB | NB | F | F | F | F | F | NB | M |
| Unemployed | F | F | NB | NB | NB | NB | P | F | F | F | F | NB | M |
| Homemaker | F | F | NB | NB | NB | NB | P | F | F | F | F | NB | M |
| Student full time | P | P | NB | NB | NB | NB | P | P | P | F | P | NB | M |
| Student part time | P | P | NB | NB | NB | NB | P | P | P | F | F | NB | M |
| Unknown | М | М | M | M | M | M | M | M | M | M | M | NB | M |

F = Fully Back; P = Partially Back; NB = Not Back; M = Missing.

# 14.4 Adverse events of special interest

This appendix contains the search criteria (provided as MedDRA PTs and PT codes) for the following AESIs:

- Brain oedema
- Cerebral hemorrhage
- Anaemia
- Lung complications
- Hypotension
- Oedema and fluid retention
- Tachyarrhythmia
- Hepatic disorders

# Overview of search criteria for clazosentan AESI

**Hepatic disorders** 

| MedDRA v25.0 |
|----------------------------|
| <u>Brain oedema</u> |
| <u>Cerebral hemorrhage</u> |
| <u>Anaemia</u> |
| Lung complications |
| <u>Hypotension</u> |
| Oedema and fluid retention |
| Tachyarrhythmia_ |

#### Brain oedema

MedDRA v25.0 code

The case will be included in this subgroup if it contains an event within the MedDRA HLGT "Increased intracranial pressure and hydrocephalus" (primary or secondary path), i.e., any of the following MedDRA PTs:

| Aqueductal stenosis | 10067575 |
|-----------------------------------------------|----------|
| Benign enlargement of the subarachnoid spaces | 10078477 |
| Brain compression | 10006112 |
| Brain dislocation syndrome | 10082220 |
| Brain herniation | 10006126 |
| Brain oedema | 10048962 |
| Cerebral ventricle collapse | 10073706 |
| Cerebrospinal fluid circulation disorder | 10075604 |
| Cerebrospinal fluid retention | 10065532 |
| Cerebrospinal thrombotic tamponade | 10052173 |
| Congenital aqueductal stenosis | 10066084 |
| Congenital hydrocephalus | 10010506 |
| Cytotoxic oedema | 10067276 |
| Dandy-Walker syndrome | 10048411 |
| Dialysis disequilibrium syndrome | 10059256 |
| External hydrocephalus | 10076670 |
| Hydrocephalus | 10020508 |
| Hypertensive hydrocephalus | 10058025 |
| Idiopathic intracranial hypertension | 10078904 |
| Intracranial pressure increased | 10022773 |
| Normal pressure hydrocephalus | 10029773 |
| Oval pupil | 10085734 |
| Papilloedema | 10033712 |
| Posthaemorrhagic hydrocephalus | 10079859 |
| Vasogenic cerebral oedema | 10067275 |

MedDRA v25.0 code

All PTs from the Haemorrhagic central nervous system vascular conditions (SMQ): The case will be included in this subgroup if it contains an event within the "Haemorrhagic central nervous system vascular conditions" SMQ, i.e., if it contains an event with any of the following MedDRA PTs:

| Basal ganglia haematoma | 10077031 |
|--------------------------------------------------|----------|
| Basal ganglia haemorrhage | 10067057 |
| Basal ganglia stroke | 10071043 |
| Basilar artery perforation | 10075736 |
| Brain stem haematoma | 10073230 |
| Brain stem haemorrhage | 10006145 |
| Brain stem microhaemorrhage | 10071205 |
| Brain stem stroke | 10068644 |
| Carotid aneurysm rupture | 10051328 |
| Carotid artery perforation | 10075728 |
| Central nervous system haemorrhage | 10072043 |
| Cerebellar haematoma | 10061038 |
| Cerebellar haemorrhage | 10008030 |
| Cerebellar microhaemorrhage | 10071206 |
| Cerebellar stroke | 10079062 |
| Cerebral aneurysm perforation | 10075394 |
| Cerebral aneurysm ruptured syphilitic | 10008076 |
| Cerebral arteriovenous malformation haemorrhagic | 10008086 |
| Cerebral artery perforation | 10075734 |
| Cerebral cyst haemorrhage | 10082099 |
| Cerebral haematoma | 10053942 |
| Cerebral haemorrhage | 10008111 |
| Cerebral haemorrhage foetal | 10050157 |
| Cerebral haemorrhage neonatal | 10008112 |
| Cerebral microhaemorrhage | 10067277 |
| Cerebrovascular accident | 10008190 |
| Cerebrovascular disorder | 10008196 |
| Epidural haemorrhage | 10073681 |
| Extra-axial haemorrhage | 10078254 |
| Extradural haematoma | 10015769 |
| Extradural haematoma evacuation | 10082797 |
| Extraischaemic cerebral haematoma | 10080347 |
| Foville syndrome | 10082594 |
| Haemorrhage intracranial | 10018985 |
| Haemorrhagic cerebellar infarction | 10085944 |
| Haemorrhagic cerebral infarction | 10019005 |
| Haemorrhagic stroke | 10019016 |
| Haemorrhagic transformation stroke | 10055677 |
| Intracerebral haematoma evacuation | 10062025 |
| Intracranial haematoma | 10059491 |

| Intracranial haemorrhage neonatal | 10086946 |
|---------------------------------------|----------|
| Intracranial tumour haemorrhage | 10022775 |
| Intraventricular haemorrhage | 10022840 |
| Intraventricular haemorrhage neonatal | 10022841 |
| Meningorrhagia | 10052593 |
| Perinatal stroke | 10073945 |
| Periventricular haemorrhage neonatal | 10076706 |
| Pituitary apoplexy | 10056447 |
| Pituitary haemorrhage | 10049760 |
| Putamen haemorrhage | 10058940 |
| Ruptured cerebral aneurysm | 10039330 |
| Spinal cord haematoma | 10076051 |
| Spinal cord haemorrhage | 10048992 |
| Spinal epidural haematoma | 10050162 |
| Spinal epidural haemorrhage | 10049236 |
| Spinal stroke | 10082031 |
| Spinal subarachnoid haemorrhage | 10073564 |
| Spinal subdural haematoma | 10050164 |
| Spinal subdural haemorrhage | 10073563 |
| Stroke in evolution | 10059613 |
| Subarachnoid haematoma | 10076701 |
| Subarachnoid haemorrhage | 10042316 |
| Subarachnoid haemorrhage neonatal | 10042317 |
| Subdural haematoma | 10042361 |
| Subdural haematoma evacuation | 10042363 |
| Subdural haemorrhage | 10042364 |
| Subdural haemorrhage neonatal | 10042365 |
| Thalamus haemorrhage | 10058939 |
| Vertebral artery perforation | 10075735 |
| Vertebrobasilar stroke | 10082484 |

MedDRA v25.0 code

The case will be included in this subgroup if it contains an event within the "Haematopoietic erythropenia" SMQ or the "Haematopoietic cytopenias affecting more than one type of blood cell" SMQ, or it contains an event with any MedDRA Preferred Term containing the text "anaemia" (with the exception of the PT "Melanaemia"), or with the PT "Haemodilution"

i.e., any of the following MedDRA PTs:

| Anaemia | 10002034 |
|-----------------------------------------------------|----------|
| Anaemia folate deficiency | 10002043 |
| Anaemia Heinz body | 10002058 |
| Anaemia macrocytic | 10002064 |
| Anaemia megaloblastic | 10002065 |
| Anaemia neonatal | 10002068 |
| Anaemia of chronic disease | 10002073 |
| Anaemia of malignant disease | 10049105 |
| Anaemia of pregnancy | 10066468 |
| Anaemia postoperative | 10048861 |
| Anaemia prophylaxis | 10050250 |
| Anaemia splenic | 10049009 |
| Anaemia vitamin B12 deficiency | 10002080 |
| Anaemia vitamin B6 deficiency | 10002081 |
| Aplasia pure red cell | 10002965 |
| Aplastic anaemia | 10002967 |
| Aspiration bone marrow abnormal | 10003506 |
| Autoimmune anaemia | 10080243 |
| Autoimmune aplastic anaemia | 10071576 |
| Autoimmune haemolytic anaemia | 10073785 |
| Autosomal recessive megaloblastic anaemia | 10081878 |
| Bicytopenia | 10058956 |
| Biopsy bone marrow abnormal | 10004738 |
| Blood disorder | 10061590 |
| Blood incompatibility haemolytic anaemia of newborn | 10056369 |
| Blood loss anaemia | 10082297 |
| Blood loss anaemia neonatal | 10005644 |
| Bone marrow disorder | 10061729 |
| Bone marrow failure | 10065553 |
| Bone marrow infiltration | 10075173 |
| Bone marrow myelogram abnormal | 10057528 |
| Bone marrow necrosis | 10058822 |
| Cardiac haemolytic anaemia | 10072202 |
| Cold type haemolytic anaemia | 10009868 |
| Congenital anaemia | 10010329 |
| Congenital aplastic anaemia | 10053138 |
| Congenital dyserythropoietic anaemia | 10081457 |

| Coombs negative haemolytic anaemia | 10010940 |
|---------------------------------------------------------|----------|
| Coombs positive haemolytic anaemia | 10010940 |
| Cytopenia | 10066274 |
| Deficiency anaemia | 10060274 |
| Erythroblast count abnormal | 10051101 |
| Erythroblast count decreased | 10058505 |
| Erythroid dysplasia | 10036303 |
| Erythroid maturation arrest | 10030470 |
| Erythropenia Erythropenia | 10015277 |
| Erythropoiesis abnormal | 10013287 |
| Erythropoietin deficiency anaemia | 10043467 |
| Febrile bone marrow aplasia | 10063236 |
| Foetal anaemia | 10033213 |
| Full blood count decreased | 10077377 |
| Gelatinous transformation of the bone marrow | |
| | 10078097 |
| Haematocrit abnormal | 10049221 |
| Haematocrit decreased | 10018838 |
| Haematotoxicity | 10061188 |
| Haemodilution | 10059484 |
| Haemoglobin abnormal | 10018879 |
| Haemoglobin decreased | 10018884 |
| Haemolytic anaemia | 10018916 |
| Haemolytic anaemia enzyme specific | 10018919 |
| Haemolytic icteroanaemia | 10054920 |
| Hand and foot syndrome secondary to sickle cell anaemia | 10048775 |
| Hereditary haemolytic anaemia | 10060893 |
| Hereditary microcytic anaemia | 10085905 |
| Hereditary sideroblastic anaemia | 10019902 |
| Hexokinase deficiency anaemia | 10020022 |
| Hyperchromic anaemia | 10020605 |
| Hypochromic anaemia | 10020969 |
| Hypoplastic anaemia | 10021074 |
| Immune-mediated cytopenia | 10084828 |
| Iron deficiency anaemia | 10022972 |
| Leukoerythroblastic anaemia | 10053199 |
| Microangiopathic haemolytic anaemia | 10027527 |
| Microcytic anaemia | 10027538 |
| Myelodysplastic syndrome | 10028533 |
| Myelodysplastic syndrome transformation | 10067387 |
| Myelofibrosis | 10028537 |
| Myeloid metaplasia | 10028561 |
| Myelosuppression | 10028584 |
| Nephrogenic anaemia | 10058116 |
| Normochromic anaemia | 10029782 |
| Normochromic normocytic anaemia | 10029783 |
| Normocytic anaemia | 10029784 |
| Pancytopenia | 10033661 |
| Panmyelopathy | 10050026 |
| Pernicious anaemia | 10034695 |

| Plasmablast count decreased | 10058774 |
|---------------------------------------------|----------|
| Primary myelofibrosis | 10077161 |
| Proerythroblast count abnormal | 10060227 |
| Proerythroblast count decreased | 10060229 |
| Protein deficiency anaemia | 10037006 |
| Pyruvate kinase deficiency anaemia | 10037682 |
| Radiation anaemia | 10085644 |
| Red blood cell count abnormal | 10038151 |
| Red blood cell count decreased | 10038153 |
| Refractory anaemia with an excess of blasts | 10038270 |
| Refractory anaemia with ringed sideroblasts | 10038272 |
| Reticulocyte count abnormal | 10038788 |
| Reticulocyte count decreased | 10038790 |
| Reticulocyte percentage decreased | 10059921 |
| Reticulocytopenia | 10038795 |
| Scan bone marrow abnormal | 10053504 |
| Scorbutic anaemia | 10086662 |
| Sickle cell anaemia | 10040641 |
| Sickle cell anaemia with crisis | 10040642 |
| Sideroblastic anaemia | 10040661 |
| Spherocytic anaemia | 10041509 |
| Spur cell anaemia | 10052483 |
| Warm autoimmune haemolytic anaemia | 10087091 |

MedDRA v25.0 MedDRA v25.0 code

The case will be included in this subgroup if it contains an event with the PTs "Bronchospasm", "Bronchospasm paradoxical", "Unilateral bronchospasm",

or with a PT containing "pneumonia" from within the following MedDRA High Level terms:

Bacterial lower respiratory tract infections

Fungal lower respiratory tract infections

Lower respiratory tract and lung infections

Lower respiratory tract infections NEC

Lower respiratory tract inflammatory and immunologic conditions

Viral lower respiratory tract infections

#### Or with a PT within any of the following MedDRA HLTs:

Conditions associated with abnormal gas exchange

Parenchymal lung disorders NEC

Pneumothorax and pleural effusions NEC

Pulmonary oedemas

Pulmonary thrombotic and embolic conditions

Respiratory failures (excl neonatal)

i.e. any of the following MedDRA PTs (exact match):

| Acute interstitial pneumonitis | 10066728 |
|-------------------------------------|----------|
| Acute lung injury | 10069351 |
| Acute pulmonary oedema | 10001029 |
| Acute respiratory distress syndrome | 10001052 |
| Acute respiratory failure | 10001053 |
| Alveolar aeration excessive | 10001874 |
| Alveolar lung disease | 10073344 |
| Alveolar proteinosis | 10001881 |
| Anaemic hypoxia | 10051899 |
| Anaphylactoid syndrome of pregnancy | 10067010 |
| Anoxia | 10002660 |
| Antisynthetase syndrome | 10068801 |
| Asphyxia | 10003497 |
| Atelectasis | 10003598 |
| Atypical mycobacterial pneumonia | 10071075 |
| Atypical pneumonia | 10003757 |
| Brain hypoxia | 10006127 |
| Bronchopulmonary disease | 10053420 |
| Bronchospasm | 10006482 |
| Bronchospasm paradoxical | 10006486 |
| Candida pneumonia | 10053158 |
| Capnothorax | 10070771 |
| Cardiopulmonary failure | 10051093 |
| Cardio-respiratory arrest | 10007617 |
| Cardio-respiratory distress | 10049874 |
| Catamenial pneumothorax | 10086100 |

| | 40050404 |
|---|---|
| Cement embolism | 10050484 |
| Chronic respiratory failure | 10009126 |
| Chylothorax | 10051228 |
| Combined pulmonary fibrosis and emphysema | 10076515 |
| Complications of transplanted lung | 10010187 |
| Confirmed e-cigarette or vaping product use associated lung injury | 10085189 |
| Congenital chylothorax | 10078770 |
| Congenital emphysema | 10010456 |
| Congenital pneumonia | 10010594 |
| COPA syndrome | 10083948 |
| Coronavirus pneumonia | 10084381 |
| COVID-19 pneumonia | 10084380 |
| Cyanosis | 10011703 |
| Cyanosis central | 10011704 |
| Cystic lung disease | 10078811 |
| Diffuse idiopathic pulmonary neuroendocrine cell hyperplasia | 10082591 |
| Embolic pneumonia | 10065680 |
| Emphysema | 10014561 |
| Engraftment syndrome | 10050684 |
| Enterobacter pneumonia | 10054218 |
| Eosinophilic pleural effusion | 10080148 |
| Eosinophilic pneumonia | 10014962 |
| Eosinophilic pneumonia acute | 10052832 |
| Eosinophilic pneumonia chronic | 10052833 |
| Haemorrhagic pneumonia | 10077933 |
| Haemothorax | 10019027 |
| Hepatic hydrothorax | 10067365 |
| Herpes simplex pneumonia | 10065046 |
| Hydrothorax | 10048612 |
| Hypercapnia | 10020591 |
| Hypercapnic coma | 10072597 |
| Hyperoxia | 10058490 |
| Hypobarism | 10077606 |
| Hypocapnia | 10020952 |
| Нурохіа | 10021143 |
| Hypoxia intolerance | 10080129 |
| Hypoxic ischaemic encephalopathy neonatal | 10086943 |
| Hypoxic-ischaemic encephalopathy | 10070511 |
| Idiopathic interstitial pneumonia | 10078268 |
| Idiopathic pneumonia syndrome | 10063725 |
| Idiopathic pulmonary fibrosis | 10003723 |
| Interstitial lung disease | 10021210 |
| Leukostasis syndrome | 10074608 |
| Low lung compliance | 10074000 |
| Lung consolidation | 10030117 |
| Lung cyst | 10023080 |
| Lung induration | 10057261 |
| Lung infiltration | 10037201 |
| _ | |
| Lung perforation | 10076279 |

| | 10010150 |
|------------------------------------------------|----------|
| Lymphangioleiomyomatosis | 10049459 |
| MacLeod's syndrome | 10025375 |
| Metapneumovirus pneumonia | 10085550 |
| Metastatic pulmonary embolism | 10069909 |
| Middle lobe syndrome | 10056652 |
| Miliary pneumonia | 10055088 |
| Multifocal micronodular pneumocyte hyperplasia | 10057109 |
| Negative pressure pulmonary oedema | 10080589 |
| Neonatal pneumonia | 10053584 |
| Neonatal pneumothorax | 10082056 |
| Neuroendocrine cell hyperplasia of infancy | 10072968 |
| Non-cardiogenic pulmonary oedema | 10029538 |
| Obstetrical pulmonary embolism | 10029925 |
| Oesophageal-pulmonary fistula | 10083015 |
| Organising pneumonia | 10067472 |
| Paracancerous pneumonia | 10080986 |
| Paraneoplastic pleural effusion | 10075715 |
| Parasitic pneumonia | 10078883 |
| Pleural effusion | 10035598 |
| Pleuroparenchymal fibroelastosis | 10084305 |
| Pleuroperitoneal communication | 10068641 |
| Pneumocystis jirovecii pneumonia | 10073755 |
| Pneumonia | 10035664 |
| Pneumonia acinetobacter | 10079866 |
| Pneumonia adenoviral | 10035665 |
| Pneumonia anthrax | 10035667 |
| Pneumonia aspiration | 10035669 |
| Pneumonia bacterial | 10060946 |
| Pneumonia bordetella | 10035672 |
| Pneumonia chlamydial | 10035673 |
| Pneumonia cryptococcal | 10067565 |
| Pneumonia cytomegaloviral | 10035676 |
| Pneumonia escherichia | 10035699 |
| Pneumonia fungal | 10061354 |
| Pneumonia haemophilus | 10035702 |
| Pneumonia herpes viral | 10035703 |
| Pneumonia influenzal | 10035714 |
| Pneumonia klebsiella | 10035717 |
| Pneumonia legionella | 10035718 |
| Pneumonia lipoid | 10035720 |
| Pneumonia measles | 10035722 |
| Pneumonia moraxella | 10035723 |
| Pneumonia mycoplasmal | 10035724 |
| Pneumonia necrotising | 10055672 |
| Pneumonia parainfluenzae viral | 10035727 |
| Pneumonia pneumococcal | 10035728 |
| Pneumonia proteus | 10079867 |
| Pneumonia pseudomonal | 10035731 |
| Pneumonia respiratory syncytial viral | 10035732 |

| Pneumonia salmonella | 10035733 |
|-------------------------------------------------------------------|----------|
| Pneumonia serratia | 10079868 |
| Pneumonia staphylococcal | 10035734 |
| Pneumonia streptococcal | 10035735 |
| Pneumonia tularaemia | 10035736 |
| Pneumonia viral | 10035737 |
| Pneumothorax | 10035759 |
| Pneumothorax spontaneous | 10035763 |
| Pneumothorax traumatic | 10035765 |
| Polymer fume fever | 10077266 |
| Post procedural pneumonia | 10066590 |
| Post procedural pulmonary embolism | 10063909 |
| Postoperative respiratory distress | 10054809 |
| Postoperative respiratory failure | 10072651 |
| Probable e-cigarette or vaping product use associated lung injury | 10085188 |
| Procedural pneumothorax | 10077574 |
| Progressive massive fibrosis | 10036805 |
| Pulmonary air leakage | 10067826 |
| Pulmonary alveolar haemorrhage | 10037313 |
| Pulmonary alveolar microlithiasis | 10037315 |
| Pulmonary amyloidosis | 10063945 |
| Pulmonary artery thrombosis | 10037340 |
| Pulmonary atypical adenomatous hyperplasia | 10084570 |
| Pulmonary bullae rupture | 10086936 |
| Pulmonary calcification | 10051200 |
| Pulmonary cavitation | 10051738 |
| Pulmonary congestion | 10037368 |
| Pulmonary contusion | 10037370 |
| Pulmonary embolism | 10037377 |
| Pulmonary fibrosis | 10037383 |
| Pulmonary fistula | 10065873 |
| Pulmonary haemosiderosis | 10037396 |
| Pulmonary infarction | 10037410 |
| Pulmonary interstitial emphysema syndrome | 10037415 |
| Pulmonary microemboli | 10037421 |
| Pulmonary necrosis | 10058824 |
| Pulmonary nodular lymphoid hyperplasia | 10077412 |
| Pulmonary oedema | 10037423 |
| Pulmonary oedema neonatal | 10050459 |
| Pulmonary oedema post fume inhalation | 10037427 |
| Pulmonary oil microembolism | 10069388 |
| Pulmonary ossification | 10070310 |
| Pulmonary pneumatocele | 10063749 |
| Pulmonary thrombosis | 10037437 |
| Pulmonary toxicity | 10061924 |
| Pulmonary tumour thrombotic microangiopathy | 10079988 |
| Pulmonary venous thrombosis | 10037459 |
| Reexpansion pulmonary oedema | 10064715 |
| Respiratory acidosis | 10038661 |

| Respiratory alkalosis | 10038664 |
|-----------------------------------------------------------|----------|
| Respiratory failure | 10038695 |
| Respiratory gas exchange disorder | 10062105 |
| Respiratory paralysis | 10038708 |
| Restrictive allograft syndrome | 10077506 |
| Restrictive pulmonary disease | 10048667 |
| Rheumatoid arthritis-associated interstitial lung disease | 10085517 |
| Septic pulmonary embolism | 10083093 |
| Transfusion-related acute lung injury | 10052235 |
| Traumatic haemothorax | 10074487 |
| Traumatic lung injury | 10069363 |
| Unilateral bronchospasm | 10072338 |
| Varicella zoster pneumonia | 10074254 |

The case will be included in this subgroup if it contains an event with a PT containing ("Blood pressure" AND "decreased"), or with the PT "Blood pressure immeasurable", "Mean arterial pressure decreased", "Circulatory collapse", "Hypotensive crisis", "Peripheral circulatory failure" or with a PT containing "hypotension" (with the exception of the PTs Dialysis hypotension, Intracranial hypotension, Neonatal hypotension"), or with any of the following selected PTs containing "shock" (Cardiogenic shock, Distributive shock, Hypovolaemic shock, Procedural shock, Shock, Shock haemorrhagic, Shock symptom), i.e., if it contains any of the following MedDRA PTs:

| Blood pressure ambulatory decreased | 10005731 |
|-----------------------------------------------|----------|
| Blood pressure systolic inspiratory decreased | 10005761 |
| Blood pressure systolic decreased | 10005758 |
| Blood pressure orthostatic decreased | 10053356 |
| Blood pressure diastolic decreased | 10005737 |
| Blood pressure decreased | 10005734 |
| Blood pressure immeasurable | 10005748 |
| Mean arterial pressure decreased | 10026983 |
| Circulatory collapse | 10009192 |
| Peripheral circulatory failure | 10034567 |
| Hypotensive crisis | 10083659 |
| Hypotension | 10021097 |
| CT hypotension complex | 10078280 |
| Diastolic hypotension | 10066077 |
| Procedural hypotension | 10062300 |
| Post procedural hypotension | 10084013 |
| Orthostatic hypotension | 10031127 |
| Shock | 10040560 |
| Cardiogenic shock | 10007625 |
| Distributive shock | 10070559 |
| Hypovolaemic shock | 10021138 |
| Procedural shock | 10080894 |
| Shock haemorrhagic | 10049771 |
| Shock symptom | 10040581 |

MedDRA v25.0 code

The case will be included in this subgroup if it contains an event within the SMQ "Haemodynamic oedema, effusions and fluid overload (SMQ)" or with the PTs Swelling of eyelid, Swelling face, Eyelid oedema, Face oedema, i.e. the case will be included if it contains an event with any of the following MedDRA PTs:

| Acute pulmonary oedema | 10001029 |
|-------------------------------------------------------|----------|
| Administration site joint effusion | 10075944 |
| Administration site oedema | 10075104 |
| Administration site swelling | 10075107 |
| Amyloid related imaging abnormalities | 10072599 |
| Amyloid related imaging abnormality-microhaemorrhages | |
| and haemosiderin deposits | 10072601 |
| Amyloid related imaging abnormality-oedema/effusion | 10072260 |
| Application site joint effusion | 10076010 |
| Application site joint swelling | 10076016 |
| Application site oedema | 10003050 |
| Application site swelling | 10053424 |
| Ascites | 10003445 |
| Bone marrow oedema | 10051763 |
| Bone marrow oedema syndrome | 10064269 |
| Bone swelling | 10053631 |
| Brain oedema | 10048962 |
| Bronchial oedema | 10056695 |
| Capillary leak syndrome | 10007196 |
| Catheter site oedema | 10055909 |
| Cerebral mass effect | 10067086 |
| Cerebral oedema management | 10008128 |
| Cervix oedema | 10063817 |
| Circumoral swelling | 10081703 |
| Compression garment application | 10079209 |
| Cytotoxic oedema | 10067276 |
| Durotomy procedure | 10081615 |
| Effusion | 10063045 |
| Elephantiasis nostras verrucosa | 10071025 |
| Extensive swelling of vaccinated limb | 10065106 |
| Eyelid oedema | 10015993 |
| Face oedema | 10016029 |
| Flood syndrome | 10084797 |
| Fluid retention | 10016807 |
| Gallbladder oedema | 10017637 |
| Gastrointestinal oedema | 10058061 |
| Generalised oedema | 10018092 |
| Gestational oedema | 10063412 |
| Gravitational oedema | 10018713 |

| Hook and are | 10010240 |
|-----------------------------------------------------|----------------------|
| Heat oedema<br>Hydraemia | 10019340<br>10060374 |
| Hydrothorax | 10060374 |
| Hydrovarium | 10048012 |
| Hypervolaemia | 10081346 |
| Hypoosmolar state | 10020919 |
| | 10074867 |
| Implant site oedema | 10063776 |
| Implant site swelling | |
| Inadequate peritoneal dialysis Incision site oedema | 10085005 |
| | 10065614 |
| Incision site swelling | 10074758 |
| Infusion site joint effusion | 10076072 |
| Infusion site joint swelling | 10076078 |
| Infusion site oedema | 10053998 |
| Infusion site swelling | 10053505 |
| Injection site joint swelling | 10049260 |
| Injection site oedema | 10022085 |
| Injection site swelling | 10053425 |
| Instillation site oedema | 10073619 |
| Joint effusion | 10023215 |
| Joint swelling | 10023232 |
| Lipoedema | 10063955 |
| Localised oedema | 10048961 |
| Lumbar subcutaneous oedema | 10086593 |
| Lymphoedema | 10025282 |
| Lymphovenous bypass | 10084980 |
| Medical device site joint effusion | 10076117 |
| Medical device site joint swelling | 10076123 |
| Modified Rodnan skin score abnormal | 10081776 |
| Mouth swelling | 10075203 |
| Muscle oedema | 10071759 |
| Muscle swelling | 10064470 |
| Myocardial oedema | 10064966 |
| Negative pressure pulmonary oedema | 10080589 |
| Non-cardiogenic pulmonary oedema | 10029538 |
| Non-pitting oedema | 10083903 |
| Oedema | 10030095 |
| Oedema blister | 10080039 |
| Oedema due to cardiac disease | 10049632 |
| Oedema due to hepatic disease | 10049631 |
| Oedema due to renal disease | 10049630 |
| Oedema mucosal | 10030111 |
| Oedema neonatal | 10061317 |
| Oedema peripheral | 10030124 |
| Oedematous kidney | 10073381 |
| Oesophageal oedema | 10064342 |
| Omental oedema | 10087030 |
| Oropharyngeal oedema | 10078783 |
| Pelvic fluid collection | 10065388 |
| | . 5 5 5 5 5 5 6 6 |

| 10034474 |
|----------|
| 10059209 |
| 10078818 |
| 10049779 |
| 10048959 |
| 10035598 |
| 10074880 |
| 10037423 |
| 10050459 |
| 10074069 |
| 10064715 |
| 10063637 |
| 10038983 |
| 10055953 |
| 10084563 |
| 10058679 |
| 10053262 |
| 10063036 |
| 10054797 |
| 10042674 |
| 10042682 |
| 10042690 |
| 10086724 |
| 10043354 |
| 10076172 |
| 10076178 |
| 10067275 |
| 10065768 |

MedDRA v25.0 MedDRA v25.0 code

A case will be included in this subgroup if it contains an event within the following SMQ: Tachyarrhythmias (incl supraventricular and ventricular tachyarrhythmias) (SMQ) including all its sub-SMQs, or within the SMQ Torsade de pointes/QT prolongation (broad scope), i.e., any of the following MedDRA PTs:

| contains | aupu | ıcate | PIS |
|----------|------|-------|-----|
|----------|------|-------|-----|

| Arrhythmic storm | 10067339 |
|----------------------------------------------|----------|
| Cardiac arrest | 10007515 |
| Cardiac death | 10049993 |
| Cardiac fibrillation | 10061592 |
| Cardio-respiratory arrest | 10007617 |
| Electrocardiogram QT interval abnormal | 10063748 |
| Electrocardiogram QT prolonged | 10014387 |
| Electrocardiogram repolarisation abnormality | 10052464 |
| Electrocardiogram U wave inversion | 10062314 |
| Electrocardiogram U wave present | 10057913 |
| Electrocardiogram U-wave abnormality | 10055032 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Loss of consciousness | 10024855 |
| Sudden cardiac death | 10049418 |
| Sudden death | 10042434 |
| Syncope | 10042772 |
| Torsade de pointes | 10044066 |
| Ventricular arrhythmia | 10047281 |
| Ventricular fibrillation | 10047290 |
| Ventricular flutter | 10047294 |
| Ventricular tachyarrhythmia | 10065341 |
| Ventricular tachycardia | 10047302 |
| Accelerated idioventricular rhythm | 10049003 |
| Anomalous atrioventricular excitation | 10002611 |
| Arrhythmia supraventricular | 10003130 |
| Arrhythmic storm | 10067339 |
| Atrial fibrillation | 10003658 |
| Atrial flutter | 10003662 |
| Atrial parasystole | 10071666 |
| Atrial tachycardia | 10003668 |
| Cardiac fibrillation | 10061592 |
| Cardiac fibrillation | 10061592 |
| Cardiac flutter | 10052840 |
| Congenital supraventricular tachycardia | 10082343 |
| Early repolarisation syndrome | 10086230 |
| ECG P wave inverted | 10057526 |
| Electrocardiogram P wave abnormal | 10050384 |
| Extrasystoles | 10015856 |
| Frederick's syndrome | 10082089 |

| 10074640 |
|----------|
| 10033929 |
| 10071187 |
| 10039111 |
| 10040752 |
| 10042602 |
| 10065342 |
| 10042604 |
| 10049447 |
| 10044066 |
| 10047281 |
| 10047289 |
| 10047290 |
| 10047294 |
| 10058184 |
| 10049761 |
| 10065341 |
| 10047302 |

MedDRA v25.0 code

The case will be included in this subgroup if it contains an event within the "Hepatic disorders" SMQ.

| 5'nucleotidase increased | 10000028 |
|---------------------------------------------|----------|
| Accessory liver lobe | 10050020 |
| Acquired antithrombin III deficiency | 10074561 |
| Acquired factor IX deficiency | 10082747 |
| Acquired factor V deficiency | 10086006 |
| Acquired factor VIII deficiency | 10082745 |
| Acquired factor XI deficiency | 10082746 |
| Acquired hepatocerebral degeneration | 10080860 |
| Acquired protein S deficiency | 10068370 |
| Acute fatty liver of pregnancy | 10000746 |
| Acute graft versus host disease in liver | 10066263 |
| Acute hepatic failure | 10000804 |
| Acute hepatitis B | 10059193 |
| Acute hepatitis C | 10065051 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Adenoviral hepatitis | 10056885 |
| Alagille syndrome | 10053870 |
| Alanine aminotransferase abnormal | 10001547 |
| Alanine aminotransferase increased | 10001551 |
| Alcoholic encephalopathy | 10085656 |
| Alcoholic liver disease | 10001627 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Ammonia abnormal | 10001942 |
| Ammonia increased | 10001946 |
| Anorectal varices | 10068924 |
| Anorectal varices haemorrhage | 10068925 |
| Anti factor X activity abnormal | 10077670 |
| Anti factor X activity decreased | 10077674 |
| Anti factor X activity increased | 10077671 |
| Anti-liver cytosol antibody type 1 positive | 10086970 |
| Antithrombin III decreased | 10049547 |
| Ascites | 10003445 |
| Aspartate aminotransferase abnormal | 10003477 |
| Aspartate aminotransferase increased | 10003481 |
| AST to platelet ratio index increased | 10084175 |
| AST/ALT ratio abnormal | 10082832 |
| Asterixis | 10003547 |
| Asymptomatic viral hepatitis | 10063838 |
| Autoimmune hepatitis | 10003827 |
| Bacterascites | 10068547 |
| Benign hepatic neoplasm | 10004269 |

| Benign hepatobiliary neoplasm | 10077922 |
|---|---|
| Benign recurrent intrahepatic cholestasis | 10087038 |
| Bile output abnormal | 10051344 |
| Bile output decreased | 10051343 |
| Biliary ascites | 10074150 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Bilirubin conjugated abnormal | 10067718 |
| Bilirubin conjugated increased | 10004685 |
| Bilirubin excretion disorder | 10061009 |
| Bilirubin urine present | 10077356 |
| Biopsy liver abnormal | 10004792 |
| Blood alkaline phosphatase abnormal | 10059571 |
| Blood alkaline phosphatase increased | 10059570 |
| Blood bilirubin abnormal | 10058477 |
| Blood bilirubin increased | 10005364 |
| Blood bilirubin unconjugated increased | 10005370 |
| Blood cholinesterase abnormal | 10005429 |
| Blood cholinesterase decreased | 10005430 |
| Blood fibrinogen abnormal | 10005518 |
| Blood fibrinogen decreased | 10005520 |
| Blood thrombin abnormal | 10005818 |
| Blood thrombin decreased | 10005820 |
| Blood thromboplastin abnormal | 10005824 |
| Blood thromboplastin decreased | 10005826 |
| Bromosulphthalein test abnormal | 10006408 |
| Cardiohepatic syndrome | 10082480 |
| Cerebrohepatorenal syndrome | 10053684 |
| Child-Pugh-Turcotte score abnormal | 10077020 |
| Child-Pugh-Turcotte score increased | 10068287 |
| Cholaemia | 10048611 |
| Cholangiosarcoma | 10077861 |
| Cholestasis | 10008635 |
| Cholestasis of pregnancy | 10049055 |
| Cholestatic liver injury | 10067969 |
| Cholestatic pruritus | 10064190 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatic failure | 10057573 |
| Chronic hepatitis | 10008909 |
| Chronic hepatitis B | 10008910 |
| Chronic hepatitis C | 10008912 |
| Cirrhosis alcoholic | 10009208 |
| Coagulation factor decreased | 10009736 |
| Coagulation factor IX level abnormal | 10061770 |
| Coagulation factor IX level decreased | 10009746 |
| Coagulation factor V level abnormal Coagulation factor V level decreased | 10061771<br>10009754 |
| Coagulation factor V level decreased Coagulation factor VII level abnormal | 10009754 |
| Coagulation factor VII level decreased | 10061772 |
| Coagulation ractor virtevel decreased | 10009701 |

| Coagulation factor X level abnormal | 10061774 |
|----------------------------------------------------|----------|
| Coagulation factor X level decreased | 10009775 |
| Coma hepatic | 10010075 |
| Complications of transplanted liver | 10010186 |
| Computerised tomogram liver abnormal | 10078360 |
| Congenital absence of bile ducts | 10010317 |
| Congenital hepatic fibrosis | 10056533 |
| Congenital hepatitis B infection | 10010496 |
| Congenital hepatitis C infection | 10084252 |
| Congenital hepatobiliary anomaly | 10061065 |
| Congenital hepatomegaly | 10051130 |
| Congenital viral hepatitis | 10084251 |
| Congestive hepatopathy | 10084058 |
| Cryptogenic cirrhosis | 10063075 |
| Cystic fibrosis hepatic disease | 10068289 |
| Cytokeratin 18 increased | 10068471 |
| Cytomegalovirus hepatitis | 10011830 |
| Deficiency of bile secretion | 10071634 |
| Diabetic hepatopathy | 10071265 |
| Dilatation intrahepatic duct congenital | 10013003 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Fatty liver alcoholic | 10016262 |
| Flood syndrome | 10084797 |
| Focal nodular hyperplasia | 10052285 |
| Foetor hepaticus | 10052554 |
| Galactose elimination capacity test abnormal | 10059710 |
| Galactose elimination capacity test decreased | 10059712 |
| Gallbladder varices | 10072319 |
| Gamma-glutamyltransferase abnormal | 10017688 |
| Gamma-glutamyltransferase increased | 10017693 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Gianotti-Crosti syndrome | 10053842 |
| Glutamate dehydrogenase increased | 10049483 |
| Glycocholic acid increased | 10080824 |
| Glycogen storage disease type I | 10018464 |
| Glycogen storage disease type III | 10053250 |
| Glycogen storage disease type IV | 10053249 |
| Glycogen storage disease type VI | 10053240 |
| Graft versus host disease in liver | 10064676 |
| Granulomatous liver disease | 10018704 |
| Guanase increased | 10051333 |
| Haemangioma of liver | 10018821 |
| Haemorrhagic ascites | 10059766 |
| Haemorrhagic hepatic cyst | 10067796 |

| HBV-DNA polymerase increased | 10058937 |
|------------------------------------|----------|
| Hepaplastin abnormal | 10019621 |
| Hepaplastin decreased | 10019622 |
| Hepatectomy | 10061997 |
| Hepatic adenoma | 10019629 |
| Hepatic amoebiasis | 10063741 |
| Hepatic angiosarcoma | 10067388 |
| Hepatic artery flow decreased | 10068997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cancer | 10073069 |
| Hepatic cancer metastatic | 10055110 |
| Hepatic cancer recurrent | 10073070 |
| Hepatic cancer stage I | 10059318 |
| Hepatic cancer stage II | 10059319 |
| Hepatic cancer stage III | 10059324 |
| Hepatic cancer stage IV | 10059325 |
| Hepatic candidiasis | 10049653 |
| Hepatic cirrhosis | 10019641 |
| Hepatic cyst | 10019646 |
| Hepatic cyst infection | 10051705 |
| Hepatic cyst ruptured | 10053973 |
| Hepatic cytolysis | 10049199 |
| Hepatic echinococciasis | 10019659 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic enzyme abnormal | 10062685 |
| Hepatic enzyme decreased | 10060794 |
| Hepatic enzyme increased | 10060795 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic fibrosis marker abnormal | 10074084 |
| Hepatic fibrosis marker increased | 10074413 |
| Hepatic function abnormal | 10019670 |
| Hepatic gas gangrene | 10077055 |
| Hepatic haemangioma rupture | 10054885 |
| Hepatic hamartoma | 10079685 |
| Hepatic hydrothorax | 10067365 |
| Hepatic hypertrophy | 10076254 |
| Hepatic hypoperfusion | 10084751 |
| Hepatic infection | 10056522 |
| Hepatic infection bacterial | 10065215 |
| Hepatic infection fungal | 10065217 |
| Hepatic infection helminthic | 10065216 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic lipoma | 10086088 |
| Hepatic lymphocytic infiltration | 10079686 |
| Hepatic mass | 10057110 |

| Hepatic necrosis | 10019692 |
|--------------------------------------------|----------|
| Hepatic neoplasm | 10019695 |
| Hepatic neuroendocrine tumour | 10085864 |
| Hepatic pain | 10019705 |
| Hepatic perfusion disorder | 10083840 |
| Hepatic sarcoma | 10086958 |
| Hepatic sequestration | 10066244 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatic vascular resistance increased | 10068358 |
| Hepatic venous pressure gradient abnormal | 10083172 |
| Hepatic venous pressure gradient increased | 10083171 |
| Hepatitis | 10019717 |
| Hepatitis A | 10019719 |
| Hepatitis A antibody abnormal | 10019722 |
| Hepatitis A antibody positive | 10019725 |
| Hepatitis A antigen positive | 10058751 |
| Hepatitis A immunity confirmed | 10086044 |
| Hepatitis A virus test positive | 10070216 |
| Hepatitis acute | 10019727 |
| Hepatitis alcoholic | 10019728 |
| Hepatitis B | 10019731 |
| Hepatitis B antibody abnormal | 10019733 |
| Hepatitis B antibody positive | 10019736 |
| Hepatitis B antigen positive | 10063411 |
| Hepatitis B core antibody positive | 10071344 |
| Hepatitis B core antigen positive | 10052328 |
| Hepatitis B DNA assay positive | 10060047 |
| Hepatitis B DNA increased | 10068379 |
| Hepatitis B e antibody positive | 10071348 |
| Hepatitis B e antigen positive | 10052329 |
| Hepatitis B immunity confirmed | 10086043 |
| Hepatitis B reactivation | 10058827 |
| Hepatitis B surface antibody positive | 10071346 |
| Hepatitis B surface antigen positive | 10019742 |
| Hepatitis B virus test positive | 10070217 |
| Hepatitis C | 10019744 |
| Hepatitis C antibody positive | 10019747 |
| Hepatitis C core antibody positive | 10077052 |
| Hepatitis C RNA increased | 10068377 |
| Hepatitis C RNA positive | 10019750 |
| Hepatitis C virus test positive | 10070218 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis D | 10019762 |
| Hepatitis D antibody positive | 10059528 |
| Hepatitis D antigen positive | 10058436 |
| Hepatitis D RNA positive | 10059540 |

| | 40070606 |
|------------------------------------|----------|
| Hepatitis D virus test positive | 10070626 |
| Hepatitis E | 10019768 |
| Hepatitis E antibody abnormal | 10057994 |
| Hepatitis E antibody positive | 10057985 |
| Hepatitis E antigen positive | 10060049 |
| Hepatitis E immunity confirmed | 10086045 |
| Hepatitis E RNA positive | 10086906 |
| Hepatitis E virus test positive | 10070220 |
| Hepatitis F | 10019771 |
| Hepatitis fulminant | 10019772 |
| Hepatitis G | 10019773 |
| Hepatitis H | 10019776 |
| Hepatitis infectious mononucleosis | 10019781 |
| Hepatitis mumps | 10019783 |
| Hepatitis neonatal | 10019785 |
| Hepatitis non-A non-B | 10019786 |
| Hepatitis non-A non-B non-C | 10019787 |
| Hepatitis post transfusion | 10019791 |
| Hepatitis syphilitic | 10019794 |
| Hepatitis toxic | 10019795 |
| Hepatitis toxoplasmal | 10019798 |
| Hepatitis viral | 10019799 |
| Hepatitis viral test positive | 10072748 |
| Hepatobiliary cancer | 10073073 |
| Hepatobiliary cancer in situ | 10073074 |
| Hepatobiliary cyst | 10079889 |
| Hepatobiliary disease | 10062000 |
| Hepatobiliary infection | 10056523 |
| Hepatobiliary neoplasm | 10061203 |
| Hepatobiliary scan abnormal | 10066195 |
| Hepatoblastoma | 10062001 |
| Hepatoblastoma recurrent | 10019823 |
| Hepatocellular carcinoma | 10073071 |
| Hepatocellular damage neonatal | 10019834 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepato-lenticular degeneration | 10019819 |
| Hepatomegaly | 10019842 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatosplenic abscess | 10077631 |
| Hepatosplenic candidiasis | 10051590 |
| Hepatosplenomegaly | 10019847 |
| Hepatosplenomegaly neonatal | 10019848 |
| Hepatotoxicity | 10019851 |
| Hereditary haemochromatosis | 10057873 |
| Herpes simplex hepatitis | 10067389 |
| Hyperammonaemia | 10020575 |
| 21 | |

| Hyperbilirubinaemia | 10020578 |
|--------------------------------------------|----------|
| Hyperbilirubinaemia neonatal | 10020580 |
| Hypercholia | 10051924 |
| Hyperfibrinolysis | 10074737 |
| Hypertransaminasaemia | 10068237 |
| Hypoalbuminaemia | 10020942 |
| Hypocoagulable state | 10020973 |
| Hypofibrinogenaemia | 10051125 |
| Hypoprothrombinaemia | 10021085 |
| Hypothrombinaemia | 10058517 |
| Hypothromboplastinaemia | 10058518 |
| Icterus index increased | 10021209 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Immune-mediated hepatitis | 10078962 |
| Increased liver stiffness | 10082444 |
| International normalised ratio abnormal | 10022592 |
| International normalised ratio increased | 10022595 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Intrahepatic portal hepatic venous fistula | 10072629 |
| Ischaemic hepatitis | 10023025 |
| Jaundice | 10023126 |
| Jaundice cholestatic | 10023129 |
| Jaundice hepatocellular | 10023136 |
| Jaundice neonatal | 10023138 |
| Kayser-Fleischer ring | 10023321 |
| Kernicterus | 10023376 |
| Leucine aminopeptidase increased | 10024275 |
| Liver abscess | 10024652 |
| Liver and pancreas transplant rejection | 10051603 |
| Liver carcinoma ruptured | 10050842 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver function test abnormal | 10024690 |
| Liver function test decreased | 10077677 |
| Liver function test increased | 10077692 |
| Liver induration | 10052550 |
| Liver injury | 10067125 |
| Liver iron concentration abnormal | 10074352 |
| Liver iron concentration increased | 10074354 |
| Liver opacity | 10084071 |
| Liver operation | 10062040 |
| Liver palpable | 10075895 |
| Liver sarcoidosis | 10068664 |
| Liver scan abnormal | 10061947 |
| Liver tenderness | 10024712 |
| Liver transplant | 10024714 |
| Liver transplant failure | 10083175 |

| Liver transplant rejection | 10024715 |
|------------------------------------------------------------|----------|
| Liver-kidney microsomal antibody positive | 10060107 |
| Lupoid hepatic cirrhosis | 10025129 |
| Lupus hepatitis | 10067737 |
| Magnetic resonance imaging hepatobiliary abnormal | 10085121 |
| Magnetic resonance proton density fat fraction measuremen | 10082443 |
| Mitochondrial aspartate aminotransferase increased | 10064712 |
| Mixed hepatocellular cholangiocarcinoma | 10027761 |
| Mixed liver injury | 10066758 |
| Model for end stage liver disease score abnormal | 10077291 |
| Model for end stage liver disease score increased | 10077292 |
| Molar ratio of total branched-chain amino acid to tyrosine | 10066869 |
| Multivisceral transplantation | 10082450 |
| Necrolytic acral erythema | 10084061 |
| Neonatal cholestasis | 10056528 |
| Neonatal hepatomegaly | 10049995 |
| Nodular regenerative hyperplasia | 10051081 |
| Non-alcoholic fatty liver | 10029530 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Ocular icterus | 10058117 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Omental oedema | 10087030 |
| Osteopontin increased | 10082708 |
| Parenteral nutrition associated liver disease | 10074151 |
| Perihepatic discomfort | 10054125 |
| Perinatal HBV infection | 10075233 |
| Peripancreatic varices | 10073215 |
| Periportal oedema | 10068821 |
| Peritoneal fluid protein abnormal | 10069000 |
| Peritoneal fluid protein decreased | 10068999 |
| Peritoneal fluid protein increased | 10068998 |
| Peritoneovenous shunt | 10052716 |
| Pneumobilia | 10066004 |
| Polycystic liver disease | 10048834 |
| Porphyria acute | 10036182 |
| Porphyria non-acute | 10036186 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal pyaemia | 10036202 |
| Portal shunt | 10036204 |
| Portal shunt procedure | 10077479 |
| Portal tract inflammation | 10075331 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |

| Portal vein flow decreased | 10067337 |
|-----------------------------------------------------|----------|
| Portal vein pressure increased | 10064936 |
| Portal venous system anomaly | 10076609 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Progressive familial intrahepatic cholestasis | 10076033 |
| Protein C decreased | 10037005 |
| Protein S abnormal | 10051736 |
| Protein S decreased | 10051120 |
| Prothrombin level abnormal | 10037048 |
| Prothrombin level decreased | 10037050 |
| Prothrombin time abnormal | 10037057 |
| Prothrombin time prolonged | 10037063 |
| Prothrombin time ratio abnormal | 10061918 |
| Prothrombin time ratio increased | 10037068 |
| Radiation hepatitis | 10051015 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retinol binding protein decreased | 10048473 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Schistosomiasis liver | 10039610 |
| Small-for-size liver syndrome | 10069380 |
| Spider naevus | 10041519 |
| Splenic artery embolisation | 10083795 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Splenorenal shunt | 10041661 |
| Splenorenal shunt procedure | 10077281 |
| Spontaneous bacterial peritonitis | 10061135 |
| Spontaneous intrahepatic portosystemic venous shunt | 10076239 |
| Steatohepatitis | 10076331 |
| Stomal varices | 10075186 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Sustained viral response | 10076041 |
| Thrombin time abnormal | 10051319 |
| Thrombin time prolonged | 10051390 |
| Total bile acids increased | 10064558 |
| Transaminases abnormal | 10062688 |
| Transaminases increased | 10054889 |
| Ultrasound liver abnormal | 10045428 |
| Urine bilirubin increased | 10050792 |
| Urobilinogen urine decreased | 10070480 |
| Urobilinogen urine increased | 10070479 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| Viral hepatitis carrier | 10047458 |

| Weil's disease | 10047903 |
|------------------------------|----------|
| White nipple sign | 10078438 |
| Withdrawal hepatitis | 10071220 |
| X-ray hepatobiliary abnormal | 10056536 |
| Yellow skin | 10048245 |
| Zieve syndrome | 10048255 |

#### 14.5 Definitions of marked abnormalities

Where more than one assessment falls on the same day, the scheduled assessment is used above any non-scheduled (repeat or re-test or local) assessment for that parameter.

Laboratory analyses are based central laboratory data.

Marked laboratory abnormalities are displayed in Table 9, as described in the company standards

Table 9 Marked abnormalities in laboratory parameters for reporting

| Laboratory parameter | Criteria for marked laboratory abnormalities |
|---|---|
| Hematology (SI unit) | Circina for marked insortatory assistrations |
| | .00 |
| Hemoglobin (g/L) | < 80 |
| | < 100 |
| | > 20 above ULN or > 20 above baseline if baseline > ULN |
| | > 40 above ULN or > 40 above baseline if baseline > ULN |
| Hematocrit (L/L) | < 0.20 |
| | < 0.32 (Male) or < 0.28 (Female) |
| | > 0.60 (Male) or > 0.55 (Female) |
| | > 0.65 |
| Platelets (10 <sup>9</sup> /L) | < 50 |
| | < 75 |
| | > 600 |
| | > 999 |
| Leukocytes (10 <sup>9</sup> /L) | < 2.0 |
| | < 3.0 |
| | > 20.0 |
| | > 100.0 |
| Lymphocytes (10 <sup>9</sup> /L) | < 0.5 |
| | < 0.8 |
| | > 4.0 |
| | > 20.0 |
| Blood chemistry (SI unit) | |
| Alkaline phosphatase (U/L) | > 2.5 × ULN |
| | > 5 × ULN |
| Alanine aminotransferase | > 3 × ULN |
| (U/L) | > 5 × ULN |
| | > 8 × ULN |
| | > 10 × ULN |
| Aspartate aminotransferase | > 3 × ULN |
| (U/L) | > 5 × ULN |

| Laboratory parameter | Criteria for marked laboratory abnormalities |
|---|---|
| | > 8 × ULN |
| | > 10 × ULN |
| Total bilirubin (μmol/L) | >2 × ULN |
| | > 5 × ULN |
| Creatinine (µmol/L) | > 1.5 × ULN or > 1.5 × baseline if baseline < ULN |
| | $> 3 \times \text{ULN or} > 3 \times \text{baseline if baseline} < \text{ULN}$ |
| Potassium (mmol/L) | < 3.0 |
| | < 3.2 |
| | > 5.5 |
| | > 6.0 |
| Sodium (mmol/L) | < 130 |
| | > 150 |
| | > 155 |
| Gamma-glutamyl | > 2.5 × ULN |
| transferase (U/L) | > 5 × ULN |
| Urea nitrogen (mmol/L) | > 2.5 × ULN |
| | > 5 × ULN |

SI = standard international; ULN = upper limit of normal.